Official Title: PHASE I/IIA, OPEN-LABEL, SAFETY, TOLERABILITY, AND IMMUNOGENICITY

STUDY OF INO-3112 DELIVERED BY ELECTROPORATION (EP) IN WOMEN WITH CERVICAL CANCER AFTER CHEMORADIATION FOR NEWLY DIAGNOSED

DISEASE OR THERAPY FOR RECURRENT AND/OR PERSISTENT DISEASE

NCT Number: NCT02172911

**Document Date:** Protocol Version 2.1: 27 April 2016



# **HPV-004**

# PHASE I//IIA, OPEN-LABEL, SAFETY, TOLERABILITY, AND IMMUNOGENICITY STUDY OF INO-3112 DELIVERED BY ELECTROPORATION (EP) IN WOMEN WITH CERVICAL CANCER AFTER CHEMORADIATION FOR NEWLY DIAGNOSED DISEASE OR THERAPY FOR RECURRENT AND/OR PERSISTENT DISEASE

**Sponsored by:** 

Inovio Pharmaceuticals, Inc.

**BB-IND # 15,946** 

Version 2.1 27 April 2016

# PHASE I/IIA, OPEN-LABEL, SAFETY, TOLERABILITY, AND IMMUNOGENICITY STUDY OF INO-3112 DELIVERED BY ELECTROPORATION (EP) IN WOMEN WITH CERVICAL CANCER AFTER CHEMORADIATION FOR NEWLY DIAGNOSED DISEASE OR THERAPY FOR RECURRENT AND/OR PERSISTENT DISEASE

**Biologic Products:** INO-3112 (VGX-3100 and INO-9012)

**Protocol Number:** HPV-004

**Sponsor:** Inovio Pharmaceuticals, Inc.

660 West Germantown Pike, Suite 110

Plymouth Meeting, PA 19462

Principal Investigator:

Medical Monitor: , MD

Version and Date: Version 2.1 27 April 2016

# **CONFIDENTIAL**

The information in this document is considered privileged and confidential by Inovio Pharmaceuticals and may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Ethics committee approval and informed consent, or as required by local regulatory authorities. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Inovio Pharmaceuticals. Any supplemental information added to this document is also confidential and proprietary information of Inovio Pharmaceuticals and must be kept in confidence in the same manner as the contents of this document.

# **SUMMARY OF CHANGES**

The following is a list of significant protocol changes from v2.0 dated 12 June 2015 to v2.1 dated 27 April 2016. All other changes are administrative and do not significantly affect the safety of subjects, study scope, or scientific quality of the protocol.

- 1. The duration of the study changed from 3 years from last study treatment/EP to 36 weeks. This change still fulfills the study primary objectives, which include safety, tolerability and immunogenicity in subjects with cervical cancer and received INO-3112/EP treatment.
- 2. Updated the estimated number of Study Centers
- 3. Number of subjects to be enrolled in the study changed from 30 to 10 subjects. This is mainly due to study primary objectives and the challenge in trial operation/enrollment.
- 4. Specified in section 6.1.1 and 6.7 that the subjects with HPV-16 and/or HPV-18 positive from In-situ hybridization (ISH) or polymerase chain reaction (PCR) assays will be eligible for the study.
- 5. Added the option to conduct Weeks 2, 6, 8 and 10 visits as phone visit or inperson office visit. This change intends to be more convenient for study subjects.
- 6. Eliminated collection of the blood samples at Weeks 2, 4, 6, 10 and 14.
- 7. The medical monitor and associated contact information was updated to reflect a resourcing update by the Sponsor. All responsibilities of the updated medical monitor will remain the same.

# PROTOCOL ACKNOWLEDGEMENT

I have read this Protocol and agree that it contains all necessary details for carrying out the study described. I understand that it must be reviewed by the Institutional Review Board or Independent Ethics Committee overseeing the conduct of the study and approved or given favorable opinion before implementation.

The signature of the Principal Investigator and Sponsor below constitute their approval of this protocol and proved the necessary assurances that this study will be conducted according to The Declaration of Helsinki, GCP, ICH guidelines, local legal and regulatory regulations as well as to all stipulations of the protocol in both the clinical and administrative sections, including statements regarding confidentiality.

| Investigator's printed name and signature | Date |
|-------------------------------------------|------|
| , MD | Date |
| Medical Monitor | |

Protocol Number: HPV-004

Site Number:

Version Number/Version Date: v2.1/27 April 2016

# TABLE OF CONTENTS

| S | UMMA | RY OF CHANGES | 3 |
|---|---|---|---|
| T | ABLE | OF CONTENTS | 5 |
| C | LINICA | AL PROTOCOL SYNOPSIS | 9 |
| | Table | 1: HPV-004 Schedule of Events | .14 |
| 1 | | INTRODUCTION | . 16 |
| | 1.1 | Background and Rationale | . 16 |
| | 1.1.1 | Epidemiology of HPV Infection and Cervical Cancer | .16 |
| | 1.1.2 | Primary Prevention of HPV Disease: Screening and Prophylactic Vaccination 16 | on |
| | 1.1.3 | Rationale for a HPV Immunotherapy | .17 |
| | 1.1.4 | Target Organ for a Therapeutic HPV Immunotherapy – Skeletal Muscle | .20 |
| | 1.1.5 | Delivery Method – Injection / Electroporation (EP) | .20 |
| | 1.2 | Plasmid DNA Immunotherapy Agents (INO-3112) | .21 |
| | 1.2.1 V | VGX-3100 | .21 |
| | 1.2.2 I | NO-9012 | .21 |
| | 1.3 | Dose and Regimen Rationale | .21 |
| | 1.3.1 | Previous Human Experience with VGX-3100 | .22 |
| | 1.3.2 | Previous Human Experience with INO-9012 | .24 |
| | 1.4 | Risks/Benefit Assessment | . 25 |
| | 1.4.1 | Current Therapy for Stage IB-IVB Cervical Cancer | .25 |
| | 1.4.2 | Rationale for Study Design | .26 |
| | 1.4.3 | Potential Risks of DNA Immunotherapy Delivery with Electroporation | .28 |
| | 2 | HYPOTHESIS AND STUDY OBJECTIVES | . 29 |
| | 2.1 | Hypothesis | . 29 |
| | 2.2 | Primary Objective | . 29 |
| | 2.3 | Secondary Objective | . 29 |
| | 2.4 | Exploratory Objective | . 29 |
| 3 | | STUDY DESIGN | .30 |
| 4 | | SELECTION AND ENROLLMENT OF SUBJECTS | .32 |

| | 4.1 | Inclusion Criteria | 32 |
|---|---------|----------------------------------------------------------|-----|
| | | Exclusion Criteria | |
| | 4.3 | Supplementation of Study Subjects | |
| | 4.4 | Discontinuation/Withdrawal of Study Subjects | |
| 5 | | INVESTIGATIONAL PRODUCTS | |
| 3 | | | |
| | | Investigational Product | |
| | | Packaging and Labeling | |
| | 5.3 | Handling of INO-3112 | 36 |
| | 5.4 | Dispensing of INO-3112 | 37 |
| | 5.5 | Records of INO-3112 Disposition at Investigational Sites | 37 |
| | 5.6 | Return and Destruction of Investigational Products | 37 |
| | 5.7 | Use of CELLECTRA®-5P Electroporation Device | 38 |
| | 5.8 | Investigational Device Accountability | 38 |
| 6 | | STUDY PROCEDURES AND TREATMENTS | 39 |
| | 6.1 | Procedure by Visit | 39 |
| | 6.1.1 | Screening Evaluations | 39 |
| | 6.1.2 | Study Evaluations | 40 |
| | 6.2 | Timing and Evaluations | 43 |
| | 6.2.1 | Informed Consent | 43 |
| | 6.2.2 | Assignment of Screening/Allocation Numbers | 43 |
| | 6.2.3 | Medical History | 43 |
| | 6.2.4 | Safety Assessments | 44 |
| | 6.2.4.2 | Physical Assessments | 44 |
| | 6.2.4.3 | Post-Treatment Reaction Assessment | 44 |
| | 6.2.4.4 | Participant Reminder C | ard |
| | 6.2.4.5 | Vital Signs | 45 |
| | 6.2.4.6 | Weight and Height | 45 |
| | 6.2.4.7 | 12-lead ECGs | 45 |
| | 6.2.4.8 | Pregnancy Test | 45 |
| | 6.2.4.9 | Laboratory Evaluations | 46 |

| | 6.2.4. | 10 | Γ/CT Scan |
|---|---|---|---|
| | 6.3 | Study Treatment/EP with INO-3112 | 47 |
| | 6.3.1 | Management of anxiety and pain due to EP procedure | 47 |
| | 6.4 | Assessment of Clinical Adverse Events | 48 |
| | 6.5 | Assessment of Laboratory Abnormalities | 48 |
| | 6.6 | Assessment of Injection Site Reactions | 48 |
| | 6.7 | Cervical Virologic and Peripheral Blood Immunogenicity Assessment | t49 |
| | 6.8 | Disease Status | 52 |
| | 6.9 | Concomitant Medications/Medical Care | 52 |
| | 6.10 | Permitted Supportive Therapy | 52 |
| | 6.11 | HLA Testing | 52 |
| | 6.12 | Downloading of EP data from CELLECTRA®-5P device | 52 |
| | 6.13 | Restrictions | 52 |
| 7 | | EVALUATION OF SAFETY AND MANAGEMENT OF TOXICITY | Y 53 |
| | 7.1 | Safety Parameters | 53 |
| | 7.1.2 | Serious Adverse Events (SAEs) | 54 |
| | 7.1.3 | Severity Codes for AEs | 55 |
| | 7.2 | Causal Relationship of Clinical Material to AEs | 56 |
| | 7.2.1 | Abnormal Laboratory Value | 56 |
| | 7.2.2 | Post-Study Reporting Requirements | 57 |
| | 7.3 | Methods and Timing of the Collection and Recording of Safety Data. | 57 |
| | 7.4 | Procedures for Documenting Pregnancy During Study | 58 |
| | 7.5 | Toxicity Management | 58 |
| | 7.5.1 | Criteria for Halting of Study Enrollment | 58 |
| | 7.5.2 | Events Requiring Expedited Reporting | 59 |
| | 7.5.3 | Stopping Rules (Criteria for Pausing of Study) | 59 |
| 8 | | STATISTICAL CONSIDERATIONS | 60 |
| | 8.1 | Sample Size Considerations | 60 |
| | 8.3 | Analysis of Immune Responses | 60 |
| | 8.4 | Analysis of Clinical Responses | 60 |

| 8.5 | Summary of Demographic and Other Baseline Characteristics | .60 |
|---|---|---|
| 8.6 | Missing Values | .60 |
| 8.7 | Site Effects | . 60 |
| 9 | DATA COLLECTION, MONITORING, AND AE REPORTING | .61 |
| 9.1 | Records to Be Kept | .61 |
| 9.2 | Safety and Quality Monitoring and Record Availability | .61 |
| 9.3 | Adverse Experience (AE) Reporting | . 62 |
| 9.3.1 | Study Reporting Period of Adverse Events | .62 |
| 9.3.2 | Study Reporting Period of Serious Adverse Events | .62 |
| 9.3.3 | Notification of Serious Adverse Events | .63 |
| 9.4 | Reporting of Device Related Complaints | . 64 |
| 9.5 | Study Discontinuation | . 64 |
| 10 | PUBLICATION OF RESEARCH FINDINGS | . 64 |
| 11 | LIST OF ABBREVIATIONS | . 66 |
| 12 | REFERENCES | . 68 |
| 13 | APPENDICES | .73 |
| 13.1 | Appendix 1: Subject Identification Fax Form | .73 |
| 13.2 | Appendix 2: ECOG Performance Status | . 74 |
| 13.3 | Appendix 3: Standard Chemoradiation Guidelines | .75 |
| 13.4 | Appendix 4: Common Terminology Criteria for Adverse Events (CTCAE) | ) |
| | Version 4.03 dated June 14, 2010 | .85 |
| 13.5 | Appendix 5: Acute Radiation Morbidity Scoring Criteria (RTOG) | . 86 |
| 13.6 | Appendix 6: Preparation of Investigational Products | .88 |
| 13.7 | Appendix 7: CELLECTRA®-5P Error Reporting Form | . 89 |
| 13.8 | Appendix 8: New York Heart Association (NYHA) Functional | 1 |
| | Classification | .90 |
| 13.9 | Appendix 9: Participant Reminder Card | .91 |
| 13.10 | Appendix 10: RECIST | .92 |

# CLINICAL PROTOCOL SYNOPSIS

**Title of Study**: Phase I/IIA, Open-Label, Safety, Tolerability, and Immunogenicity Study of INO-3112 Delivered by Electroporation (EP) in Women with Cervical Cancer after Chemoradiation for Newly Diagnosed Disease or Therapy for Recurrent and/or Persistent Disease

**Estimated Number of Study Centers and Countries/Regions:** 2 sites (United States)

Number of Subjects : Approximately 10 subjects

Study Phase: I/IIa

**Research Hypothesis:** Immunotherapy with INO-3112 delivered by intramuscular (IM) injection followed by EP with CELLECTRA®-5P will be immunogenic and well tolerated in women with newly diagnosed, inoperable cervical cancer associated with HPV-16 and/or HPV-18 after completion of standard chemoradiation therapy with curative intent (Cohort 1) or in women with persistent and/or recurrent cervical cancer associated with HPV-16 and/or HPV-18 following salvage therapy (Cohort 2) and will not be associated with any significant increased toxicity compared to that expected/reported with "standard" therapy alone.

# **Primary Objective:**

• Evaluate the safety and tolerability of immunotherapy with INO-3112 when delivered IM followed by EP with CELLECTRA®-5P in women with newly diagnosed, inoperable cervical cancer associated with HPV-16 and/or HPV-18 after completion of standard chemoradiation therapy with curative intent (Cohort 1) or in women with persistent and/or recurrent cervical cancer associated with HPV-16 and/or HPV-18 following salvage therapy (Cohort 2) compared to that expected/reported with "standard" therapy alone.

# **Secondary Objective:**

• Evaluate the cellular and humoral immune responses to immunotherapy with INO-3112 delivered IM followed by EP with CELLECTRA®-5P in women with newly diagnosed, inoperable cervical cancer associated with HPV-16 and/or HPV-18 after completion of standard chemoradiation therapy with curative intent (Cohort 1) or in women with persistent and/or recurrent cervical cancer associated with HPV-16 and/or HPV-18 following salvage therapy (Cohort 2).

# **Exploratory Objective:**

• Evaluate clinical responses (disease-free survival and progression-free survival) following treatment with INO-3112 delivered intramuscularly followed by EP with CELLECTRA®-5P in women with newly diagnosed, inoperable cervical cancer associated with HPV-16 and/or HPV-18 after completion of standard chemoradiation therapy with curative intent (Cohort 1) or in women with persistent and/or recurrent cervical cancer associated with HPV-16 and/or HPV-18 following salvage therapy (Cohort 2).

**Study Design:** This is a Phase I/IIa, open-label study to evaluate the safety, tolerability, and immunogenicity of INO-3112 [6 mg of VGX-3100 (2 separate DNA plasmids encoding E6 and E7 proteins of HPV 16 and HPV 18) and 1 mg of INO-9012 (DNA plasmid encoding human interleukin 12)] delivered IM by EP in approximately 10 female subjects with biopsy-proven, Stage IB-IVB inoperable invasive cervical carcinoma associated with HPV-16 and/or HPV-18 who have completed treatment with standard chemoradiation therapy with curative intent (Cohort 1) or in subjects with persistent and/or recurrent cervical cancer associated with HPV-16 and/or HPV-18 following salvage therapy (Cohort 2).

Eligible subjects who consent to participate in the study will receive a 1.1 mL IM injection of INO-3112 in the deltoid followed immediately by EP with CELLECTRA®-5P. If the deltoid is not a suitable location, the IM injection should be in the lateral quadriceps followed immediately by EP with CELLECTRA®-5P. All subjects (Cohorts 1 and 2) will receive a 4-dose series of INO-3112. The first study treatment/EP after completion of standard chemoradiation (Cohort 1) or salvage therapy (Cohort 2) will be designated as "Day 0", the second dose will be administered at Week 4, the third dose at Week 8, and the fourth (final) treatment will be administered at Week 12.

# Cohort 1:

Cohort 1 will include subjects with biopsy-proven, Stage IB-IVB inoperable, newly diagnosed, invasive cervical carcinoma associated with HPV-16 and/or HPV-18 treated with standard chemoradiation therapy with curative intent.

All subjects in Cohort 1 must receive their first study treatment (Day 0) within 2 weeks after completing a course of standard radiation therapy (external beam and brachytherapy) administered concurrently with platinum based therapy with curative intent. (Refer to Appendix 3: Standard Chemoradiation Guidelines)

# Cohort 2:

Cohort 2 will include subjects with persistent and/or recurrent cervical carcinoma associated with HPV-16 and/or HPV-18 treated with salvage therapy (chemotherapy and/or radiation therapy).

All subjects in Cohort 2 must receive their first study treatment (Day 0) no sooner than 2 weeks and no later than 4 weeks after completing a course of salvage therapy. If in the investigators opinion, there are no additional salvage therapy options, the subject may be enrolled in Cohort 2 without having received salvage therapy immediately prior to enrollment.

# **Primary Safety Endpoints:**

- 1. Incidence of adverse events (all, severe [graded per Common Toxicity Criteria for Adverse Events (CTCAE) v4.03], unexpected, serious) classified by system organ class (SOC), preferred term, severity, and relationship to study medication and schedule
- 2. Injection site reactions including pain, tenderness, erythema and induration at the administration site
- 3. Rates of acute gastrointestinal, genitourinary, or other chemoradiation side effects above the expected, graded per Acute Radiation Morbidity Scoring Criteria (RTOG)
- 4. Changes in laboratory parameters from baseline

# **Study Design Contd.:**

# Secondary Immunologic Endpoints:

- 1. Antigen-specific cellular immune responses to INO-3112 in blood samples obtained from subjects per study schedule:
  - a. Interferon- $\gamma$  secreting T lymphocytes in PBMC by ELISpot
  - b. Flow Cytometry for T-cell activation, cytolytic phenotype, and memory phenotype in PBMC
- 2. Antigen-specific humoral responses to HPV–E6 and –E7 by ELISA per study schedule

# **Exploratory Clinical Endpoints:**

- Changes in standard uptake volume (SUV) on PET/CT scans performed at baseline vs followup PET/CT scans obtained at specified time points
- 2. Evaluation of subjects relative immune competence longitudinally throughout the study starting at the screening visit (for details refer to Section 6.7: Cervical Virologic and Peripheral Blood Immunogenicity Assessment)
- 3. Changes in cervical histology from the screening biopsy as compared to the week 16 biopsy
- 4. Local immune responses to INO-3112 in tumor tissue samples obtained at week 16
- 5. Disease-free survival assessed in accordance with RECIST v1.1 (refer to Appendix 10) as follows:
  - Clinical evaluations for disease response will be conducted at all study visits (as assessed by clinical signs and symptoms of disease progression)
  - A baseline PET/CT scan will be obtained on each subject within 4 weeks prior to Day 0 and then PET/CT scans for disease progression will be obtained for all subjects 3-4 months after Day 0 and 3-5 months thereafter per standard of care/in accordance with local guidelines and institutional practices. Additional PET/CT scans may be obtained at other time points if clinically indicated to confirm a clinical diagnosis of disease progression based on signs and symptoms.

# Inclusion Criteria

- a) Written informed consent in accordance with institutional guidelines. If required by local law, candidates must also authorize the release and use of protected health information (PHI);
- b) Female subjects age 18 years or older;
- c) Histological diagnosis of squamous cell carcinoma, adenocarcinoma or adenosquamous cell carcinoma of the cervix. Not accepted are small cell, clear cell and other rare variants of the classical adenocarcinoma;
- d) Histologically confirmed, Stage IB-IVB, invasive cervical carcinoma associated with HPV-16 and/or HPV-18 and meeting the following eligibility criteria for either Cohort 1 or Cohort 2;

# Inclusion Criteria Contd.

## 1. Cohort 1

- Newly diagnosed inoperable cervical cancer treated with chemoradiation therapy with curative intent and a life expectancy of at least 12 months as assessed by the investigator.
  - No CNS/spinal metastases
- Able to initiate study treatment (Day 0) within 2 weeks of completion of last chemoradiation treatment;
  - Platinum based treatment (alone or in combination with other drugs); 5 weekly courses of Cisplatin 40 mg/m² completed within 10 weeks of its initiation
  - Standard radiation therapy (external beam and brachytherapy); completed within 10 weeks of its initiation
  - o Brachytherapy; must be the last treatment if the subject is receiving sequential brachytherapy following the chemoradiation therapy

# 2. Cohort 2

- Persistent and/or recurrent cervical cancer
  - No CNS/spinal metastases
- Able to initiate study treatment (Day 0) at least 2 weeks after but no more than 4 weeks after completion of salvage therapy (If in the investigators opinion, there are no additional salvage therapy options, the subject may be enrolled in Cohort 2 without having received salvage therapy immediately prior to enrollment.)
- Subject has a life expectancy of at least 12 months as assessed by the investigator
- e) ECG with no clinically significant findings as assessed by the investigator performed within 30 days of signing the informed consent form (ICF);
- f) Chemistry, liver function tests, renal function, total creatine phosphokinase (CPK) and hematology lab results must be ≤ Grade 1 at the time of screening, in accordance with the CTCAE v4.03;
- g) Eastern Cooperative Oncology Group (ECOG) Performance status of  $\leq 1$ ;
- h) Adequate venous access for repeated blood sampling according to study schedule;
- i) Women of child-bearing potential must have a negative serum pregnancy test and agree to remain sexually abstinent, have a partner who is sterile (i.e., vasectomy), or use two medically effective methods of contraception (e.g., oral contraception, barrier methods, spermicide, intrauterine device (IUD)). This requirement should be followed from screening through 24 weeks after last study treatment/EP. Whole pelvis external beam radiation therapy (EBRT) followed by intracavitary (IC) therapy for cervical cancer is considered to be an irreversible form of contraception;
- j) Able and willing to comply with all study procedures.

# Exclusion Criteria:

- a) Pregnancy or breastfeeding;
- b) History of previous <u>therapeutic</u> HPV vaccination (individuals who have been immunized with licensed prophylactic HPV vaccines (e.g. Gardasil®, Cervarix®) are not excluded);
- c) Prior exposure to an investigational agent or device within 30 days of signing the ICF. Of note, the subject may participate in observational studies;
- d) Positive serological test for human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C or history of HIV infection, Hepatitis B or Hepatitis C (women with cured HCV will be allowed; subject must have had an serologic test performed within 12 months of informed consent);
- e) Prior major surgery within 4 weeks of first study treatment/EP from which the subject has not yet recovered to baseline;
- f) High medical risks because of non-malignant systemic disease or with active uncontrolled infection;
- g) Current malignancies at other sites, with the exception of adequately treated basal or squamous cell carcinoma of the skin;
  - Cancer survivors, who have undergone curative therapy for a prior malignancy, have no evidence of that disease for five years and are deemed at low risk for recurrence, are eligible for the study;
- h) Congestive heart failure or prior history of New York Heart Association (NYHA) class III/ IV cardiac disease (refer to Appendix 8);
- i) Any concurrent condition requiring the continued use of systemic or topical steroids at or near the injection site, excluding non-systemic (e.g. inhaled and eye drop-containing) corticosteroids or the use of other immunosuppressive agents. All other corticosteroids must be discontinued > 4 weeks prior to Day 0 of study product administration;
- j) Any cardiac pre-excitation syndromes (such as Wolff-Parkinson-White);
- k) History of seizures (unless seizure free for 5 years);
- 1) Less than two acceptable sites exist for IM injection and EP between use of the deltoid and lateral quadriceps muscles. A site for injection/EP is not acceptable if there are tattoos or scars within 2 cm of the injection/EP site or if there is implanted metal within the same limb. Any device implanted in the chest (e.g., cardiac pacemaker or defibrillator) excludes the use of the deltoid muscle on the same side of the body;
- m) Administration of any non-study related vaccine within 2 weeks of Day 0;
- n) Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements;
- o) Imprisonment or compulsory detainment (involuntary incarceration) for treatment of either a psychiatric or physical (i.e. infectious disease) illness;
- p) History of immunosuppressive or autoimmune disease;
- **q)** Any other illnesses or conditions that in the opinion of the investigator may affect the safety of the subject or limit the evaluation of a subject or any study endpoint.

Table 1: HPV-004 Schedule of Events

| Torde | - C | DA | Weeks <sup>a</sup> | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Tests | S | D0 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 24 | 32 | 36 |
| | | Study | Proc | edur | es | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | |
| Medical and CIN/Cancer history | X | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | X | X | | | | | | | | | | | |
| Physical exam/assessment <sup>c</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| ECOG performance status | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Medical/Clinical assessment | X | X | $X^{b}$ | X | $X^{b}$ | X | Xb | X | Xb | X | X | X | X |
| Chemo/RT Effects/Adverse Events | X <sup>m</sup> | X | $X^{b}$ | X | | | | | | | | | |
| Adverse events | X | X | $X^{b}$ | X | $X^{b}$ | X | $X^{b}$ | X | $X^{b}$ | X | X | X | X |
| Concomitant medications | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Disease Status <sup>d</sup> | X | | | | | | | | | X | | X | X |
| Vital signs (Height and Weight) <sup>e</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG | X | | | | | | | | | | | | |
| Histologic HPV assessment <sup>f</sup> | X | | | | | | | | | | | | |
| Tumor biopsy collection | X <sup>l</sup> | | | | | | | | | X | | | |
| ThinPrep <sup>TM</sup> sample (if obtainable) | X | X | | | | | | | | X | | | X |
| Digene swab (2) (if obtainable) | X | X | | | | | | | | X | | | X |
| PET/CT scan | X <sup>n</sup> | | | | | | | | | Xp | | $X^q$ | $X^q$ |
| | La | borat | ory P | roceo | lures | | • | | | | | | |
| CBC w/ differential | X | Xº | | Xº | | Xº | | Xº | | Xº | | | |
| Serum chemistry <sup>g</sup> | X | Xº | | Xº | | Xº | | Xº | | Xº | | | |
| Urinalysis <sup>h</sup> | X | | | | | | | | | | | | |
| СРК | X | | | | | | | | | Xº | | | |
| Pregnancy Test <sup>i</sup> | X | X | | X | | X | | X | | X | | | |
| HIV/ hepatitis serology | X | | | | | | | | | | | | |
| Blood immunologic samples <sup>j,</sup> | X | X | | | | X | | | | X | X | X | X |
| | Imm | unoth | erapy | Pro | cedui | res | | | | | | | |
| Immunotherapy/EP | | X | | X | | X | | X | | | | | |
| Post treatment reaction <sup>k</sup> | | X | $X^{b}$ | X | $X^{b}$ | X | $X^{b}$ | X | $X^{b}$ | X | | | |
| Download EP data | | X | | X | | X | | X | | | | | |
| Participant Reminder Card | | X | | X | | X | | X | | | | | |
| Review participant reminder card | | | $X^{b}$ | X | $X^{b}$ | X | $X^{b}$ | X | $X^{b}$ | X | | | |

Wks 2, 6, 8 and 14 visits may be performed as an in-person office visit or a telephone call. After completing medical/clinical assessment, reviewing PRC and collecting information on AE with the subject on the phone, the investigator will determine whether an office visit is needed for further evaluation.

Cohort 1: Subjects in Cohort 1 can be screened either prior to initiation of chemoradiation, or during chemoradiation and should be enrolled such that their first study treatment (Day 0) will be delivered within 2 weeks of completing their chemoradiation therapy;

Cohort 2: Subjects in Cohort 2 can be screened and enrolled such that their first study treatment (Day 0) is no sooner than 2 weeks and no later than 4 weeks after completing the salvage therapy. If in the

- investigators opinion, there are no additional salvage therapy options, the subject may be enrolled in Cohort 2 without having received salvage therapy immediately prior to enrollment.
- <sup>a</sup> Procedures and visits scheduled from Day 0 through Wk 16 must occur  $\pm 1$  week of scheduled time. Procedures and visits scheduled from Week 24 to Week 36 must occur  $\pm 2$  weeks of scheduled time.
- <sup>b</sup> assessment to be performed if visit done as phone-call
- <sup>c</sup> Targeted physical examination at all visits except full examination at screening (includes complete gynecological exam) and discharge visit
- <sup>d</sup> Disease status should be categorized into 1) No evidence of disease (NED) 2) Partial Response 3) Stable disease 4) Progressive disease
- <sup>e</sup>Temperature, respiratory rate, blood pressure, heart rate, weight and height. Height collected at screening only
- f Paraffin embedded tissue obtained for diagnosis of cervical cancer must be available for HPV testing
- <sup>g</sup> Serum chemistry includes glucose, albumin, total protein, SGPT, SGOT, alkaline phosphatase, total bilirubin, blood urea nitrogen (BUN), calcium, creatinine, electrolytes (sodium, potassium, chloride, carbon dioxide or bicarbonate)
- <sup>h</sup> Urine samples will be tested by dipstick for glucose, protein, and hematuria.
- i Serum pregnancy test required at screening. Urine pregnancy test should be used prior to tumor biopsy and prior to each study treatment/EP
- <sup>j</sup> At least 34 mL (4 x 8.5 mL tubes) whole blood in Acid Citrate Dextrose tubes and 4 mL serum per time point. A total of at least 68 mL whole blood and 4 mL serum should be collected prior to dosing on Day 0
- <sup>k</sup> Assessed 30 to 45 minutes after study treatment/EP and at post-treatment visits
- <sup>1</sup>A tumor biopsy collection is required at screening if residual tissue and/or unstained slides are not available
- <sup>m</sup> Chemo/RT effects to be assessed at screening if subject is screened during chemoradiation
- <sup>n</sup> PET/CT to include standard uptake volume, must be performed within 4 weeks prior to Day 0
- <sup>o</sup> All labs for Day 0 and those associated with any treatment visit should be available prior to treatment and collected no more than 48 hours prior to treatment
- <sup>p</sup> PET/CT will be performed 3-4 months after Day 0
- <sup>q</sup> Not required at study discharge if performed at wk 32
- <sup>r</sup>Immune competence will be evaluated longitudinally throughout the study from the time of screening visit. No additional blood collection required.

# 1 INTRODUCTION

# 1.1 Background and Rationale

# 1.1.1 Epidemiology of HPV Infection and Cervical Cancer

More than 200 genotypes of human papillomavirus (HPV) are known, of which approximately 40 can infect the anogenital mucosa [World Health Organization 2008]. Persistent infection with oncogenic HPV genotypes is the proximate cause of virtually every squamous cervical cancer. HPV types 16 and 18 are the most prevalent types of highly oncogenic HPV associated with cervical cancer, accounting for approximately two-thirds of all cases of cervical cancer [Munoz 2003].

HPV infection is characterized by ongoing viral replication and shedding, and is associated with early pathologic changes (cervical intraepithelial neoplasia; CIN). Most genital HPV infections clear spontaneously. Persistent infection with a highly oncogenic HPV type is associated with integration of the viral genome into the host genome, with subsequent constitutive expression of the viral proteins, E6 and E7. Expression of these oncoproteins is functionally required for disease initiation and persistence, as E6 binds and targets p53 for degradation, and E7 targets pRb. Viral integration is found in high grade cervical dysplasia (CIN2/3), the intraepithelial lesion which is the immediate precursor to invasive disease. The vast majority of invasive cancers of the cervix are thought to arise from untreated CIN2/3 [Munger 2002]. Because these viral, non-'self' proteins are functionally required for disease, and are expressed only in diseased tissue, not in normal cells, they present compelling antigenic targets for therapeutic vaccination.

# 1.1.2 Primary Prevention of HPV Disease: Screening and Prophylactic Vaccination

Despite screening programs that have dramatically reduced the incidence of cervical cancer, approximately 12,900 American women are diagnosed with this disease annually, and 4100 die from it [ACS 2015]. Worldwide, cervical cancer is the fourth most common cancer in women resulting in approximately 268,000 deaths yearly [GLOBOCAN 2012].

In 2006, the U.S. Food and Drug Administration (FDA) licensed a quadrivalent HPV vaccine for use in females 9-26 years of age to prevent diseases caused by HPV types 6, 11, 16 and 18 [Centers for Disease Control and Prevention 2007]. The primary analysis of a prospective, randomized, double-blind, trial involving 10,565 women 15-26 years of age with no virologic evidence of infection by HPV 16 or 18, who were randomized 1:1 to receive a 3-dose course of vaccine or placebo, found the vaccine efficacy for prevention of the primary composite endpoint (prevention of HPV-16 or 18 infection resulting in CIN2 or 3) after 3 years to be 98% (95% C.I. 86%, 100%) [Future II Study Group 2007]. In October 2009, a bivalent vaccine was approved for use in women to prevent diseases caused by HPV types 16 and 18.

Recently available prophylactic HPV vaccines are unlikely to impact the burden of disease in the near future; protection is type-specific, and vaccine delivery requires intense infrastructure, including the need for three inoculations. Indeed, in the United States, only 44% of eligible teen (13-17 years) girls received any HPV vaccine, and ~27% completed the three-vaccination series in 2009. Furthermore, ensuring vaccination prior to HPV exposure can be challenging [CDC 2010].

# 1.1.3 Rationale for a HPV Immunotherapy

While the currently available prophylactic HPV vaccines are highly effective in preventing infection and the development of high-grade CIN caused by HPV types 16 and 18, these have no therapeutic effect, and therefore are of no value for women already infected with these oncogenic types. Treatment for CIN 2/3 usually consists of either surgical removal of the affected tissue by cone biopsy or a loop electrical excision procedure (LEEP), or ablative therapy via laser, or cryotherapy. Invasive cervical cancer may be treated by radical hysterectomy, and/or combination radiation and chemotherapy.

Intraepithelial HPV disease is indolent, and not all CIN 2/3 progress to invasive disease. In fact, in immune-competent subjects, spontaneous regression of CIN 2/3 over a relatively brief timeframe of 6 months is estimated at 30-40% [Trimble 2005, Castle 2009, Moscicki 2010]. In subjects with CIN 2/3 associated with HPV-16, the rate of spontaneous regression is lower, in the range of 25% [Trimble 2005, Castle 2009, Moscicki 2010]. Boosting cell-mediated immune responses to the early HPV E6 and E7 proteins may lead to elimination of immortalized cells and so prevent the development of invasive disease. [Kenter 2009]. The ability of immunotherapy with VGX-3100 delivered by EP to reverse high grade dysplasia is currently being studied in a prospective global, placebocontrolled, randomized phase 2 study in women with CIN2 and CIN3 associated with HPV-16 and/or HPV-18. A pre-planned interim analysis of the study data completed in July 2014 revealed that the study met its primary endpoint (histopathologic regression of lesions) and secondary endpoint (histopathologic regression of lesions in the context of elimination of HPV16 and/or 18 infection) demonstrating a highly statistically significant improvement in the VGX-3100 arm (p<0.017 and p<0.001 respectively). Treatment of HPV16 and/or 18 positive patients with CIN2 or 3 was generally safe as evidenced by the lack of statistical significance between the frequencies of adverse events reported in the placebo arm as compared to the VGX-3100 treated arm. Treatment with VGX-3100 was able to induce a robust immune response in the periphery as gauged by IFNg ELISpot as well as in the tissue as examined using immunohistochemistry. These data reveal the highly promising potential of therapeutic immunization with DNA followed by electroporation for the treatment of HPV-16 and/or HPV-18 related precancerous cervical disease in women.

There is early data regarding the use of therapeutic vaccines for cervical cancer which does appear to demonstrate some HPV-specific antibody response in pre-

clinical and early clinical studies [Borysiewicz 1996, Cui 2005, Cui 2006, Jochmus 1999, Liu 2000, Ohlschlager 2009, Welters 2008].

Some clinical studies have employed the combination of radiotherapy with immunotherapy and have been shown to induce tumor-specific and innate immunity [Chi 2005, Gulley 2005]. Radiation has been shown to increase immunogenicity of solid tumors by several mechanisms, including enhancing the expression of MHC class I molecules [Reits 2006], as well as increasing expression of adhesion molecules by endothelial cells [Gaugler 1997]. These and other phenotypic changes subsequent to radiation render established disease more susceptible to T-cell-mediated lysis [Garnett 2004]. Chemotherapeutic regimens, including cisplatin (CDDP) can also render solid tumors more susceptible to immunologic intervention [Gelbard 2006, Matsuzaki 2000].

However, to date, there are limited data investigating the use of a therapeutic vaccine for cervical cancer in the setting of chemoradiotherapy. Encouraging synergistic results have been demonstrated in animal models [Tseng 2009]. It was observed that TC-1 tumor-bearing mice treated with radiotherapy combined with CRT/E7(detox) DNA vaccination generated significant therapeutic anti-tumor effects and the highest frequency of E7-specific CD8<sup>+</sup> T-cells in the tumors and spleens of treated mice. Furthermore, treatment with radiotherapy was shown to render the TC-1 tumor cells more susceptible to lysis by E7-specific CTLs (cytotoxic T lymphocytes). In addition, it was observed that treatment with radiotherapy during the second DNA vaccination generated the highest frequency of E7-specific CD8<sup>+</sup> T-cells in the tumors and spleens of TC-1 tumor-bearing mice. Finally, TC-1 tumor-bearing mice treated with the chemotherapy in combination with radiation and CRT/E7(detox) DNA vaccination generated significantly enhanced therapeutic anti-tumor effects [Tseng 2009].

Rationale for DNA based Immunotherapy: DNA vaccines have several advantages over traditional vaccines such as live attenuated virus and recombinant protein-based vaccines (engineered specificity, production, safety). To date, DNA vaccines have been well-tolerated in humans. In fact, clinical data from hundreds of subjects vaccinated with DNA vaccines suggests that intramuscular administration alone elicits barely detectable systemic immune responses to vaccine antigens. Preclinical safety studies in the literature have not demonstrated evidence of plasmid integration [Martin 1999, Nichols 1995]. Similar results were obtained in the pre-clinical safety and toxicology studies performed with VGX-3100 in rabbits. In our studies with VGX-3100, the rates of plasmid clearance from the injection site skin and muscle were similar whether the plasmid was delivered with or without electroporation suggesting that the delivery method did not result in an increased persistence at the injection site.

Unlike viral vector-based constructs, DNA vaccines can be used for repeated administration as the efficacy of plasmid vectors are not influenced by pre-existing neutralizing antibodies [Chattergoon 1997]. Furthermore, the ability to engineer specific targeting of multiple antigenic components allows the inclusion of specific immunogens, adjuvants or targeting sequences. VGX-3100 is

comprised of plasmids targeting E6 and E7 proteins of both HPV subtypes 16 and 18, and is delivered via electroporation (EP) using the CELLECTRA®-5P constant current device.

Individual candidate vaccine plasmids were developed for both HPV-16 (pCon16E6E7) and HPV-18 (pCon18E6E7), pre-clinical expression and immunogenicity were demonstrated, and then the plasmids were combined and formulated to produce VGX-3100. Preclinical toxicology and biodistribution studies with VGX-3100 have demonstrated an acceptable safety profile in the New Zealand White Rabbit.

Several pre-clinical studies were performed to further characterize the two plasmids. The immunogenicity of DNA delivered by intramuscular (IM) injection alone was compared to DNA delivery via electroporation (IM+EP). Immunogenicity was compared to vector-alone controls in mice and non-human primates (rhesus macaques).

HPV-16 and HPV-18 E6 and E7 proteins were appropriately expressed and processed in two separate animal studies (mouse and rhesus macaques). Indeed in both cases, robust cell mediated immune (CMI) responses were elicited. CMI responses were enhanced by about 3-fold using EP delivery vs. DNA alone at doses as low as 10  $\mu$ g when delivered by EP. Further, CMI was elicited for both the HPV-16 and 18 constructs based on similar ELISpot results.

A side-by-side comparison at the low DNA dose indicated that the responses were approximately 3-fold greater when delivered via IM+EP compared to IM alone. Similar levels of CMI responses were elicited when the plasmid DNA was delivered at a 10-fold higher dose using IM alone suggesting that the use of EP technology will pave the way for development of dose-sparing immunotherapy agents. Importantly, in both cases, the epitopes recognized were well characterized E6 and E7 epitopes suggesting that normal effective processing of antigens occurs following vaccination regardless of whether the antigens were delivered via IM+EP or IM alone. This phenomenon has been observed in preclinical studies with other DNA plasmid candidates as well (e.g. influenza, HIV), where the magnitude of response is increased when DNA vaccines are delivered via EP.

Finally, efficacy of the pCon16E6E7 plasmid was assessed in a mouse tumor challenge model using the TC-1 cell-line which expresses HPV-16 E6 and E7 proteins [Yan 2009]. Mice were challenged with TC-1 tumor cells at low dose (5x10<sup>4</sup>) on Day 0. Three days after TC-1 cell implantation, ten mice were immunized with pVAX, a plasmid containing HPV16 E7 only (pE7) and pCon16E6E7 and boosted twice on day 10 and 17.

Only three out of ten mice in pCon16E6E7 vaccinated group developed tumors 49 days after initial tumor implantation. All mice in the pE7 group eventually developed tumors; however, the tumors in this group were smaller than those in the control group (p<0.05). In order to further assess the therapeutic potential of pCon16E6E7, we performed another tumor regression study by increasing the

challenge dose of TC-1 cells to  $1x10^6$  and mice were not immunized with pCon16E6E7 until the average tumor size was about 6 mm (on day 7). After boosting four times, mice in pCon16E6E7 group developed significantly smaller tumors compared to those in the control group (p<0.05). Moreover, all mice in pCon16E6E7 group survived 49 days after tumor implantation. In contrast, none of the mice in the pVAX group survived 28 days after tumor implantation. These results indicate that the DNA vaccine pCon16E6E7 induced regression of well-established tumors in C57BL/6 mice. The efficacy of pCon18E6E7 was not assessed due to the lack of a suitable tumor challenge model for HPV-18 related tumors [Yan 2009].

VGX-3100, HPV therapeutic vaccine is a combination of two plasmids in equal quantities (*i.e.* the 6 mg dose will deliver 3 mg of each pGX3001 and pGX3002 plasmids):

- a) pGX3001: p16ConE6E7, a plasmid encoding for a synthetic HPV16 consensus (SynCon<sup>TM</sup>) E6 and E7 fusion gene into a pVAX1 backbone (Invitrogen, Carlsbad, CA) under the control of the cytomegalovirus immediate-early (CMV) promoter, and
- b) pGX3002: p18ConE6E7, a plasmid encoding for a synthetic HPV18 consensus (SynCon<sup>TM</sup>) E6 and E7 fusion gene into a pVAX1 backbone (Invitrogen, Carlsbad, CA) under the control of the cytomegalovirus immediate-early (CMV) promoter.

Both HPV type 16 and 18 E6 and E7 consensus nucleotide sequences were synthetically produced (GeneArt, Germany) after performing multiple alignments of the sequences described in the international genetic database (GenBank) for HPV type 16 and 18.

# 1.1.4 Target Organ for a Therapeutic HPV Immunotherapy – Skeletal Muscle

The skeletal musculature is an excellent candidate for the target tissue of gene expression, because muscle fibers have a long lifespan and can be transduced by circular plasmids, allowing the gene to be expressed efficiently in immunocompetent hosts [Davis 1993; Tripathy 1996]. Furthermore, muscle is well vascularized, allowing the newly produced transgene product to gain access to the circulation.

# 1.1.5 Delivery Method – Injection / Electroporation (EP)

The use of EP via the CELLECTRA®-5P device increases the expression of INO-3112. EP utilizes a transmembrane electric field pulse to induce microscopic pathways (pores) in a bio-membrane. The electric field allows macromolecules, ions, and water to pass from one side of the membrane to the other. The presence of a constant field influences the kinetics of directional translocation of the macromolecular plasmid, such that the plasmid delivery *in vivo* has been sufficient to achieve physiological levels of secreted proteins. Intramuscular injection of plasmid followed by EP has been used very successfully to deliver

**HPV-004** 

therapeutic genes that encode for a variety of hormones, cytokines or enzymes in a variety of species [Prud'homme 2006, 2007]. The design of software that enables constant current EP to deliver plasmids allows for the individual resistance of the treated muscle to be taken into consideration and yields highly efficient in vivo plasmid expression [Khan 2005].

In a small (10 healthy volunteers) pilot study, pain was evaluated immediately, 5, 15, 30 minutes and 1 hour after EP with the CELLECTRA® device [Diehl 2013]. Subjects used a Visual Analog Scale (VAS) questionnaire, 10 cm in length, anchored by word descriptors at each end, "No Pain" and "Worst Pain", to mark their pain related to the treatment. Subjects reported a mean (±sem) score of 6.3  $(\pm 0.7)$  immediately after treatment and 2.8  $(\pm 0.5)$  approximately 5 minutes after the procedure. These data showed that the pain associated with electroporation was brief and diminished quickly [Diehl 2013].

### 1.2 Plasmid DNA Immunotherapy Agents (INO-3112)

# 1.2.1 VGX-3100

Chemical name: Circular, double stranded, deoxyribonucleic acid consisting of 3782 base pairs for the pGX3001 plasmid and 3824 base pairs for the pGX3002 plasmid.

Distinguishing name: Eukaryotic expression plasmids containing HPV 16 and 18-E6 & E7-encoding transcription unit controlled by a synthetic, CMV promoter, and elements required for replication and selection in E. coli, namely a pUC origin of replication (pUC Ori) and a kanamycin resistance gene (Kan R).

# 1.2.2 INO-9012

Chemical name: Circular, double stranded, deoxyribonucleic acid consisting of 6259 base pairs for the pGX6001 (also called IL-12 DNA) plasmid.

Distinguishing name: Eukaryotic expression plasmids containing synthetic IL-12 p35 light chain and p 40 heavy chain (pGX6001) controlled by a dual promoter vector, a bGH poly A tract, bacterial origin of replication to support production of the plasmid in *E. coli*, and a kanamycin resistance gene (Kan R).

### 1.3 **Dose and Regimen Rationale**

The doses selected are based on previous human experience and preclinical data with VGX-3100 and other DNA vaccines. A total dose of 6 mg VGX-3100 DNA has been selected for this study based on the safety and immunogenicity data generated in the HPV-001 study, where 6 mg of DNA were delivered IM followed by EP, which showed trends toward higher response rates and magnitudes of IFN-y ELISpot responses in the high dose cohort compared to the low (0.6 mg) and mid-dose (2 mg) cohorts (Table 1.1) without significant safety issues [Bagarazzi, 2012].

This dose-trend was consistent with prior expectation, a feature of the finding that suggests it is a "real" effect rather than random variation. Adverse events from previous human studies with closely related DNA plasmid products have been limited to injection site pain from the injection and electroporation procedure. No unexpected or severe adverse events were observed in any of the three dose cohorts.

Table 1.1: Percent of subjects responding and average SFU/ $10^6$  PBMC in responders for each antigen by cohort in Protocol HPV-001 Interferon- $\gamma$  ELISpot

| Cohort | Lo | )W | M | lid | High | |
|--------|-----|-----|-----|-----|------|------|
| Antige | %RE | | %RE | | %RE | |
| n | SP | AVG | SP | AVG | SP | AVG |
| 16E6 | 33% | 107 | 50% | 243 | 50% | 1341 |
| 16E7 | 17% | 198 | 50% | 104 | 67% | 143 |
| 18E6 | 50% | 359 | 50% | 338 | 83% | 664 |
| 18E7 | 33% | 159 | 17% | 179 | 50% | 834 |
| Any | 67% | 221 | 67% | 210 | 83% | 556 |

The IL-12 plasmid dose is based on previous experience in the HVTN-080 study, where 1 mg was co-administered with PENNVAX®-B followed by EP. HIV-specific CD4+ T cell responses were generated in ~81% of PENNVAX®-B + IL-12 recipients after three vaccinations, compared to 44% with PENNVAX®-B alone. Delivery of PENNVAX®-B via EP also increased the frequency of CD8+ T cell responses. CD8+ responses were detected in 33% of PENNVAX®-B and 52% of PENNVAX®-B + IL-12 recipients after 3 vaccinations. Six months after the third vaccination 43% of individuals were still able to respond to HIV peptide pools. Overall, 89% of individuals vaccinated with PENNVAX®-B + IL-12 plasmid followed by EP developed either a CD4+ or CD8+ T-cell response after the third vaccination. No unexpected or severe adverse events were observed in HVTN-080 or earlier studies of IL-12 DNA delivered without electroporation.

In summary, a total of 7 mg VGX-3100 + INO-9012 DNA was selected for this study based on the safety and immunogenicity data generated in HPV-001, the follow-on study HPV-002, and HVTN-080. Additional human experience with related DNA plasmids informing the dose is described below.

# 1.3.1 Previous Human Experience with VGX-3100

The clinical experience with VGX-3100 is demonstrated in two phase 1 studies, HPV-001 and HPV-002 which enrolled 18 and 13 women, respectively, and a phase 2 study, HPV-003, which enrolled 167 women. There have been no significant safety findings with very few related Grade 3 Adverse Events (AE's) and no related Grade 4 AE's or Serious Adverse Events (SAEs) after 551 doses in 185 subjects. Importantly, the safety profile of the DNA immunogen /electroporation technology platform employed in this study has been consistently unremarkable in the 580 subjects and 1,548 doses in 16 different studies as of

February 4, 2015. (Refer to INO-3112 Investigator's Brochure v3.0 for additional information)

There were no significant safety findings in the 18 subjects enrolled in HPV-001, the phase 1 study of VGX-3100, with only mild to moderate adverse events, injection site reactions and laboratory abnormalities which resolved without sequelae. All subjects returned home after at least 30 minutes observation in the study unit post injection/EP. CPK and ECGs were unremarkable post electroporation. Study participants judged the injection/EP to be relatively painful (mean VAS score 6.2 immediately after and 2.8 approximately 5 minutes after EP) but transient, but did not preclude subsequent injection/EP administration. There were no serious adverse events attributed to treatment in any of the subjects and there were no early discontinuations in the study. Thirteen women participated in HPV-002 in which a fourth dose (6 mg only) of VGX-3100 was evaluated and the safety findings were consistent with those observed in the parent study, HPV-001.

The clinical trial experience in HPV-003 with the investigational product to date is consistent with those reported previously. No new safety issues have been identified with VGX-3100 delivered IM followed by EP with CELLECTRA®-5P, and no serious unexpected drug related adverse events, or other events requiring expedited reporting, have been reported for subjects dosed with VGX-3100 delivered IM followed by EP with CELLECTRA®-5P.

The mechanism of action of VGX-3100 delivered using EP is expected to be mediated through a Th1-biased cytolytic T-cell response against the HPV16 and HPV18 E6 and E7 proteins. Strong antigen-specific T-cell immune responses were observed in not only the phase 1 HPV studies but also in the previous studies using the same technology with different antigens for several disease indications (e.g. influenza, HIV) [Bagarazzi 2012]. The cellular immunity has also been demonstrated to be durable up to 25 months from the initiation of therapy [unpublished data]; strongly suggesting the development of long term memory cells in the immunized volunteers. In addition, the antigen-specific T-cells have been shown to exhibit a memory phenotype by flow cytometry [Bagarazzi 2012]. Immunoglobulin G-based antibodies have also been measured in a high percentage (>90%) of immunized volunteers in the previous human studies with this technology [Bagarazzi 2012, unpublished data].

# Ongoing study of VGX-3100 in subjects with for high grade CIN associated with HPV-16 and/or HPV-18 (HPV-003)

All current therapeutic options for cervical dysplasia are destructive, have adverse sequelae, and furthermore are not always curative. Among treated high grade CIN in immunocompetent women, the overall risk of recurrence is less than ten percent when all surgical margins are clear, but increases to approximately 25% in women with positive margins. About 90% of recurrences will occur within the first year after treatment [Felix 1994]. Moreover, tissue destruction from therapeutic interventions can make subsequent detection and treatment of recurrent disease difficult, as the healing process draws the transition zone of the

cervical epithelium proximally, into the endocervical canal [Ferris 1995]. Effective immunotherapy would obviate the need for surgery, to say nothing of preventing progression to cervical cancer. Consequently, a placebo-controlled phase 2 study is under way to determine if VGX-3100 delivered by EP will result in immune-mediated regression of high grade cervical dysplasia when administered prior to surgical intervention. The study, known as HPV-003 will evaluate histologic regression 6 months after completion of the three dose series. A pre-planned interim analysis of the study data completed in July 2014 revealed that the study met its primary endpoint (histopathologic regression of lesions) and secondary endpoint (histopathologic regression of lesions in the context of elimination of HPV16 and/or 18 infection) demonstrating a highly statistically significant improvement in the VGX-3100 arm (p<0.017 and p<0.001 respectively). Treatment of HPV16 and/or 18 positive patients with CIN2 or 3 was generally safe as evidenced by the lack of statistical significance between the frequencies of adverse events reported in the placebo arm as compared to the VGX-3100 treated arm. Treatment with VGX-3100 was able to induce a robust immune response in the periphery as gauged by IFNy ELISpot as well as in the tissue as examined using immunohistochemistry. These data reveal the highly promising potential of therapeutic immunization with DNA followed by electroporation for the treatment of HPV-16 and/or HPV-18 related precancerous cervical disease in women.

A logical next step is to determine if INO-3112 delivered by EP could also provide clinical benefit for patients with invasive squamous cell carcinoma of the cervix. In this setting, the DNA immunogen/EP platform would need to generate HPV-specific immune responses to help eliminate residual neoplastic cells after standard therapy. This study is designed to assess potential toxicity and secondarily immune responses to specific antigens in both blood and locally in the cervix, and whether the immune responses are associated with subsequent regression of neoplastic cells.

# 1.3.2 Previous Human Experience with INO-9012

The safety profile associated with IM administration of IL-12 plasmid DNA alone or followed by EP has been acceptable in clinical studies. Clinical results from three different studies substantiate the safety and tolerability profile of IL-12 plasmid DNA. IL-12 plasmid DNA has been used in several cohorts in the following four phase I clinical protocols.

| Protocol # | Co-administered with | # subjects received IL-12 DNA |
|------------|----------------------------|-------------------------------|
| HVTN-060 | HIV-1 gag p37 | 80 |
| HVTN-063 | HIV-1 gag p37 | 30 |
| HVTN-070 | PENNVAX®-B (gag, pol, env) | 30 |

| HVTN-080 | PENNVAX®-B (gag, pol, env) | 30 |
|----------|----------------------------|----|
|----------|----------------------------|----|

IL-12 DNA was delivered without EP in HVTN-060, -063 and -070 but was followed by EP in HVTN-080. In this protocol, PENNVAX®-B or placebo were delivered via IM injection followed by electroporation with the CELLECTRA®-5P device in 48 healthy volunteers. The regimen consisted of 3 mg of PENNVAX®-B with or without plasmid encoding IL-12 at months 0, 1 and 3. This study established that a highly engineered DNA vaccine delivered intramuscularly followed by EP can induce frequent and robust T-cell responses in humans.

In summary of above clinical studies, no pattern of systemic AEs emerged, and no SAEs related to the study products were observed. The plasmid DNA vaccine co-administered with IL-12 plasmid DNA as a cytokine adjuvant were well-tolerated. (See Section 5 of the INO-3112 IB for details for HVTN-080 study)

# 1.4 Risks/Benefit Assessment

# 1.4.1 Current Therapy for Stage IB-IVB Cervical Cancer

All current therapeutic options for cervical cancer involve either surgery with or without adjuvant chemotherapy and/or radiation therapy, or definitive radiation therapy, or definitive chemoradiation. Current outcomes with either radical surgery or standard chemoradiation for invasive cervical cancer results in cure rates of approximately 80 to 95 percent in early stage disease (stage I and non-bulky stage II disease) and approximately 40 to 60 percent for bulky stage II and stage III disease [Quinn 2006].

Table 1.3: Survival by FIGO stage for patients with cervical cancer: 1999 to 2001 FIGO statistics

| | # of | Overall survival, % | | |
|------------|----------|---------------------|---------|---------|
| FIGO stage | patients | 1 year | 2 years | 5 years |
| IA1 | 829 | 99.8 | 99.5 | 97.5 |
| IA2 | 275 | 98.5 | 96.9 | 94.8 |
| IB1 | 3020 | 98.2 | 95 | 89.1 |
| IB2 | 1090 | 95.8 | 88.3 | 75.7 |
| IIA | 1007 | 96.1 | 88.3 | 73.4 |
| IIB | 2510 | 91.7 | 79.8 | 65.8 |
| IIIA | 211 | 76.7 | 59.8 | 39.7 |
| IIIB | 2028 | 77.9 | 59.5 | 41.5 |
| IVA | 326 | 51.9 | 35.1 | 22 |
| IVB | 343 | 42.2 | 22.7 | 9.3 |

Original table modified for this publication. From: Quinn MA, Benedet JL, Odicino F, et al. Carcinoma of the cervix uteri. Int J Gynaecol Obstet 2006; 95:S43.

Recurrence rate by stage is as follows: for FIGO stage IB around 10%, for stage IIA 17%, for stage IIB 23%, and for stages III and IVA 42% and 74% respectively [Perez 1992].

For early stage disease, the predominant site of disease recurrences is local (*i.e.* at the vaginal apex) or regional (*i.e.* pelvic sidewall). The risk of persistent or recurrent pelvic disease increases with more advanced initial disease stage [Morely 1976, Hopkins 1991, Estape 1998].

The most frequent distant sites of recurrence are the para-aortic lymph nodes (81%), lungs (21%), and supraclavicular lymph nodes (7%), whose incidence relates to the stage of disease: it is 0–3% in stage IA, 13–16% in stage IB, 22–31% in stage IIA, 22–26% in stage IIB, 32–39% in stage III and 75% in stage IVA [Perez 1995].

The outcomes for inoperable cervical cancer have improved with the use of concurrent chemotherapy during radiation and this multi-modality approach is now standard of care [Rose 1999, Morris 1999, Grigsby 2001]. However, as noted above, recurrence rates are significant and impact not only survival but also quality of life.

Clearly, there is room to decrease recurrence rates at all stages of disease and additional investigations are warranted to further improve outcomes for this population.

# 1.4.2 Rationale for Study Design

There are data in patients with pre-invasive lesions that demonstrate the safety of immune-based therapy in immune-competent patients.

In otherwise healthy women whose CIN 2/3 lesions had already been resected, treatment with VGX-3100 delivered by EP stimulated both antibody and T-cell responses that were detectable in over 80% of subjects, without significant side effects. The potential benefit of taking part in this study is that INO-3112 could stimulate the immune system to eliminate residual neoplastic cells after standard therapy. This study is designed to assess primarily toxicity of treatment with INO-3112 delivered by EP after such standard therapy and secondarily, immune responses to the HPV antigens encoded by VGX-3100 in both peripheral blood and locally in the cervix.

Subjects enrolled in this protocol will undergo close clinical surveillance by experienced gynecologic oncologist, radiation oncologists and oncologists. Participants will be seen at screening to determine eligibility. Two cohorts will be enrolled.

In Cohort 1, prior to dosing, all subjects will have undergone standard external beam radiation therapy administered concurrently with cisplatin over 5 to 6 weeks, followed by brachytherapy and then a brief rest period (2 weeks or less) prior to the study treatment/EP (Day 0) regimen with INO-3112. The first study treatment/EP treatment (Day 0) will be administered within two weeks of completion of chemoradiation, the second study treatment/EP at Week 4

following Day 0, the third at Week 8 and the fourth (final) treatment will be administered at Week 12 following Day 0.

In cohort 2, subjects with persistent and/or recurrent disease will be treated with study treatment/EP following salvage therapy. The first study treatment/EP treatment (Day 0) will be administered no earlier than 2 weeks after completing salvage therapy, the second study treatment/EP at Week 4 following Day 0, the third at Week 8 and the fourth (final) treatment will be administered at Week 12 following Day 0.

Participants will be followed as part of this study for 6 months after the last study treatment/EP (i.e. Week 12) with INO-3112.

Radiation therapy has been shown to induce a variety of immune effects within the radiation field, including up regulation of major histocompatibility complex class I (MHC-I) expression and increased activation of CD8+ cytotoxic T lymphocytes (CTL) [Nikitina 2001]. Changes in cytokine and adhesion molecule expression facilitate homing of antigen-presenting cells and effector immune cells to the induced area [Hong 1995, Hong 1999, Hallahan 1996, Tanigawa 2001]. Decreases in CD4+ CD25+ regulatory T cells and myeloid-derived suppressor cells (MDSC) have also been noted, which leads to a more robust immune response in the irradiated area [Sutmuller 2001]. Apoptotic and necrotic tumor cells within the radiation field provide sources of antigens for dendritic cells, which in turn activate T cell maturation [Rock 2005]. The dying cells also release "danger factors" which can act as immunologic adjuvants to prevent immune tolerance to tumor antigens [Matzinger 1994, Galucci 1999, Shi 2002].

Studies revealed that radiation induces up regulation of death receptors, particularly Fas, in tumor cells, which further sensitizes them to the killing action of CTL [Sheard 1997, Chakraborty 2002, Garnett 2004]. Fractionated radiotherapy is hypothesized to impair the immune response due to deleterious effects on infiltrating immune cells whereas hypo-fractionated ablative dosing resulted in a superior immune response [Lee 2009]. Thus, concurrent vaccination at the end of brachytherapy may have a similarly activating effect on the local immune system. Previous murine studies have shown that radiation can heighten the immune response to vaccination against HPV oncogenes E6 and E7, and post-radiation vaccination with a recombinant HPV E6/E7 vector results in a significant increase in long-term survival due to cell-mediated killing [Tseng 2009].

Delivering the vaccine immediately after the conclusion of brachytherapy to harness the immunologic priming effects of radiation and complement the in situ immunization may initiate a sustained adaptive immune response against the E6 and E7-expressing tumor cells.

Monitoring will include HPV typing at screening/entry. Tumor biopsy, ThinPrep<sup>TM</sup> samples for HPV testing and cytology, and Digene swabs will be collected at screening (pre or post-chemoradiation), Day 0 and at Week 16 (one month post-dose 4) and week 36. Physical exam, vital signs, ECOG performance status and laboratory evaluations will be performed at screening and prior to first

study treatment/EP on Day 0 and at specified visits throughout the study. Imaging with PET/CT scans will be performed within 4 weeks prior to Day 0 (baseline) and 3-4 months after Day 0 and 3-5 month thereafter or at study discharge per standard of care or in accordance with local guidelines and institutional practices. Investigators will be instructed to use their clinical judgment throughout the study.

# 1.4.3 Potential Risks of DNA Immunotherapy Delivery with Electroporation

The underlying basis for all studies of plasmid DNA vaccines is the fairly substantial safety database that exists for the varied plasmid DNA vaccine candidates that have now been studied in both animals and humans. The plasmid DNA platform has been utilized for vaccine candidates for a variety of disease indications and infectious agents (*e.g.*, HIV, HPV, Influenza, SARS, West Nile virus, Ebola among others) in addition to plasmid cytokine adjuvants such as IL-2, IL-12 and IL-15.

In two companion papers by Sheets *et. al*, potential toxicities (both intrinsic and immunotoxicities) and biodistribution profiles were compared for 21 different plasmid DNA constructs, in 9 separate GLP-compliant studies [Sheets 2006a, 2006b]. Despite differing plasmid DNA backbones, promoters, and sequence inserts, toxicity and biodistribution profiles were similar for all plasmid DNA constructs. With respect to the toxicity assessments, the authors reported that toxicity was localized to the site of the injection for all 21 plasmid DNA constructs. Similarly, all plasmid DNA constructs evaluated showed evidence to be localized to the injection site and surrounding tissue in all studies. Based on the results of these GLP toxicology and biodistribution studies, Sheets et. al post a case for "refinements of preclinical safety protocols over time" as it pertains to the development pathway for plasmid DNA vaccine candidates [Sheets 2006a, 2006b].

Further, four separate GLP toxicology and biodistribution studies have been performed for eight additional plasmid DNA vaccine candidates developed by Inovio with identical backbones delivered by electroporation yielding similar toxicity and biodistribution profiles. Intramuscular co-administration of IL-12 plasmid was evaluated in nonclinical studies to support the studies of intramuscular IL-12 plasmid in humans.

DNA vaccines developed by Inovio have been delivered without electroporation (1 study) or using Inovio electroporation devices (11 studies) as shown in Table 1.4. Inovio electroporation devices have also been used to deliver DNA vaccines developed outside of Inovio in three different studies and two studies have evaluated the tolerability of Inovio electroporation devices with normal saline.

Based on clinical experience with INO-3112 from similar protocols using electroporation-mediated drug delivery and the overall safety database encompassing all studies of Inovio DNA delivered by electroporation with CELLECTRA®-5P, we do not expect to observe any severe or dose-limiting side

effects or toxicities. Side effects of vaccination with INO-3112 may include discomfort related to the electroporation technique, such as transient local edema, swelling, or pain.

In the phase I studies of VGX-3100 delivered by EP in women with a history of treated CIN 2/3 there were no serious adverse events attributed to treatment in any of the subjects enrolled and no participants discontinued early.

# 2 HYPOTHESIS AND STUDY OBJECTIVES

# 2.1 Hypothesis

Immunotherapy with INO-3112 delivered by IM injection followed by EP with CELLECTRA®-5P will be immunogenic and well tolerated in women with newly diagnosed, inoperable cervical cancer associated with HPV-16 and/or HPV-18 after completion of standard chemoradiation therapy with curative intent (Cohort 1) or in women with persistent and/or recurrent cervical cancer associated with HPV-16 and/or HPV-18 following salvage therapy (Cohort 2) and will not be associated with any significant increased toxicity compared to that expected/reported with "standard" therapy alone.

# 2.2 Primary Objective

Evaluate the safety and tolerability of immunotherapy with INO-3112 when delivered IM followed by EP with CELLECTRA®-5P in women with newly diagnosed, inoperable cervical cancer associated with HPV-16 and/or HPV-18 after completion of standard chemoradiation therapy with curative intent (Cohort 1) or in women with persistent and/or recurrent cervical cancer associated with HPV-16 and/or HPV-18 following salvage therapy (Cohort 2) compared to that expected/reported with "standard" therapy alone.

# 2.3 Secondary Objective

Evaluate the cellular and humoral immune responses to immunotherapy with INO-3112 delivered IM followed by EP with CELLECTRA®-5P in women with newly diagnosed, inoperable cervical cancer associated with HPV-16 and/or HPV-18 after completion of standard chemoradiation therapy with curative intent (Cohort 1) or in women with persistent and/or recurrent cervical cancer associated with HPV-16 and/or HPV-18 following salvage therapy (Cohort 2).

# 2.4 Exploratory Objective

Evaluate clinical response (i.e. disease-free survival) following treatment with INO-3112 delivered IM followed by EP with CELLECTRA®-5P in women with newly diagnosed, inoperable cervical cancer associated with HPV-16 and/or HPV-18 after completion of standard chemoradiation therapy with curative intent (Cohort 1) or in women with persistent and/or recurrent cervical cancer associated with HPV-16 and/or HPV-18 following salvage therapy (Cohort 2).

# 3 STUDY DESIGN

This is a Phase I/IIa, open-label study to evaluate the safety, tolerability, and immunogenicity of INO-3112 [6 mg of VGX-3100 (2 separate DNA plasmids encoding E6 and E7 proteins of HPV 16 and HPV 18) and 1 mg of INO-9012 (DNA plasmid encoding human interleukin 12)] delivered IM followed by EP in approximately 10 female subjects with biopsy-proven, Stage IB-IVB inoperable invasive cervical carcinoma associated HPV-16 and/or HPV-18 who have completed treatment with standard chemoradiation with curative intent (Cohort 1) or in subjects with persistent and/or recurrent cervical cancer associated with HPV-16 and/or HPV-18 following salvage therapy (Cohort 2).

Eligible subjects who consent to participate in the study will receive a 1.1 mL IM injection of INO-3112 in the deltoid followed immediately by EP with CELLECTRA®-5P. If the deltoid is not a suitable location, the IM injection should be in the lateral quadriceps followed immediately by EP with CELLECTRA®-5P. All subjects (Cohorts 1 and 2) will receive a 4-dose series of INO-3112. The first study treatment/EP after completion of standard chemoradiation (Cohort 1) or salvage therapy (Cohort 2) will be designated as "Day 0", the second dose will be administered at Week 4, the third dose at Week 8, and the fourth (final) treatment will be administered at Week 12.

# **Cohort 1:**

Cohort 1 will include subjects with biopsy-proven, Stage IB-IVB inoperable, newly diagnosed invasive cervical carcinoma associated with HPV-16 and/or HPV-18 treated with standard chemoradiation therapy with curative intent.

All subjects in Cohort 1 must receive their initial study treatment (Day 0) within 2 weeks after completing a course of standard radiation therapy (external beam and brachytherapy) administered concurrently with platinum based therapy with curative intent.

Subjects will have received standard external beam radiation therapy administered concurrently with cisplatin at 40 mg/m²/week followed by their brachytherapy prior to the study treatment with INO-3112. The chemoradiation must be completed within 10 weeks of initiation. Standard external beam radiation therapy should be delivered to the pelvis +/- para-aortic nodal chain to a total dose of 45 Gy in 25 fractions, in conjunction with high dose rate (HDR) or low dose rate (LDR) brachytherapy to the cervix to deliver a total dose of 80-90 Gy (LDR equivalent) to point A. Parametrial and nodal boost should be delivered as determined by the disease stage per sequencing outlined in Appendix 3, such that brachytherapy will be the last treatment administered.

Weekly cisplatin chemotherapy at 40 mg/m<sup>2</sup> should be administered during Weeks 1-5 of standard external beam radiation and during parametrial boost.

# Cohort 2:

Cohort 2 will include subjects with persistent and/or recurrent cervical carcinoma associated with HPV-16 and/or HPV-18 who have been treated with salvage therapy (chemotherapy and/or radiation therapy).

All subjects in Cohort 2 must receive their initial study treatment (Day 0) no sooner than 2 weeks and no later than 4 weeks after completing a course of salvage therapy. If in the investigators opinion, there are no additional salvage therapy options, the subject may be enrolled in Cohort 2 without having received salvage therapy immediately prior to enrollment.

# **Primary Safety Endpoints:**

- 1. Incidence of adverse events (all, severe [graded per CTCAE v4.03], unexpected, serious) classified by system organ class (SOC), preferred term, severity, and relationship to study medication and schedule
- 2. Injection site reactions including pain, tenderness, erythema and induration at administration site
- 3. Rates of acute gastrointestinal, genitourinary, or other chemoradiation side effects above the expected, graded per Acute Radiation Morbidity Scoring Criteria (RTOG)
- 4. Changes in laboratory parameters from baseline

# **Secondary Immunologic Endpoints:**

- 1. Antigen-specific cellular immune responses to INO-3112 in blood samples obtained from study subjects per study schedule:
  - a) Interferon-y secreting T lymphocytes in PBMC by ELISpot
  - b) Flow Cytometry for T-cell activation, cytolytic phenotype, and memory phenotype in PBMC
- 2. Antigen-specific humoral responses to HPV-E6 and -E7 by ELISA per study schedule

# **Exploratory Clinical Endpoints:**

- 1. Changes in standard uptake volume (SUV) on PET/CT scans performed at baseline vs follow-up PET/CT scans obtained at specified time points.
- 2. Evaluation of subjects relative immune competence longitudinally throughout the study starting at the screening visit (for details refer to Section 6.7: Cervical Virologic and Peripheral Blood Immunogenicity Assessment)
- 3. Changes in cervical histology from the screening biopsy as compared to the week 16 biopsy
- 4. Local immune responses to INO-3112 in tumor tissue samples obtained at week 16
- 5. Disease-free survival assessed in accordance with RECIST v1.1 (Refer to Appendix 10) as follows:
  - Clinical evaluations for disease response will be conducted at all study visits, (as assessed by clinical signs and symptoms of disease progression).

• A baseline PET/CT scan will be obtained on each subject 1 to 2 weeks prior to Day 0 and then PET/CT scans for disease progression will be obtained for all subjects 3-4 months after Day 0 and every 3-5 months thereafter per standard of care/in accordance with local guidelines and institutional practices. Additional PET/CT scans may be obtained at other time points if clinically indicated to confirm a clinical diagnosis of disease progression based on signs and symptoms.

# 4 SELECTION AND ENROLLMENT OF SUBJECTS

# 4.1 Inclusion Criteria

- a) Written informed consent in accordance with institutional guidelines. If required by local law, candidates must also authorize the release and use of protected health information (PHI);
- b) Female subjects age 18 years or older;
- c) Histological diagnosis of squamous cell carcinoma, adenocarcinoma or adenosquamous cell carcinoma of the cervix. Not accepted are small cell, clear cell and other rare variants of the classical adenocarcinoma;
- d) Histologically confirmed, Stage IB-IVB, invasive cervical carcinoma associated with HPV-16 and/or HPV-18 and meeting the following eligibility criteria for either Cohort 1 or Cohort 2;

# 1. Cohort 1

- Newly diagnosed inoperable cervical cancer treated with chemoradiation therapy with curative intent and life expectancy of at least 12 months as assessed by the investigator
  - No CNS/spinal metastases
- Able to initiate study treatment (Day 0) within 2 weeks of completion of last chemoradiation treatment;
  - Platinum based treatment (alone or in combination with other drugs); 5 weekly courses of Cisplatin 40 mg/m² completed within 10 weeks of its initiation
  - Standard radiation therapy (external beam and brachytherapy);
     completed within 10 weeks of its initiation
  - o Brachytherapy; must be the last treatment if the subject is receiving sequential brachytherapy following the chemoradiation therapy

# 2. Cohort 2

- Persistent and/or recurrent cervical cancer
  - o No CNS/spinal metastases
- Able to initiate study treatment (Day 0) at least 2 weeks but no more than 4 weeks after completion of salvage therapy (If in the investigators opinion, there are no additional salvage therapy options, the subject may be enrolled in Cohort 2 without having received salvage therapy immediately prior to enrollment.)
- Subject has a life expectancy of at least 12 months as assessed by the investigator

- e) ECG with no clinically significant findings as assessed by the investigator performed within 30 days of signing the informed consent form (ICF);
- f) Chemistry, liver function tests, renal function, total CPK and hematology lab results must be ≤ Grade 1 at the time of screening, in accordance with the CTCAE v4.03;
- g) Eastern Cooperative Oncology Group (ECOG) Performance status of  $\leq 1$ ;
- h) Adequate venous access for repeated blood sampling according to study schedule;
- i) Women of child-bearing potential must have a negative serum pregnancy test and agree to remain sexually abstinent, have a partner who is sterile (i.e., vasectomy), or use two medically effective methods of contraception (e.g., oral contraception, barrier methods, spermicide, intrauterine device (IUD)). This requirement should be followed from screening through 24 weeks after last study treatment/EP. Whole pelvis external beam radiation therapy (EBRT) followed by intracavitary (IC) therapy for cervical cancer is considered to be an irreversible form of contraception;
- j) Able and willing to comply with all study procedures.

# 4.2 Exclusion Criteria

- a) Pregnancy or breastfeeding;
- b) History of previous therapeutic HPV vaccination (individuals who have been immunized with licensed prophylactic HPV vaccines (e.g. Gardasil®, Cervarix®) are not excluded);
- c) Prior exposure to an investigational agent or device within 30 days of signing the ICF. Of note, the subject may participate in observational studies:
- d) Positive serological test for human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C or history of HIV infection, Hepatitis B or Hepatitis C (women with cured HCV will be allowed; subject must have had an serologic test performed within 12 months of informed consent);
- e) Prior major surgery within 4 weeks of first study treatment/EP from which the subject has not yet recovered to baseline;
- f) High medical risks because of non-malignant systemic disease or with active uncontrolled infection;
- g) Current malignancies at other sites, with the exception of adequately treated basal or squamous cell carcinoma of the skin;
  - -Cancer survivors, who have undergone curative therapy for a prior malignancy, have no evidence of that disease for five years and are deemed at low risk for recurrence, are eligible for the study;
- h) Congestive heart failure or prior history of New York Heart Association (NYHA) class III/ IV cardiac disease (refer to Appendix 8);
- i) Any concurrent condition requiring the continued use of systemic or topical steroids at or near the injection site, excluding non-systemic (e.g. inhaled and eye drop-containing) corticosteroids or the use of other immunosuppressive agents. All other corticosteroids must be discontinued > 4 weeks prior to Day 0 of study product administration;
- j) Any cardiac pre-excitation syndromes (such as Wolff-Parkinson-White);

- k) History of seizures (unless seizure free for 5 years);
- Less than two acceptable sites exist for IM injection and EP between use of the deltoid and lateral quadriceps muscles. A site for injection/EP is not acceptable if there are tattoos or scars within 2 cm of the injection/EP site or if there is implanted metal within the same limb. Any device implanted in the chest (e.g., cardiac pacemaker or defibrillator) excludes the use of the deltoid muscle on the same side of the body;
- m) Administration of any non-study related vaccine within 2 weeks of Day 0;
- n) Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements;
- o) Imprisonment or compulsory detainment (involuntary incarceration) for treatment of either a psychiatric or physical (i.e. infectious disease) illness;
- p) History of immunosuppressive or autoimmune disease;
- q) Any other illnesses or conditions that in the opinion of the investigator may affect the safety of the subject or limit the evaluation of a subject or any study endpoint.

# 4.3 Supplementation of Study Subjects

Additional subjects may be enrolled with the approval of medical monitor, if subjects withdraw prior to completion of the study treatment.

# 4.4 Discontinuation/Withdrawal of Study Subjects

The subject will be considered to have completed the study when she completes all scheduled Study Treatments and follow-up visits or death, whichever occurs first. The discharge visit will be the last follow-up visit. If subject discontinues or is withdrawn at any time after receipt of Study Treatment, the investigator should make every effort to have the subject complete all assessments designated for the discharge visit. The investigator will make every effort to have all scheduled immune assessment blood sample collected as indicated in the Schedule of Events, Table 1 of the Clinical Synopsis. Any adverse events (AEs) present at the time of discontinuation/withdrawal should be followed in accordance with the safety requirements outlined in Section 7.1 – Safety Parameters.

If the subject manifests Grade 4 toxicity attributable to study treatment/EP, she will not receive further study treatment/EP but will be encouraged to continue follow-up safety assessment through study discharge and not discontinue from the study. If a subject manifests Grade 3 toxicity attributable to study treatment/EP, the medical monitor and PI will discuss whether further treatment should be continued for that participant.

Subjects will be discontinued from the study if there is confirmed disease progression or if subject starts new anti-cancer therapy.

The reason for any discontinuation of study treatment should be discussed with the Sponsor's Medical Monitor within 24 hours. The primary reason for the subject discontinuing further study treatments or withdrawal from the study itself should be selected from the following standard categories:

- Adverse Event (Adverse Reaction): Clinical or laboratory events occurred that, in the medical judgment of the investigator for the best interest of the subject, are grounds for discontinuation. This includes serious and non-serious adverse events regardless of relation to study treatment.
- Death: The subject died.
- Withdrawal of Consent: The subject desired to withdraw from further participation in the study in the absence of an investigator-determined medical need to withdraw. If the subject gave a reason for withdrawal, it should be recorded on the Case Report Form (CRF). This reason does not allow for further data collection and should not be selected if follow-up data collection of this subject is anticipated by the subject.
- Protocol Violation: The subject's findings or conduct failed to meet the
  protocol entry criteria or failed to adhere to the protocol requirements
  (e.g., treatment noncompliance, failure to return for defined number of
  visits). The violation should be discussed with the Sponsor's Medical
  Monitor prior to discontinuation of Study Treatments or study withdrawal.
- Lost to Follow-up: The subject fails to attend study visits and study personnel are unable to contact the subject after repeated attempts including letter sent by certified mail or equivalent.
- Physician Decision: The subject was terminated for a reason other than those listed above by the physician caring for the subject.
- Other: The subject was terminated for a reason other than those listed above, such as termination of study by the Sponsor.

# 5 INVESTIGATIONAL PRODUCTS

# 5.1 Investigational Product

Investigational product is defined as a pharmaceutical form of an active ingredient being tested or used as a reference in the study, whether blinded or unblinded.

INO-3112 is combination of VGX-3100 and INO-9012.

VGX-3100, the active investigational product to be used in this study, is a mixture of two separate DNA plasmids encoding E6 and E7 proteins of HPV types 16 and 18. A second investigational product being evaluated for use in combination with VGX-3100 is known as INO-9012. INO-9012 is a DNA plasmid expressing the p35 and p40 human IL-12 subunits off of separate promoters within the same plasmid.

INO-3112 will be provided by Inovio or its designee. The site pharmacist or designee will combine VGX-3100 and INO-9012 into a single syringe to create a 1.1 mL IM formulation of INO-3112 (see Appendix 6 for details).

**Table 5.1 Investigational Products** 

| VGX-3100 | The plasmid pGX3001 and pGX3002 |
|----------------------|---------------------------------|
| Volume per container | 1.0 mL minimum/vial |
| Concentration | $6.0 \pm 0.4 \text{ mg/mL}$ | |
|-------------------------|------------------------------|--|
| Container Size and Type | 10 mL glass vial | |
| INO-9012 | The plasmid pGX6001 | |
| Volume per container | 0.2 mL minimum/vial | |
| Target Concentration | $10.0 \pm 0.5 \text{ mg/ml}$ | |
| Container Size and Type | 2 mL glass vial | |

## 5.2 Packaging and Labeling

This study is open label. Therefore the subject, the Investigator's site personnel and the Sponsor are not blinded to treatment. Each vial will be labeled with a single panel label. The following shows text that may be included on the vial labels:

| Biologic<br>Product | Specimen Label |
|---|---|
| VGX-3100 | SynCon <sup>TM</sup> VGX-3100 [6mg/mL] 1 mL/vial Lot: VGX-3100. xxxxxx Date of Manufacture: DD MMM YY Final Retest Date: DD MMM YY Store frozen at or below -15C CAUTION: New Drug – Limited by Federal Law to Clinical Trial Use Only Inovio Pharmaceuticals Inc 660 W Germantown Pike, Plymouth Meeting, PA 19462 USA |
| INO-9012 | SynCon <sup>TM</sup> INO-9012 [10 mg/mL] 0.2 mL/vial Single Use Vial Lot: INO-9012.xxxxxx Date of Manufacture: DD MMM YY Final Retest Date: DD MMM YY Store frozen at or below -15°C CAUTION: New Drug – Limited by Federal Law to Investigational Use. Inovio Pharmaceuticals Inc. Rev 000 |

## 5.3 Handling of INO-3112

Inovio will be responsible for assuring that the quality of the investigational products is adequate for the duration of the trial. All study products will be shipped frozen on dry ice. If there is no dry ice remaining in the shipment container when the shipment is received, the Sponsor or designee should be contacted immediately.

In addition, a temperature monitor will track the temperature of vials and will indicate any excursions during shipment to the site.

Investigational product(s) should be stored in a secure area according to local regulations. Vials must be stored at -20 °C upon receipt at the clinical site. The Sponsor should be notified of any deviations from this recommended storage condition.

A freezer temperature log must be monitored daily and maintained at the site.

## 5.4 Dispensing of INO-3112

It is the responsibility of the Investigator to ensure that INO-3112 is dispensed to study participants. It must be dispensed only from official study sites by authorized personnel according to local regulations and must be recorded appropriately on the investigational product accountability record.

Vial contents must be thawed at ambient room temperature and must be administered within 4 hours of removal from freezer.

VGX-3100 and INO-9012 will be combined by the site pharmacist into a single syringe for subjects using the procedure outlined in Appendix 6.

The syringe must be labeled with the date and time it was removed from the freezer and a four-hour expiration date and time from the time the vial is removed from the freezer. The label should also contain the words "administer as soon as possible".

## 5.5 Records of INO-3112 Disposition at Investigational Sites

It is the responsibility of the Investigator to ensure that a current record of investigational product disposition is maintained at each study site where investigational product is inventoried and disposed. Records or logs must comply with applicable regulations and guidelines, and should include:

- Amount received and placed in storage area;
- Amount currently in storage area;
- Label ID number or batch number and use date or expiry date;
- Dates and initials of person responsible for each investigational product inventory entry/movement;
- Amount dispensed to each subject, including unique subject identifiers;
- Amount transferred to another area/site for dispensing or storage;
- Amount returned to Sponsor;
- Amount destroyed at study site, if applicable.

#### 5.6 Return and Destruction of Investigational Products

Upon completion or termination of the study, all unused and/or partially used investigational product must be returned to Inovio, if not authorized by Inovio or local regulations to be destroyed at the site.

All investigational products returned to Inovio must be accompanied by the appropriate documentation. Returned supplies should be in the original containers. Empty containers should be retained until final reconciliation performed by the Study Monitor, but not be returned to Inovio. It is the Investigator's responsibility to arrange for disposal of all empty containers,

provided that procedures for proper disposal have been established according to applicable federal, state, local and institutional guidelines and procedures, and provided that appropriate records of disposal are kept. The return of unused investigational product(s) should be arranged by the responsible Study Monitor.

If investigational products are to be destroyed on site, it is the Investigator's responsibility to ensure that arrangements have been made for the disposal, written authorization has been granted by Inovio, procedures for proper disposal have been established according to applicable regulation and guidelines and institutional procedures, and appropriate records of the disposal have been documented. The unused investigational products can only be destroyed after being inspected and reconciled by the responsible Inovio Study Monitor.

## 5.7 Use of CELLECTRA®-5P Electroporation Device

The instructions for use of the CELLECTRA®-5P device are located in the Operations Manual. Each clinical site will receive training for the use of the CELLECTRA®-5P device. The following specifications will be used during the study:

Number of pulses = 3 Current Strength = 0.5 Amp Electroporation pulse duration = 52 milliseconds/pulse Interval separating pulses = 1 second

The <u>injection/electroporation procedure</u> must be performed by qualified personnel. Any individual designated to perform the procedure should be permitted by the relevant local authorities to administer parenteral medications to patients (e.g. MD, DO, RN) in addition to receiving device training from sponsor personnel. Individuals whose credentials do not meet the relevant local requirements may perform the injection/electroporation procedure under the conditions below:

- 1. The procedure must be performed under the direct supervision of the Principal Investigator or an approved Sub-Investigator who has already been trained by sponsor personnel.
- 2. The CV and any relevant qualifications of the individual have been reviewed and approved by the sponsor or its designee to perform the procedure.

Any deviation from the above procedures must be approved by the sponsor or its designee.

## 5.8 Investigational Device Accountability

Each clinical site is responsible for maintaining investigational device accountability. This includes recording the CELLECTRA®-5P serial number, IM applicator serial number, and IM array lot number used for injection/EP of each

subject. Site personnel will be required to download electroporation data and provide to Inovio after each treatment.

### 6 STUDY PROCEDURES AND TREATMENTS

See **Table 1** for Schedule of Events showing study procedures and the times at which they are to be carried out.

## 6.1 Procedure by Visit

### **6.1.1 Screening Evaluations**

Subjects who consent to participate in the study will be eligible for screening and will have a tumor biopsy sample (i.e. unstained slides) sent to laboratory for HPV assessment that will done either by ISH or PCR. If a subject has documented evidence of HPV-16 and/or HPV-18 infection results from cervical specimen obtained prior to anti-cancer treatment, then those results will be acceptable. If applicable, ThinPrep<sup>TM</sup> sample should also be sent simultaneously to the central lab for HPV assessment by PCR. Another cervical biopsy should be collected at screening if residual tissue is not available for additional assessment. The screening assessments, if required may be done in two parts. The first part will consist of consenting the subject and collecting cervical biopsy samples for HPV assessment. The second part of the visit will consist of performing the remaining screening assessment.

Subjects in Cohort 1 can be screened either prior to initiation of chemoradiation or during chemoradiation. Subjects should be screened and enrolled such that their first study treatment (Day 0) will be delivered within 2 weeks of completing their chemoradiation therapy.

Subjects in Cohort 2 can be screened at any time prior to the date of their first study treatment. Subjects should be screened and enrolled such that their first study treatment (Day 0) is no sooner than 2 weeks and no later than 4 weeks after completing the salvage therapy.

The following evaluations will be performed at **screening** visit prior to Day 0:

- Signed informed consent
- o Histologic diagnosis of cervical cancer
- Collect demographic information
- o Determination of eligibility per inclusion and exclusion criteria
- Medical and CIN/cancer history
- Medical/clinical assessment
- o Adverse event (AE)/Serious adverse event (SAE) assessment
- o Determine disease status
- o Concomitant medications review
- Assessment of systemic reaction/toxicity/side effects of standard (chemoradiation) therapy (only if subject is screened during chemoradiation therapy)

- o Full physical exam to include complete gynecological exam and ECOG performance status
- Vital Signs (including body temperature, respiratory rate, blood pressure, heart rate and height/weight)
- o 12-lead ECG
- o HPV assessment
- Tumor biopsy collection (required only if residual tissue or unstained slides are not available at screening)
- ThinPrep<sup>TM</sup> sample for HPV testing (if applicable)
- o Digene swab (2 samples) (if applicable)
- o Baseline PET/CT scan (must be performed within 4 weeks prior to Day 0)
- Complete blood count with differential
- Serum chemistry evaluation including glucose, albumin, total protein, SGPT,
   SGOT, alkaline phosphatase, total bilirubin, blood urea nitrogen (BUN),
   calcium, creatinine, electrolytes (chloride, carbon dioxide or bicarbonate,
   potassium, sodium)
- o Baseline CPK
- o Urinalysis
- Serum pregnancy test
- o HIV, Hepatitis B and C serology (not required if performed within 12 months of signing of informed consent)
- O Whole blood and serum for immunologic assays

## 6.1.2 Study Evaluations

Visit dates and windows must be calculated from the date of the Day 0 visit.

The following study evaluations will be performed on **Day 0 prior to study treatment/EP 1**:

- o Determination of eligibility per inclusion and exclusion criteria
- Medical/clinical assessment
- o Targeted physical assessment (including ECOG performance status)
- o AE/SAE event assessment
- Assessment of systemic reaction/toxicity/side effects of standard (chemoradiation) therapy to be completed immediately prior to the first study treatment/EP on Day 0
- o Concomitant medications review
- Vital Signs and Weight
- ThinPrep<sup>TM</sup> sample for HPV testing (if applicable)
- o Digene swab (2 samples) (if applicable)
- Complete blood count with differential
- Serum chemistry evaluation including glucose, albumin, total protein, SGPT, SGOT, alkaline phosphatase, total bilirubin, blood urea nitrogen (BUN), calcium, creatinine, electrolytes (chloride, carbon dioxide or bicarbonate, potassium, sodium)
- Urine pregnancy test
- Whole blood and serum for immunologic assays

# The following study evaluations will be performed on **Day 0, post study** treatment/EP 1:

- O Post-treatment adverse event and injection site reaction assessment within 30-45 minutes after EP
- Distribute Participant Reminder Card (PRC)
- Download EP data

# The following study evaluations will be performed at <u>Weeks 2, 6, 10 and 14 post study treatment/EP</u> ( $\pm$ 1 week):

- Medical/clinical assessment \*
- o Targeted physical assessment (including ECOG performance status)
- Assessment of systemic reaction/toxicity/side effects of standard (chemoradiation) therapy
- Post-treatment injection site reaction assessment\*
- AE/SAE assessment\*
- Concomitant medications review\*
- Review of PRC\*
- Vital Signs and Weight

Weeks 2, 6, 10 and 14 visits may be performed as an in-person office visit or a telephone call. The type of visit will be documented on the case report form. All study procedures listed above should be performed for an in-person visit. The assessments that are required for a telephone call are indicated above with an asterisk (\*).

If the visit will be conducted by telephone, the subject should submit their PRC (i.e. mail, fax, email) to site personnel prior to the phone visit. If the PRC is not received in advance, site personnel should review all PRC elements verbally (see Protocol Section 6.2.4.4). The hard copy of the PRC should be collected and reviewed at the next in-person study visit. After completing a medical/clinical assessment, reviewing the post-vaccination diary and assessing for adverse events and injection site reactions with the subject on the phone, the Investigator will determine whether an office visit is needed for further evaluation.

## The following study evaluations will be performed on Weeks 4, 8 and 12 prior to each study treatment/EP (±1 week):

- o Medical/clinical assessment
- o Targeted physical assessment (including ECOG performance status)
- o Adverse event/serious adverse event assessment
- O Assessment of systemic reaction/toxicity/side effects of standard (chemoradiation) therapy at Week 4 only
- o Concomitant medications review
- Vital Signs and Weight

- Complete blood count with differential
- Serum chemistry evaluation including glucose, albumin, total protein, SGPT, SGOT, alkaline phosphatase, total bilirubin, blood urea nitrogen (BUN), calcium, creatinine, electrolytes (chloride, carbon dioxide or bicarbonate, potassium, sodium)
- Urine pregnancy test
- o Whole blood and serum for immunologic assays at Week 8 only

# The following study evaluations will be performed on **Weeks 4, 8 and 12 post study treatment/EP**:

- O Post-treatment adverse event and injection site reaction assessment within 30-45 minutes after EP
- Distribute and review PRC
- Download EP data

## The following study evaluations will be performed on Week 16 ( $\pm 1$ weeks):

- Medical/clinical assessment
- o Targeted physical assessment (including ECOG performance status)
- o AE/SAE assessment
- Concomitant medications
- o Determine disease status
- o PET/CT scan (must be done EVERY 3-4 months after Day 0)
- Vital Signs and Weight
- Urine pregnancy test
- Tumor biopsy collection
- o ThinPrep™ sample for HPV testing (if applicable)
- o Digene swab (2 samples) (if applicable)
- o Complete blood count with differential
- Serum chemistry evaluation including glucose, albumin, total protein, SGPT,
   SGOT, alkaline phosphatase, total bilirubin, blood urea nitrogen (BUN),
   calcium, creatinine, electrolytes
- o CPK
- Whole blood and serum for immunologic assays

#### The following study evaluations will be performed on Weeks 24 (±2 weeks):

- Medical/clinical assessment
- o Targeted physical assessment (including ECOG performance status)
- o AE/SAE assessment
- Concomitant medications
- Vital Signs and Weight
- Whole blood and serum for immunologic assays

## The following study evaluations will be performed on Weeks 32 (±2 weeks):

- Medical/clinical assessment with ROS
- o Targeted physical assessment (including ECOG performance status)
- o AE/SAE assessment
- Concomitant medications

- Vital Signs and Weight
- o PET/CT scan
- Whole blood and serum for immunologic assays

The following study evaluations will be performed on Week 36 or discharge visit (±2 weeks):

- Medical/clinical assessment
- o Full physical exam (including ECOG performance status)
- o AE/SAE assessment
- Concomitant medications
- o Determine disease status
- Vital Signs and Weight
- o PET/CT scan (not required if performed at wk 32)
- ThinPrep<sup>TM</sup> sample for HPV testing (if applicable)
- o Digene swab (2 samples) (if applicable)
- Whole blood and serum for immunologic assays

## 6.2 Timing and Evaluations

### **6.2.1** Informed Consent

No study specific-assessments or procedures can be conducted until a signed informed consent form (ICF) has been obtained from the subject.

Study personnel will meet with prospective study subjects, explain the study, and provide them with an ICF that describes the screening tests, eligibility criteria for entering the study, and study treatments and follow-up procedures.

#### **6.2.2** Assignment of Screening/Allocation Numbers

Study personnel will screen subjects and assign unique subject identification number (SID). Subject ID numbers are a combination of site number plus a 3-digit number starting with XX1. Information regarding subject's screening number and screen date must be documented on a screening log.

When a subject has been deemed eligible by criteria listed in protocol Section 4 - Selection and Enrollment of Subjects, the clinical site will contact the Sponsor to register the subject and provide the required eligibility information. The site will complete a Subject Identification Form (Appendix 1) and fax or email to the Sponsor prior to enrolling the subject. The Sponsor will assign the subject a unique allocation number based on the cohort the subject will be enrolled and return via fax or email the completed form to the site. Once assigned, the allocation number cannot be reused for any reason.

## **6.2.3** Medical History

Subjects will be asked to report any current or past medical conditions and illnesses at their screening visit and should include treatment detailed information on all therapy directed against cervical cancer, or CIN, e.g. past surgical and/or

radiation regimens. Any prior chemotherapy or immunotherapies, adjuvants, etc. should be recorded on the CRFs.

Any worsening of a condition recorded in the medical history should be recorded as an Adverse Event on the CRFs.

#### **6.2.4** Safety Assessments

Safety evaluations and management of toxicities are detailed in Section 7. Assessments for safety are described within this section.

#### **6.2.4.1** Medical and Clinical Assessments

New onset disease and concomitant medications will be collected on Day 0 and at all subsequent study visits through discharge.

Assessment of systemic reaction/toxicity/side effects of standard (chemoradiation) therapy will be collected at specified visits and be reported using the "Acute Radiation Morbidity Scoring Criteria (RTOG)", (Appendix 5).

Assessment of all other adverse events will be collected form the time of informed consent through discharge and will be will be assessed using the CTCAE v4.03 issued by the US Department of Health and Human Services on June 14, 2010 (Appendix 4).

Clinical evaluations for disease response will be conducted at all of the study visits (as assessed by clinical signs and symptoms of disease progression). PET/CT scans for disease progression will be obtained for all subjects 3-5 months after Day 0 and every 3-5 months thereafter per standard of care or in accordance with local guidelines and institutional practices.

#### **6.2.4.2 Physical Assessments**

A full examination including complete gynecological exam and ECOG performance status will be conducted during screening and study discharge. A targeted physical assessment (including ECOG performance) will be performed at other visits as determined by the Investigator or directed per subject complaints.

#### **6.2.4.3 Post-Treatment Reaction Assessment**

The Investigator will assess local and systemic reactions post-treatment (within 30-45 minutes after study treatment/EP) and at specified visits. Any reported local post treatment reactions will be graded per the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials and any reported systemic post treatment reactions will be graded per CTCAE v4.03 and recorded on the CRFs (see Section 6.6 for more details).

## 6.2.4.4 Participant Reminder Card

Subjects will be given an oral thermometer and participant reminder card (PRC) at each study treatment/EP visit. Subjects will be instructed to take and record their temperature daily (at the same time each day). They will also be advised to record local and systemic events on a PRC as shown in Appendix 9.

If Weeks 2, 6, 10 and 12 visits are conducted by telephone, the subject should submit their PRC (i.e. mail, fax, email) to the site personnel prior to the phone visit. If the PRC is not received in advance, site personnel should verbally review all PRC elements listed above. The hard copy of the PRC should be collected at the next in-person study visit. Any entry on PRC determined to meet the criteria for a Grade 1 or higher adverse event should be documented as adverse event. If the PRC entry does not meet the criteria of a Grade 1 or higher AE as per the CTCAE v4.0, clinical judgment can be used to determine whether the entry should be recorded as an AE. For cases where the PRC entry and final AE reporting (i.e., grading) do not agree, the reasoning should be recorded in the source documents.

## 6.2.4.5 Vital Signs

Vital signs including body temperature, respiration rate, blood pressure and heart rate will be measured at all the study visits.

## 6.2.4.6 Weight and Height

Weight (kg) and height (cm) will be collected at the screening visit. Weight will be collected at each additional visit from Day 0 through discharge.

#### 6.2.4.7 12-lead ECGs

An ECG will be performed at screening within 30 days of signing of ICF for all subjects to determine subject eligibility. Abnormal ECGs should be interpreted as clinically significant or not clinically significant.

### 6.2.4.8 Pregnancy Test

For women of reproductive potential, a negative result for serum pregnancy test (test must have a sensitivity of at least 25 mIU/mL) must be available at the screening visit and urine  $\beta$ -HCG (pregnancy test) prior to each administration of INO-3112 and prior to tumor biopsy collection. If at any point, the  $\beta$ -HCG (pregnancy) test is positive, indicating that the subject is pregnant, no additional study treatment/EP will be administered, but the subject will be followed for the duration of the study and beyond to determine the outcome of the pregnancy (with the subject's consent).

#### **6.2.4.9 Laboratory Evaluations**

At screening, blood samples will be collected for serum chemistry and hematology. A urine sample will also be obtained to determine eligibility. At other visits, blood samples will be collected as specified in Table 1 - Schedule of Events. All labs for Day 0 and those associated with any treatment visit should be collected no more than 48 hours prior to treatment and reviewed/evaluated by the PI prior to treatment. Approximately 4 cups of blood will be drawn from each subject during the entire duration of the study.

## Complete blood count (CBC)

White blood cell (WBC) count w/ differential

Red blood cell (RBC) count

Hemoglobin, Hematocrit

Platelet count

## Serum Chemistry

Glucose

Albumin

Total protein

SGPT (serum glutamic-pyruvic transaminase)/ALT

SGOT (serum glutamic-oxaloacetic transaminase)/AST

Alkaline phosphatase

Bilirubin (total)

BUN (blood urea nitrogen)

Calcium

Creatinine

Electrolytes (Sodium, Potassium, Chloride, Carbon Dioxide or Bicarbonate)

## CPK (Creatine Phosphokinase)

Serology (required only at screening if serologic test was performed  $\geq 12$  months of informed consent)

Antibody to HIV

Hepatitis B surface antigen

Antibody to Hepatitis C

### **Urinalysis**

Urine samples will be tested by dipstick for glucose, protein, and hematuria. If abnormal (presence of protein, hematuria, or glucose  $\geq 1+$ ) a microscopic examination will be performed.

#### 6.2.4.10 PET/CT Scan

Baseline PET or CT scan must be performed within 4 weeks prior to Day 0.

The follow-up scan will be performed 3-4 months after Day 0 to evaluate subject disease status. Thereafter, PET/CT scans can be performed 3-5 months or at study discharge in accordance with local guidelines and institutional practices.

FDG-PET imaging is based on the increased glucose metabolism of tumor cells compared to normal tissue resulting in higher standard uptake volume (SUV). Increased SUV<sub>max</sub> at diagnosis has been associated with persistent abnormal FDG uptake after curative chemoradiation and biopsy-proven local recurrence [Kidd 2007]. FDG-PET is already utilized as a follow-up evaluation modality in a variety of cancers, including lymphomas, head and neck cancers, and breast cancer [Schelling 2000, Smith 2000, Weber 2001, Ott 2003, Weber 2003, Brun 2002].

In a prospective study of cervical cancer patients, FDG-PET was demonstrated to be a metabolic biomarker of response and a potential prognostic marker for progression-free survival at 3 years [Schwarz 2007]. A meta-analysis of 16 studies also demonstrated statistical significance for prediction of event-free and overall survival using metabolic response derived from PET and PET/CT imaging [Zhao 2013].

Studies have previously described the abscopal effect of radiation therapy on non-irradiated tumor sites in a variety of cancers [Postow 2012, Prise 2009]. Post-treatment FDG-PET may further provide elucidation of this mechanism by highlighting sites of residual activity. Retrospective and prospective studies have demonstrated that the use of positron emission tomography (PET) with F-18 fluorodeoxyglucose (FDG) in the post-therapy evaluation of patients with cervical carcinoma is predictive of survival outcome [Grigsby 2004, Grigsby 2003].

These studies evaluated patients with similar disease stage to our current investigation and found that SUV PET response at 3 months after chemoradiation correlated with survival and patterns of failure. We propose to describe qualitatively the rates of complete metabolic response (CMR), partial metabolic response (PMR), and progressive disease (PD) in our patient population and compare these rates to patients treated per standard of care in the aforementioned studies to preliminarily explore any differential outcomes.

## 6.3 Study Treatment/EP with INO-3112

The timing of the first dose will be designated Day 0.

## 6.3.1 Management of anxiety and pain due to EP procedure

Subjects will be offered topical anesthetic (e.g. EMLA), to prevent significant discomfort from the study treatment/EP procedure. If EMLA (lidocaine 2.5% and prilocaine 2.5%) is used, an approximately 1.5 cm diameter amount will be applied with occlusion to the site of injection ~30 minutes prior to study treatment/EP.

Subjects may be offered a mild sedative (e.g. 0.5-1 mg lorazepam) for anxiety related to the EP procedure. Mild sedatives may be administered approximately 1 hour prior to EP at Weeks 0, 4, 8 and/or 12. Subjects who receive a mild sedative must not be allowed to operate a motor vehicle for 3-4 hours after receiving medication and must have arranged transportation to depart the study site.

Subjects will be offered an analgesic (e.g. ibuprofen, ketorolac) after study treatment/EP. [Note: The use of any narcotic (including Tylenol with codeine) for pain meets the definition of severe pain (Grade 3) as per the "Guidance for Industry - Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, September 2007" (Table 6.1) and therefore do not offer this to the patient unless clinically indicated.]

Subjects who are allergic to or have contraindications to ibuprofen, ketorolac or lorazepam will be offered a suitable alternative.

#### **6.4** Assessment of Clinical Adverse Events

The injection site will be assessed by study personnel prior to and within 30-45 minutes after study treatment/EP and at next visit prior to study treatment/EP.

Subjects will also be queried regarding the occurrence of any possible adverse events, concomitant medications and new onset chronic disease during their clinic visits. Subjects will be reminded to contact study personnel and immediately report any event that may happen for the duration of the study. These events will be recorded on the subject's CRF.

At specific visits the Acute Radiation Morbidity Scoring Criteria (RTOG) (Appendix 5) will be used to assess systemic reaction/toxicity/side effects of standard (chemoradiation) therapy.

### 6.5 Assessment of Laboratory Abnormalities

Investigators may use clinical judgment to enroll subjects with isolated Grade 1 abnormalities in screening CBC, serum chemistry or CPK values if there is no indication of disease process in the remainder of the history and physical examination.

Blood will be drawn for serum chemistry, hematology and serology assessments as well as pregnancy testing at screening for inclusion into the study as listed in sections 6.2.4.8 and 6.2.4.9.

Urinalysis will be performed at screening to fulfill eligibility criteria. CPK will be performed at Screening and Week 16.

Complete blood count with differential and serum chemistry will be performed at each study treatment/EP and Week 16.

### 6.6 Assessment of Injection Site Reactions

When evaluating injection site reactions throughout the study, the investigator will be instructed to use the following grading scale:

**Table 6.1: Grading Scale for Injection Site Reactions** 

| Local Reaction to<br>Injectable Product<br>(Grade) | Mild(1) | Moderate(2) | Severe(3) | Potentially Life<br>Threatening(4) |
|---|---|---|---|---|
| Pain | Does not interfere with activity | Repeated use of<br>non-narcotic<br>pain reliever<br>>24 hours or<br>interferes with<br>activity | Any use of<br>narcotic pain<br>reliever or<br>prevents daily<br>activity | Emergency room<br>(ER) visit or<br>hospitalization |
| Tenderness | Mild discomfort to touch | Discomfort with movement | Significant discomfort at rest | ER visit or hospitalization |
| Erythema/Redness* | 2.5-5 cm | 5.1-10 cm | >10 cm | Necrosis or exfoliative dermatitis |
| Induration/Swelling** | 2.5-5 cm and does not interfere with activity | 5.1-10 cm or interferes with activity | >10 cm or<br>prevents daily<br>activity | Necrosis |

September 2007 "FDA Guidance for Industry—Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials"

## 6.7 Cervical Virologic and Peripheral Blood Immunogenicity Assessment

Whole blood and serum samples to be tested for antibodies to the HPV E6 and E7 proteins and/or T-lymphocytes producing IFN- $\gamma$  will be obtained at baseline (Screening and Day 0 prior to dosing) and at each study treatment/ EP and follow-up visits for the duration of the trial. Other immunological testing may be performed to further define the immune responses to the INO-3112. Details of the immunology sample collection and shipment will be provided in laboratory manual.

Binding antibody responses against HPV E6 and E7 induced by INO-3112 will be measured using ELISA. Commercially available recombinant human HPV-16 and HPV-18 proteins will be used to assess induction of binding antibodies to each of the antigen components.

Using antigen-specific IFN- $\gamma$  ELISpot assays, the number of antigen-specific IFN- $\gamma$ -secreting T-cells in response to stimulation with overlapping peptide libraries spanning consensus antigens HPV16 E6, HPV16 E7, HPV18 E6 and HPV18 E7 will be determined. As previously described [Bagarazzi et al Sci Tran Med]. PBMCs will be incubated with HPV peptide pools at a concentration of 2  $\mu$ g/ml. IFN- $\gamma$  release will be detected after an overnight incubation. Spot forming units (SFU) will be adjusted to 1 × 10<sup>6</sup> PBMCs for each HPV peptide pool.

Flow cytometric assays will be employed to examine any or all of the following characteristics of Study Treatment: induction of T-cells to 1) exhibit phenotypic

<sup>\*</sup>in addition to grading the measured local reaction at the greatest single diameter, the measurement should be recorded as a continuous variable.

<sup>\*\*</sup>Induration/Swelling should be evaluated and graded using the functional scale as well as the actual measurement.

markers associated with cytolytic potential after short-term stimulation by HPV antigen (i.e., CTL phenotyping); 2) remain active in the presence of long-term antigen exposure and efficiently synthesize proteins used in lytic activity (i.e., Lytic granule loading); and 3) effectively employ lytic degranulation to drive killing of target cells expressing HPV antigens (i.e., Killing Assay)

**HPV-004** 

Clinical Protocol

- 1. The CTL phenotyping assay employs short term (4-6 hours) in vitro stimulation of unfractionated PBMC using peptides spanning HPV antigens and appropriate controls. The external cellular markers employed in this assay might include CD3, CD4, CD8 (T-cell identification), CD45RO, CCR7 (memory subset identification) and CD107a (lytic degranulation). The CTL Phenotyping assay may additionally analyze the following intracellular markers: IFN-γ (Th1 biasing cytokine), Tumor Necrosis Factor-α (TNF-α), Granzyme A, Granzyme B and Perforin (involved in lytic degranulation and cytotoxic potential). This panel may vary as additional relevant markers are identified.
- 2. The lytic granule loading assay employs long term (115-120 hours) in vitro stimulation of unfractionated PBMC using peptides spanning HPV antigens and appropriate controls. The external cellular markers employed in this assay might include CD3, CD4, CD8 (T-cell identification) and CD137 (also known as 41BB, T-cell activation). The Lytic granule loading assay may additionally analyze the following intracellular markers: Granzyme B, Perforin and Granulysin (cytotoxic potential). This panel may vary as additional relevant markers are identified.
- 3. The killing assay employs long term (115-120 hours) in vitro stimulation of unfractionated PBMC using peptides spanning HPV antigens. After the initial long term incubation, stimulated whole PBMC or CD8+ T-cells (hereafter referred to as Effector Cells) are co-incubated for ~1 hr with target cells treated with a stain (Target Stain) that differentiates them from Effector Cells and have additionally been pulsed with a substrate reagent which is activated only by the activity of Granzyme B or a substrate which is activated by the activity of terminal caspases involved in the induction and perpetuation of apoptosis. Enumeration of target cells identified by the Target Stain and the presence of an active substrate reagent within the Target population represents a measure of a functional T cell response that is capable of Target cell killing.

A standardized binding ELISA will be performed to measure the anti–HPV16/HPV-18 E6 or E7 antibody response induced by INO-3112. 96-well enzyme immunoassay plates will be coated with HPV16 or HPV18 E6 or E7 proteins (1  $\mu$ g/ml).

PBMC responses against a pool of known antigenic epitopes pooled from Cytomegalovirus, Epstein Barr Virus and Influenza (CEF) will be tested in order to track general cellular immune competence during the study. Assessment of the

response to these reference antigens that are not related to the study antigens will give a baseline reading of immunocompetency at study entry. Observation for variation of response against these reference antigens during the progression of study treatment may therefore give insight as to general immune competency and aid in accounting for variation in response against study antigens encoded by INO-3112 in the same manner as HPV response described above.

## Cervical Virologic Assessment

Subjects must have positive HPV-16 and/or HPV-18 genotype result from ISH or PCR assays at screening or prior to screening for inclusion in the study. Subjects whose specimens also test positive for other HPV genotypes are not excluded as long as they have a positive result for HPV 16 and/or HPV 18. If a subject has documented evidence of HPV-16 and/or HPV-18 infection results from cervical specimen obtained prior to anti-cancer treatment, then those results will be eligible for inclusion in the study.

If applicable, a liquid based cytology sample (ThinPrep<sup>™</sup>) will be collected for HPV PCR at screening and at Weeks 16 and 36. Samples will be sent to a central laboratory to be analyzed for the presence of HPV infection by PCR.

## Cervical Immunologic Assessment

If applicable, two Digene cervical brushes will be collected at baseline (screening and Day 0), Weeks 16 and 36 and will be banked and frozen for immunological testing.

Tissue specimens obtained as routine diagnostic and therapeutic specimens will be analyzed to characterize the presence, density, and co-localization of immune cell subsets, including macrophages, dendritic cells, T cells (CD8 and regulatory T cells), and NK cells. As tissue availability permits, the specimens will also be analyzed for cytokine expression.

At visits where multiple cervical samples are collected, the two Digene cervical brushes will be collected prior to the ThinPrep<sup>TM</sup> sample.

If adequate residual specimen is available, immunohistochemistry (IHC) studies will be performed on either tumor tissue block or unstained slides from tumor(s) from the following time points: (1) at screening; (2) at Week 16 (one month postdose 4).

A tumor biopsy will be used to investigate the post-radiation changes at a cellular level, with particular focus on the presence and populations of immune cells to compare to pre radiation characterization.

Characterization of the various cell populations present in the primary tumor site will allow for elucidation of long-term effects of radiation-induced changes, potential cell-mediating killing in microscopic colonies of residual tumor, and mechanisms of immune cell interactions in the post-radiation setting. The maturation and clonal expansion of T cells in response to repeated immunotherapy should result in the production of a memory T cell subset in the immune cell population.

Biopsy samples can also be compared to the post-dose peripheral blood samples to study shifts in cell populations or HPV-specific proliferative response. In addition, biomarkers may be identified as predictors of early response, resistance, or recurrence, and contribute to patient outcome stratification.

#### 6.8 Disease Status

Diseases status will be determined based on RECIST (version 1.1). Disease status should be categorized into:

- 1. No evidence of disease (NED)
- 2. Partial Response
- 3. Stable disease
- 4. Progressive disease

#### 6.9 Concomitant Medications/Medical Care

All medications taken or medical procedures performed within 12 weeks prior to Day 0 and during the study must be recorded on the case report forms (CRFs).

## 6.10 Permitted Supportive Therapy

Anti-emetics, anti-diarrheals, analgesics, nutritional and fluid supplementation, and packed red blood cell transfusions are permitted as supportive therapy during the study. All medications and interventions must be recorded as concomitant medications in the CRFs.

## 6.11 HLA Testing

A blood sample will be collected at the Day 0 visit and sent to a central laboratory for HLA typing. If the subject has a record of previous high resolution HLA testing and access to the results, this HLA testing is not required.

### 6.12 Downloading of EP data from CELLECTRA®-5P device

Within 48 hours following each treatment with INO-3112, data should be downloaded from the EP device and the data file that is created should be sent to the Sponsor or designee by email to CELLECTRAdata@inovio.com. Instructions on how to download the data are provided in Appendix 7. Training will be provided.

#### 6.13 Restrictions

Subjects should not be vaccinated (e.g. influenza vaccine) within 2 weeks of (before or after) any dose of INO-3112.

Subjects should not receive a course of systemic corticosteroids (≥2 mg/kg of prednisone or equivalent for 5 days) within 2 weeks before or after any dose of INO-3112.

### 7 EVALUATION OF SAFETY AND MANAGEMENT OF TOXICITY

## 7.1 Safety Parameters

The safety of the INO-3112 DNA plasmid vaccines will be measured and graded in accordance with the document entitled "Common Terminology Criteria for Adverse Events (CTCAE)", version 4.03 issued by the US Department of Health and Human Services on June 14, 2010 (Appendix 4).

### 7.1.1 Adverse Events (AEs)

An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body, or worsening of a pre-existing condition, temporally associated with the use of a product whether or not considered related to the use of the product. In this study, such changes will be monitored, classified, and summarized, and as <u>Clinical</u> or <u>Laboratory</u> AEs, respectively. Medical condition/diseases present before starting the investigational drug will be considered adverse events only if they worsen after starting study treatment.

An <u>unexpected</u> AE is one not identified in the Clinical Investigator's Brochure (CIB) or otherwise not expected from the characteristics of the clinical material. AEs include the following:

- Pre- or post-treatment complications that occur as a result of protocol mandated procedure during or after the first screening visit (before the administration of study drug)
- Any pre-existing condition that increases in severity, or changes in nature during or as a consequence of the study drug phase of a human clinical trial, will also be considered an AE
- Complications and termination of pregnancy; see Section 7.4 for additional information
- All AEs that occur from the study screening visits onwards and throughout the duration of the study, including the follow-up off study treatment period should be recorded as an AE

AEs do not include the following:

- Medical or surgical procedures (e.g., surgery, endoscopy, tooth extraction, transfusion) performed; the condition that leads to the procedure is an AE
- Pre-existing diseases or conditions or laboratory abnormalities present or detected before the screening visits that do not worsen
- Situations where an untoward medical occurrence has not occurred (e.g., hospitalization for elective surgery, social and/or convenience admissions).
- Overdose without clinical sequelae

- Any medical condition or clinically significant laboratory abnormality
  with an onset date before the consent form is signed and not related to
  a protocol associated procedure is not an AE. It is considered to be
  pre-existing and should be documented on the medical history CRF
- Uncomplicated pregnancy (documented on a pregnancy CRF)
- An induced elective abortion to terminate a pregnancy without medical reason (documented on a pregnancy CRF)

#### 7.1.2 Serious Adverse Events (SAEs)

A serious adverse event (SAE) is any AE that meets one of the following conditions:

- Death during the period of surveillance defined by the protocol;
- Is immediately life-threatening (e.g., subject was, in the view of the Investigator, at immediate risk of death from the event as it occurred). This does not include an AE that, had it occurred in a more serious form, might have caused death;
- An event requiring inpatient hospitalization or prolongation of existing hospitalization during the period of protocol defined surveillance (including any overnight stay in the hospital, regardless of the length of stay, even if the hospitalization is only a precautionary measure to allow continued observation. However, hospitalization (including hospitalization for an elective procedure) for a pre-existing condition that has not worsened, does not constitute an SAE;
- Results in congenital anomaly or birth defect;
- Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions;
- Is an important medical event that may not result in death, be life threatening, or require hospitalization, but based upon appropriate medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse;
- Is medically significant or requires intervention to prevent one or other of the outcomes listed above. Examples of "other medically significant events" are:
  - Intensive treatment in an emergency room or at home for allergic bronchospasm
  - o Blood dyscrasias or convulsions that do not result in hospitalization
  - o Development of drug dependency or drug abuse

## Development of malignancies

#### Clarification of Serious Adverse Events

- Death is an outcome of an AE, and not an adverse event in itself
- The subject may not have been on investigational medicinal product at the occurrence of the event. Dosing may have been given as treatment cycles or interrupted temporarily before the onset of the SAE, but may have contributed to the event
- "Life-threatening" means that the subject was at immediate risk of death from the event as it occurred. This does not include an event that might have led to death if it had occurred with greater severity
- Complications that occur during hospitalizations are AEs. If a complication prolongs the hospitalization, it is an SAE
- Inpatient hospitalization means the subject has been formally admitted to a hospital for medical reasons, for any length of time. This may or may not be overnight. It does not include presentation and care within an emergency department

The investigator should attempt to establish a diagnosis of the event on the basis of signs, symptoms, and/or other clinical information. In such cases, the diagnosis should be documented as the AE and/or SAE and not the individual signs/symptoms.

Serious adverse events that are ongoing should be followed until resolution. The reporting period for SAEs is described in Section 9.3.2.

#### 7.1.3 Severity Codes for AEs

Study personnel will grade laboratory AEs and clinical AEs (based on discussions with study participants) with respect to the following levels of severity as defined in Common Terminology Criteria for adverse events (CTCAE) of the National Cancer Institute for reporting of all serious adverse events (SAE) or the Acute Radiation Morbidity Scoring Criteria (RTOG).

- Mild (Grade 1);
- Moderate (Grade 2)
- Severe (Grade 3);
- Potentially Life Threatening (Grade 4)
- Death (Grade 5)

A copy of the CTCAE version 4.03 is provided in Appendix 4 and may be downloaded from the CTEP home page (http://ctep.cancer.gov/reporting/ctc.html):

A copy of the Acute Radiation Morbidity Scoring Criteria can be downloaded from the Radiation Oncology Therapy Group home page (<a href="http://www.rtog.org/ResearchAssociates/AdverseEventReporting/AcuteRadiationMorbidityScoringCriteria.aspx">http://www.rtog.org/ResearchAssociates/AdverseEventReporting/AcuteRadiationMorbidityScoringCriteria.aspx</a>).

## 7.2 Causal Relationship of Clinical Material to AEs

A causally related AE is one judged to have a possible, probable or definite relationship to the administration of the clinical material (INO-3112). An AE may also be assessed as not related to the investigational product. The Investigator is responsible for reporting adverse events and judging the relationship between the administration of the clinical material and a subsequent AE because the investigator is knowledgeable about the subject (e.g., medical history, concomitant medications), administers the investigational product, and monitors the subject's response to the investigational product. The Investigator is aware of the subject's clinical state and thus may be sensitive to distinctions between events due to the underlying disease process versus events that may be product related and may have observed the event. The Sponsor will assess the overall safety of the investigational product and determine whether to report expeditiously to the FDA.

The following guidance should also be taken into consideration:

- Temporal relationship of event onset to the initiation of study drug;
- Course of the event, considering especially the effects of dose reduction, discontinuation of study drug, or reintroduction of study drug (where applicable);
- Known association of the event with the study drug or with similar treatments;
- Known association of the event with the disease under study;
- Presence of risk factors in the Study Subject or use of concomitant medications known to increase the occurrence of the event:
- Presence of non-treatment-related factors that are known to be associated with the occurrence of the event

### 7.2.1 Abnormal Laboratory Value

Laboratory abnormalities are usually not recorded as AEs or SAEs. However, laboratory abnormalities (e.g., serum chemistry, hematology, CPK, urinalysis) independent of the underlying medical condition that require medical or surgical intervention or lead to study treatment interruption or discontinuation must be recorded as an AE, as well as an SAE, if applicable. In addition, laboratory or other abnormal assessments (e.g., electrocardiogram, x-rays, vital signs) that are associated with signs and/or symptoms must be recorded as an AE or SAE if they meet the definition of an AE (or SAE) as described in Sections 7.1.1 and 7.1.2. If the laboratory abnormality is part of a syndrome, record the syndrome or diagnosis (e.g., anemia) not the laboratory result (e.g., decreased hemoglobin). Any laboratory abnormality that is new in onset or worsened in severity or

Any laboratory abnormality that is new in onset or worsened in severity or frequency from the baseline condition and meets one of the following criteria will be recorded as an AE:

- Requires the rapeutic intervention or diagnostic tests
- Leads to discontinuation of study treatment
- Has accompanying or inducing symptoms or signs

## • Is judged by the investigator as clinically significant

Grade is an essential element of these criteria. Each CTCAE grading term in the current version is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT).

Investigators are asked to take the CTCAE grading criteria into account when assessing if a laboratory abnormality qualifies as a laboratory AE. Their clinical judgment ultimately determines whether the abnormality in question is "clinically significant (CS)" or "not clinically significant (NCS)" and the severity of the event. CTCAE grading can be used as a reference when making this determination. It is the responsibility of the Investigators to ensure all AEs are accurately reported and graded.

## 7.2.2 Post-Study Reporting Requirements

All AEs and SAEs including deaths, regardless of cause or relationship, must be reported for subjects on study (including any protocol-required post-treatment follow-up).

Investigators are not obligated to actively seek AEs or SAEs beyond study discharge for subjects. However, if the investigator learns of an AE or SAE that occurs after the completion or termination visit and the event is deemed by the investigator to be probably or possibly related to the Study Treatment, he/she should promptly document and report the event to Inovio Pharmaceuticals.

## 7.3 Methods and Timing of the Collection and Recording of Safety Data

After study treatment/EP: Study subjects will be directly observed by study personnel for 30-45 minutes after each administration of study treatment/EP for immediate reactions. Injection sites will also be assessed at the subsequent study visit.

The occurrence and severity of any AE during this period or the lack of same will be recorded on the appropriate CRF. Subjects will be given an oral thermometer and instructed to take and record their temperature daily (at the same time each day).

Days 0-3 following study treatment/EP: Subjects will also be instructed to record local and systemic events in a PRC for 3 days following treatment visit as shown in Appendix 9.

<u>Throughout the Study:</u> Subjects will also be queried regarding the occurrence of any possible adverse events, concomitant medications and new onset chronic disease during their clinic visits. Subjects will be reminded to contact study personnel and immediately report any event that may happen for the duration of the study. These events will be recorded on the subject's CRF.

At specified visit the Acute Radiation Morbidity Scoring Criteria (RTOG) form will be completed for each patient to assess systemic reaction/toxicity/side effects of standard (chemoradiation) therapy.

On study treatment/EP visits, the assessments will be performed prior to dosing. Study subjects will be queried at each clinic visit regarding the occurrence of any AEs, including SAEs that may have occurred since the last visit. They will be reminded to contact study personnel and immediately report any such event that happens during the course of the study. These events will be recorded on the CRFs.

## 7.4 Procedures for Documenting Pregnancy During Study

Subjects who are pregnant or expect to become pregnant during the course of the study will be excluded from participation in the study. Should a subject become pregnant after enrolling in the study, she will not be given any further treatments with INO-3112. The Investigator will report this event to Inovio Pharmaceuticals, Inc., or its designee, within 24 hours and to the IRB. The Investigator should counsel the participant and discuss risks of continuing with the pregnancy and the possible effects on the fetus. Sites must request the subject's permission to query pregnancy outcome and follow each subject to determine the outcome of the pregnancy. Results will be summarized in the clinical study report (CSR).

Subjects who become pregnant at any point during the study should continue to be followed for safety assessments without receiving further treatments. Procedures that are contraindicated during pregnancy, including additional vaccinations, must not be performed. Investigators should use clinical judgment regarding subsequent study-related blood collection based on the presence or absence of anemia in each subject. Subjects who are not withdrawn should continue to be followed for safety assessments through discharge per protocol.

All pregnancies that occur from the time of first screening procedure through the follow up visits must be reported. Monitoring of the subject and the outcome of the pregnancy should be followed by the investigator. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Inovio Pharmaceuticals.

### 7.5 Toxicity Management

The Sponsor's Medical Monitor will be responsible for the overall safety monitoring of the study.

## 7.5.1 Criteria for Halting of Study Enrollment

Study enrollment (enrollment of new subjects) will be halted if there is a report of Grade 3 anaphylaxis from study treatment/EP with INO-3112. The study may resume enrollment after the safety data has been reviewed and deemed safe to continue by the Medical Monitor and Investigator.

## 7.5.2 Events Requiring Expedited Reporting

Events requiring expedited reporting (ERER) will be defined as treatment- or EP-related adverse events including any of the following:

- Grade 3 or greater injection site pain, tenderness, erythema, and/or induration recorded ≥ 1 hour after study treatment (see Table 6.1)
- Grade 3 or greater fever assessed by the Principal Investigator as possibly, probably or definitely related to study treatment
- Grade 3 or greater systemic symptoms assessed by the Principal Investigator as possibly, probably or definitely related to study treatment

as defined in the "Common Terminology Criteria for Adverse Events (CTCAE)", version 4.03 issued by the US Department of Health and Human Services on June 14, 2010 (Appendix 4). The worse grade for that particular event is to be documented on the CRFs.

Sites should inform the Sponsor of any ERER within 72 hours to discuss whether further dosing should continue for that participant.

## 7.5.3 Stopping Rules (Criteria for Pausing of Study)

- 7.5.3.1 If at any time during the study one third (1/3) or more subjects experience an ERER assessed as possibly, probably or definitely related to study treatment, further enrollment and study treatments will be halted immediately until a thorough investigation has been conducted by the Medical Monitor and Principal Investigator.
- 7.5.3.2 After any SAE, potentially life threatening AE or death assessed as possibly, probably or definitely related to study treatment, further enrollment and study treatments will be halted immediately until a thorough investigation has been conducted by the Medical Monitor, Principal Investigator and IRB (if applicable).
- 7.5.3.3 If three or more subjects in this study, experience the same grade 3 or 4 adverse event, assessed as possibly, probably or definitely related to study treatment, further enrollment and study treatments will be halted immediately until a thorough investigation has been conducted by the Medical Monitor and Principal Investigator.
- 7.5.3.4 In the event of any unexpected Grade 4 toxicities, assessed as possibly, probably or definitely related to study treatment, further enrollment and study treatments will be halted immediately until a thorough investigation has been conducted by the Medical Monitor, Principal Investigator and IRB (if applicable).

7.5.3.5 The study will be halted for any report of Grade 3 anaphylaxis from immunotherapy/EP with INO-3112 in two or more patients (as graded per "Common Terminology Criteria for Adverse Events (CTCAE)", version 4.03 issued by the US Department of Health and Human Services on June 14, 2010 (Appendix 4)).

#### 8 STATISTICAL CONSIDERATIONS

## 8.1 Sample Size Considerations

Per Rose et al., the percentage of patients with grade 3 or 4 hematologic toxicity was 23%. With n=10 patients in this study, there is approximately a 92% chance of observing of at least one grade 3 or 4 hematologic toxicity. If 0 out of 10 adverse events are observed, the study provides 95% confidence that the true proportion of such events is <31%.

## 8.2 Safety Analysis

With the toxicity results, data from the Acute Radiation Morbidity Scoring Criteria and CTCAE will be recorded for each patient during each visit. For the toxicity results, and for AEs and injection site reactions, descriptive statistics will be generated tabulating the percentage of subjects with events by type and grade along with associated exact 95% Clopper-Pearson confidence intervals.

### 8.3 Analysis of Immune Responses

Binary responses, i.e., responders/non-responders, will be analyzed by calculating the percentage of responders along with associated exact 95% Clopper-Pearson confidence intervals. Continuous responses, e.g., immune levels, will be analyzed by calculating the mean or median responses along with associated 95% confidence intervals.

## 8.4 Analysis of Clinical Responses

Disease status frequencies based on RECIST criteria categories will be summarized.

## 8.5 Summary of Demographic and Other Baseline Characteristics

Demographic and baseline characteristics will be summarized with means, medians, standard deviations, ranges or percentages.

### 8.6 Missing Values

Missing data will not be imputed.

### 8.7 Site Effects

The data will be summarized by site and compared observationally among sites.

## 9 DATA COLLECTION, MONITORING, AND AE REPORTING

## 9.1 Records to Be Kept

CRFs will be provided for each subject. Subjects must not be identified by name on any CRFs. Subjects will be identified by their subject identification number (SID) provided by Inovio Pharmaceuticals, Inc.

## 9.2 Safety and Quality Monitoring and Record Availability

### Monitoring

Monitoring of the clinical trial will be performed by experienced monitors, who will report to the Sponsor. Records for all clinical subjects in this trial will be monitored. The following clinical site monitoring tasks will be performed at all sites:

- Prior to trial initiation, a site visit will be conducted to review all relevant forms and documentation, to ensure compliance with all applicable requirements.
- All clinical site monitoring visits will be documented.
- Periodic site visits will be performed on a per dose group basis.
- The site monitor will be responsible for addressing and documenting the following study conduct activities and obligations and will:
  - o Assure that the study is being conducted in accordance with the protocol, applicable regulatory agency regulations, and IRB policies.
  - Discuss study conduct issues and incidents of noncompliance with the Investigator and/or study personnel and document them on the resolution trip report. Report any significant unresolved problems immediately to the sponsor.
  - Remind the Investigator as necessary of the obligation to immediately report SAE and provide subsequent follow-up report of the final outcome to the IRB.
  - o Review all CRF pages for completeness, logic, and internal consistency throughout the study.
  - Assure that the study facilities continue to be acceptable.
  - o Compare the study CRFs with source documents to assure that the data are accurate and complete and that the protocol is being followed.
  - Assure that investigational product and device accountability and reconciliation records are complete and accurate.
  - Assure that all subject specimens are being stored and forwarded properly for testing.

## **Record Availability**

The investigator will make study documents (e.g., ICFs, drug distribution forms, CRFs) and pertinent hospital or clinic records readily available for inspection by the local IRB, the site monitors, the FDA, Inovio or its designee or confirmation of the study data.

## 9.3 Adverse Experience (AE) Reporting

To assure the safety of the participants, information about all AEs (see Section 7.1 Safety Parameters for definitions), whether volunteered by the subject, discovered by investigator or study staff questioning, or detected through physical examination, laboratory test or other means, will be collected and recorded in the subject's source documents and followed as appropriate.

### 9.3.1 Study Reporting Period of Adverse Events

The reporting period for AEs due to chemoradiation therapy toxicity is the period immediately following initiation of chemoradiation through the Week 4 visit of the study.

The reporting period for all other AEs is the period immediately following informed consent through the end of the study

## 9.3.2 Study Reporting Period of Serious Adverse Events

The reporting period for SAEs (without regard to causality) is the entire period following informed consent until the end of the study.

Each AE will be assessed to determine whether it meets seriousness criteria. If the AE is considered serious, the investigator should report this event to Inovio Pharmaceuticals as outlined below and also to the Ethics Committee according to its standard operating procedures.

Expectedness of SAEs will be determined by Inovio Pharmaceuticals using reference safety information specified in the Investigator's Brochure. An event may qualify for expedited reporting to regulatory authorities if it is a SAE, serious adverse drug reaction, or suspected unexpected serious adverse reaction (SUSAR) in line with relevant legislation. All investigators will receive a safety letter notifying them of relevant SUSAR reports. The investigator should notify the Ethics Committee as soon as is practical, of serious events in writing where this is required by local regulatory authorities, and in accordance with the local institutional policy. The investigator should send the initial report to sponsor within 24 hours of becoming aware of the event. At minimum, the initial report should include the following information:

- Event
- Study code
- Subject number, initials and date of birth
- Investigational study product
- Reporter name and contact information

In the case of a "minimum report" (one that is solely comprised of the information bulleted above), a more detailed follow-up report should be sent as soon as more information becomes available but no later than 7 calendar days after the date of the initial report. Each SAE should be followed up until resolution or stabilization and for a reported death, the

investigator should provide Inovio Pharmaceuticals and the Ethics Committee with any additional requested information (e.g., autopsy reports and terminal medical reports).

The original SAE form should be kept at the study site. Inovio Pharmaceuticals or its representative will be responsible for determining and in turn, reporting SAEs to regulatory authorities according to the applicable regulatory requirements.

SAEs must be followed by the investigator until resolution, even if this extends beyond the study-reporting period. Resolution of an SAE is defined as the return to baseline status or stabilization of the condition with the expectation that it will remain chronic.

At any time after completion of the SAE reporting period, if an investigator becomes aware of an SAE that is suspected by the investigator to be related to Study Treatment, the event should be reported to the Sponsor or its designee.

#### 9.3.3 Notification of Serious Adverse Events

In accordance with 21 CFR 312.32, the Sponsor shall notify FDA and all participating investigators in a written IND safety report of any adverse experience associated with the use of the drug that is both serious and unexpected. Reports of serious adverse events shall be made as soon as possible and in no event later than 7 calendar days if the event is a death or is life threatening and 15 calendar days for all other reportable events after the Sponsor's initial receipt of the information. Each written notification may be submitted on FDA Form 3500A or in a narrative format and shall bear prominent identification of its contents. Each written notification to FDA shall be transmitted to the FDA new product review division that has responsibility for review of the IND. In each written IND safety report, the Sponsor shall identify all safety reports previously filed with the IND concerning a similar adverse experience, and shall analyze the significance of the adverse experience in light of the previous, similar reports. The Sponsor shall also notify FDA by telephone or by facsimile transmission of all deaths regardless of causality and any unexpected fatal or lifethreatening experience associated with the use of the drug as soon as possible but in no event later than 7 calendar days after the sponsor's initial receipt of the information. Each telephone call or facsimile transmission to FDA shall be transmitted to the FDA new product review division that has responsibility for review of the IND.

Follow up information to a safety report shall be submitted as soon as the relevant information is available. If the results of a Sponsor's event investigation show that an adverse drug experience not initially determined to be reportable is, in fact, reportable, the Sponsor shall report such experience in a written safety report as soon as possible, but in no event later than 15 calendar days after the determination is made. Results

of investigations of other safety information shall be submitted, as appropriate, in an information amendment or annual report.

In the event of death, if an autopsy is performed, a copy of the report should be sent to Inovio Pharmaceuticals.

SAE reporting email: safety@inovio.com

SAE FAX transmission:

SAE Phone:

SAE MAILING ADDRESS Inovio Pharmaceuticals, Inc. 660 W. Germantown Pike Suite 110 Plymouth Meeting, PA 19462

MEDICAL MONITOR:



## 9.4 Reporting of Device Related Complaints

Any problems experienced during the treatment procedure including potential malfunctions of the CELLECTRA®-5P device, error messages displayed on the device screen following treatment or errors that occur during the treatment procedure should be reported to the Sponsor or designee immediately for evaluation. The error reporting form provided in Appendix 7 should be completed and emailed to the Sponsor at

## 9.5 Study Discontinuation

Inovio Pharmaceuticals reserves the right to discontinue the study at this site or at multiple sites for safety or administrative reasons at any time. Should the study be terminated and/or the site closed for whatever reason, all documentation and study product pertaining to the study must be returned to Inovio Pharmaceuticals or its representative.

#### 10 PUBLICATION OF RESEARCH FINDINGS

The results of this trial will be submitted for presentation and/or publication within 1 year of study completion and data availability. All data obtained, recorded in the CRF and analyzed during the course of this study are the property of the Sponsor (Inovio). Any use of these data must be approved in writing by the Sponsor. At least 60 days before any of the data or results of this study are submitted for presentation or publication, the abstract, poster, presentation, or manuscript must be sent to the Sponsor for review and approval to determine if any confidential information, trade secret, or patentable information is present. The Sponsor must approve or deny all requests for data presentation or

publication in writing within 30 days. In the event Inovio makes such objection, the researcher(s) shall refrain from making such submission for publication or presentation for a maximum of three (3) months from the date of receipt of such objection in order for patent application(s) directed to the patentable subject matter contained in the proposed publication or presentation to be filed with the United States Patent and Trademark Office and/or foreign patent office(s).

11 LIST OF ABBREVIATIONS

AE Adverse Event
BMI Body Mass Index

CEF Cytomegalovirus, Epstein Barr Virus and Influenza

CFR Code of Federal Regulations
CIB Clinical Investigator's Brochure
CIN Cervical Intraepithelial Neoplasia

CMI Cell-mediated immunity

CMR Complete Metabolic Response

CMV CytoMegalo Virus
CRF Case Report Forms
CPK Creatine Phosphokinase
CT Computed Tomography

CTL Cytotoxic T-cells
CSR Clinical Study Report

CTCAE Common Terminology Criteria for Adverse Events
DAIDS Division of Acquired Immunodeficiency Syndrome

DNA Deoxyribonucleic Acid
DLT Dose Limiting Toxicity

EBRT External Beam Radiation Therapy

ECG Electrocardiogram

ECOG Eastern Cooperative Oncology Group

EP Electroporation

ERER Events Requiring Expedited Reporting ELISA Enzyme Linked Immunosorbent Assay

ELISpot Enzyme Linked Immunosorbent Spot-forming Assay

FDA Food and Drug Administration

FDG Fluordeoxyglucose
GCP Good Clinical Practice
GLP Good Laboratory Practice
GMP Good Manufacturing Practice
HCG Human Chorionic Gonadotropin
HIV Human Immunodeficiency Virus
HLA Human Leukocyte Antigen

IC Intracavitary

**HPV** 

ICF Informed Consent Form

ICH International Conference on Harmonization

Human Papillomavirus

IFN-γ Interferon GammaIL-12 Interleukin 12IM Intramuscular

IND Investigational New Drug Application

IRB Institutional Review Board

IUD Intrauterine Device

LEEP Loop Electrosurgical Excision Procedure

| MedDRA® | Medical Dictionary for Drug Regulatory Affairs |
|---------|------------------------------------------------|
| NED | No Evidence of Disease |
| NIH | National Institutes of Health |
| NYHA | New York Heart Association |
| PBMC | Peripheral Blood Mononuclear Cells |
| PD | Progressive Disease |
| PET | Positron Emission Tomography |
| PHI | Protected Health Information |
| PFS | Progression Free Survival |
| PMR | Partial Metabolic Response |
| PRC | Participant Reminder Card |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| ROS | Review of Systems |
| RTOG | Radiation Therapy Oncology Group |
| SAE | Serious Adverse Event |
| SARS | Severe Acute Respiratory Syndrome |
| SID | Subject Identification |
| SOC | System Organ Class |
| SUV | Standard Uptake Volume |
| ULN | Upper Limit of Normal |
| VAS | Visual Analog Scale |
| WOCBP | Women of Childbearing Potential |

### 12 REFERENCES

- 1. World Health Organization. Viral cancers: Human papillomavirus. Initiative for vaccine research. Available at <<a href="http://www.who.int/vaccine\_research/diseases/viral-cancers/en/index3.html">http://www.who.int/vaccine\_research/diseases/viral-cancers/en/index3.html</a>>. Accessed January 12, 2008.
- 2. Munoz N, Bosch FX, de Sanjose S, et al. (2003) Epidemiologic classification of human papillomavirus types associated with cervical cancer. N Engl J Med. 348:518-527.
- 3. Munger K, Howley PM (2002) Human papillomavirus immortalization and transformation functions. Virus Res 89:213-228.
- 4. GLOBOCAN 2012: Estimated Cancer Incidence, Mortality and Prevalence Worldwide in 2012. Available at <a href="http://globocan.iarc.fr/Pages/fact-sheets-cancer.aspx">http://globocan.iarc.fr/Pages/fact-sheets-cancer.aspx</a>.
- 5. Centers for Disease Control and Prevention (2007) Quadrivalent human papillomavirus vaccine. Recommendations of the Advisory Committee on Immunization Practices. Morb Mort Wkly Rep. 56(RR02):1-24.
- 6. Future II Study Group (2007) Quadrivalent vaccine against human papillomavirus to prevent high-grade cervical lesions. N Engl J Med. 356:1915-27.
- 7. Centers for Disease Control and Prevention (2010) National, State, and Local Area Vaccination Coverage among Adolescents Aged 13-17 Years United States, 2009. Morb Mort Wkly Rep. 59(32):1018-1023.
- 8. Trimble C, Piantadosi S, Gravitt P, Ronnett B, Pizer E, Elko A, Wilgus B, Yutzy W, Daniel R, Shah K, Peng S, Hung C, Roden R, Wu TC, Pardoll D (2005) Spontaneous Regression of High-Grade Cervical Dysplasia: Effects of Human Papillomavirus Type and HLA Phenotype. Clin Cancer Res 11: 4717-4723.
- 9. Castle PE, Schiffman M, Wheeler CM, Solomon D (2009). Evidence for Frequent Regression of Cervical Intraepithelial Neoplasia-Grade 2. Obstet Gynecol 113:18-25
- 10. Moscicki AB, Ma Y, Wibbelsman C, Darragh T, Powers A, Farhat S, Shiboski S (2010) Rate of and Risks for Regression of Cervical Intraepithelial Neoplasia 2 in Adolescents and Young Women. Obstetrics & Gynecology. 116: 1373-1380.
- 11. Kenter GG, Welters M, Valentijn A, Lowik M, Berends-van der Meer D, Vloon A, Essahsah F, Fathers LM, Offringa R, Drijfhour JW, Wafelman AR, Oostendorp J, Fleuren GJ, van der Burg SH, Melief C (2009) Vaccination against HPV-16 Oncoproteins for Vulvar Intraepithelial Neoplasia. N Engl J Med 361: 1838-47.
- 12. Borysiewicz LK, Fiander A, Nimako M, Man S, Wilkinson GW, Westmoreland D, Evans AS, Adams M, Stacey SN, Boursnell ME, Rutherford E, Hickling JK, Inglis SC (1996) A recombinant vaccinia virus encoding human papillomavirus types 16 and 18, E6 and E7 proteins as immunotherapy for cervical cancer. Lancet 347:1523-1527.
- 13. Cui Z, Huang L. Liposome-polycation-DNA (LPD) particle as a carrier and adjuvant for protein-based vaccines: therapeutic effect against cervical cancer. Cancer Immunol Immunother 2005; 54(12):1180-1190.

- 14. Cui Z, Qiu F. Synthetic double-stranded RNA poly(I:C) as a potent peptide vaccine adjuvant: therapeutic activity against human cervical cancer in a rodent model. Cancer Immunol Immunother 2006; 55(10):1267-1279.
- 15. Jochmus I, Schafer K, Faath S, Muller M, Gissmann L. Chimeric virus-like particles of the human papillomavirus type 16 (HPV 16) as a prophylactic and therapeutic vaccine. Arch Med Res 1999; 30(4):269-274.
- 16. Liu DW, Tsao YP, Kung JT, Ding YA, Sytwu HK, Xiao X, et al. Recombinant adeno-associated virus expressing human papillomavirus type 16 E7 peptide DNA fused with heat shock protein DNA as a potential vaccine for cervical cancer. J Virol 2000; 74(6):2888-2894.
- 17. Ohlschlager P, Quetting M, Alvarez G, Durst M, Gissmann L, Kaufmann AM. Enhancement of immunogenicity of a therapeutic cervical cancer DNA-based vaccine by co-application of sequence-optimized genetic adjuvants. Int J Cancer 2009; 125(1):189-198.
- 18. Welters MJ, Kenter GG, Piersma SJ, Vloon AP, Lowik MJ, Berends-van der Meer DM, et al. Induction of tumor-specific CD4+ and CD8+ T-cell immunity in cervical cancer patients by a human papillomavirus type 16 E6 and E7 long peptides vaccine. Clin Cancer Res 2008; 14(1):178-187.
- 19. Chi KH, Liu SJ, Li CP, Kuo HP, Wang YS, Chao Y et al 2005 Combination of conformal radiotherapy and intratumoral injection of adoptive dendritic cell immunotherapy in refractory hepatoma. J Immunother 28:p.129–35
- 20. Gulley JL, Arlen PM, Bastian A, Morin S, Marte J, Beetham P et al 2005 Combining a recombinant cancer vaccine with standard definitive radiotherapy in patients with localized prostate cancer. Clin Cancer Res 11:3353–3362
- 21. Reits EA, Hodge JW, Herberts CA, Groothuis TA, Chakraborty M, Wansley EK et al (2006) Radiation modulates the peptide repertoire, enhances MHC class I expression, and induces successful antitumor immunotherapy. J Exp Med 203:1259–1271
- 22. Gaugler MH, Squiban C, van der Meeren A, Bertho JM, Vandamme M, Mouthon MA (1997) Late and persistent up-regulation of intercellular adhesion molecule-1 (ICAM-1) expression by ionizing radiation in human endothelial cells in vitro. Int J Radiat Biol 72:201–209
- 23. Garnett CT, Palena C, Chakraborty M, Tsang KY, Schlom J, Hodge JW (2004) Sublethal irradiation of human tumor cells modulates phenotype resulting in enhanced killing by cytotoxic T lymphocytes. Cancer Res 64:p.7985–94.
- 24. Gelbard A, Garnett CT, Abrams SI, Patel V, Gutkind JS, Palena C et al (2006) Combination chemotherapy and radiation of human squamous cell carcinoma of the head and neck augments CTL-mediated lysis. Clin Cancer Res 12: p.1897–1905.
- 25. Matsuzaki I, Suzuki H, Kitamura M, Minamiya Y, Kawai H, Ogawa J (2000) Cisplatin induces fas expression in esophageal cancer cell lines and enhanced cytotoxicity in combination with LAK cells. Oncology 59: p.336–343
- 26. Tseng CW, Trimble C, Zeng Q, Monie A, Alvarez RD, Huh WK, Hoory T, Wang MC, Hung CF, Wu TC. Cancer Immunol Immunotherapy. 2009 May;58(5):737-48. doi: 10.1007/s00262-008-0596-0. Epub 2008 Sep 25. Low-dose radiation enhances therapeutic HPV DNA vaccination in tumor-bearing hosts.

- 27. Martin T, Parker SE, Hedstrom R, Le T, Hoffman SL, Norman J, Hobart P, Lew D (1999) Plasmid DNA malaria vaccine: the potential for genomic integration after intramuscular injection. Hum Gene Ther. 10:759-768
- 28. Nichols WW, Ledwith BJ, Manam SV, Troilo PJ (1995) Potential DNA vaccine integration into host cell genome. Ann N Y Acad Sci. 772:30-39
- 29. Chattergoon M, Boyer J, Weiner DB (1997) Genetic immunization: a new era in vaccines and immune therapeutics. FASEB J 11:753-763
- 30. Yan J, Reichenbach DK, Corbitt N, Hokey DA, Ramanathan MP, McKinney KA, Weiner DB, Sewell D (2009) Induction of antitumor immunity *in vivo* following delivery of a novel HPV-16 DNA vaccine encoding an E6/E7 fusion antigen. Vaccine 27: 431-440.
- 31. Davis HL, Whalen RG, Demeneix BA (1993) Direct gene transfer into skeletal muscle in vivo: factors affecting efficiency of transfer and stability of expression. Hum Gene Ther. 4:151-9.
- 32. Tripathy SK, Svensson EC, Black HB, Godwasser E, Margalith M, Hobart PM, Leiden JM (1996) Long-term expression of erythropoietin in the systemic circulatin of mice after intramuscular injection of a plasmid DNA vector. Proc Nat Acad Sci USA. 93:10876-80.
- 33. Prud'homme GJ, Glinka Y, Khan AS, Draghia-Akli R (2006) Electroporation-enhanced nonviral gene transfer for the prevention or treatment of immunological, endocrine and neoplastic diseases. Curr Gene Ther. 6:243-73.
- 34. Prud'homme GJ, Draghia-Akli R, Wang Q (2007) Plasmid-based gene therapy of diabetes mellitus. Gene Ther. 14:553-564.
- 35. Khan AS, Pope MA, Draghia-Akli R (2005) Highly efficient constant-current electroporation increases in vivo plasmid expression. DNA & Cell Biology. 24:810-18.
- 36. Diehl M, Lee J, Daniels S, Tebas P, Khan A, Giffear M, Sardesai N, Bagarazzi M, Tolerability of intramuscular and intradermal delivery by CELLECTRA® adaptive constant current electroporation device in healthy volunteers. Human Vaccines & Immunotherapeutics 9:10, 1–7; October 2013.
- 37. Bagarazzi M, Yan J, Morrow M, Shen X, Parker R, Lee J, Giffear M, Pankhong P, Khan S, Broderick K, Knott C, Lin F, Boyer J, Draghia-Akli R, White C, Kim J, Weiner D, Sardesai N, Immunotherapy Against HPV16/18 Generates Potent TH1 and Cytotoxic Cellular Immune Response. Science Translational Medicine 10 October 2012 Vol 4 Issue 155 155ra138.
- 38. Felix, J., et al., The significance of positive margins in loop electrosurgical cone biopsies. Obstet Gynecol, 1994. 84(6): p. 996-1000.
- 39. Ferris, D., et al., Electrosurgical loop excision of the cervical transformation zone: the experience of family physicians. Journal of Family Practice, 1995. 41(4): p. 337-44.
- 40. Kalams SA, Parker S, Jin X, Elizaga M, Metch B, Wang M, *et al.* Safety and immunogenicity of an HIV-1 gag DNA vaccine with or without IL-12 and/or IL-15 plasmid cytokine adjuvant in healthy, HIV-1 uninfected adults. *PLoS One* 2012; 7(1):e29231.
- 41. Quinn MA, Benedet JL, Odicino F, Maisonneuve P, Beller U, Creasman WT, Heintz AP, Ngan HY, Pecorelli S. Int J Gynaecol Obstet. 2006 Nov;95 Suppl

Date: 27 April 2016 v 2.1

- 1:S43-103. Carcinoma of the cervix uteri. FIGO 26th Annual Report on the Results of Treatment in Gynecological Cancer.
- 42. Perez CA, Grigsby PW, Nene SM, Camel HM, Galakatos A, Kao MS, Lockett MA. Cancer. Effect of tumor size on the prognosis of carcinoma of the uterine cervix treated with irradiation alone. 1992 Jun 1;69(11):2796-806.
- 43. Morley GW, Seski JC. Radical pelvic surgery versus radiation therapy for stage I carcinoma of the cervix (exclusive of microinvasion). Am J Obstet Gynecol, 126 (7) (1976), pp. 785–798.
- 44. Hopkins MP, Morley GW. Radical hysterectomy versus radiation therapy for stage IB squamous cell cancer of the cervix. Cancer, 68 (2) (1991), pp. 272–277.
- 45. Estape RE, Angioli R, Madrigal M, Janicek M, Gomez C, Penalver M, Averette H. Close vaginal margins as a prognostic factor after radical hysterectomy. Gynecol Oncol, 68 (3) (1998), pp. 229–232.
- 46. Perez CA, Grigsby PW, Camel HM, Galakatos AE, Mutch D, Lockett MA.. Irradiation alone or combined with surgery in stage IB, IIA, and IIB carcinoma of uterine cervix: update of a nonrandomized comparison. Int J Radiat Oncol Biol Phys, 31 (1995), pp. 703–716.
- 47. Rose PG, Bundy BN, Watkins J, et al: Concurrent cisplatin-based chemotherapy and radiotherapy for locally advanced cervical cancer. N Engl J Med 340:1144-1153, 1999.
- 48. Grigsby PW, Heydon K, Mutch DG, Kim RY, Eifel P. Long-term follow-up of RTOG 92-10: cervical cancer with positive para-aortic lymph nodes. Int J Radiat Oncol Biol Phys. 2001 Nov 15;51(4):982-7.
- 49. Morris M, Eifel PJ, Lu J, et al: Pelvic radiation with concurrent chemotherapy compared with pelvic and paraaortic radiation for high-risk cervical cancer. N Engl J Med 340:1137-1143, 1999
- 50. Sheets RL, Stein J, Manetz TS, Duffy C, Nason M, Andrews C, et al. Biodistribution of DNA plasmid vaccines against HIV-1, Ebola, Severe Acute Respiratory Syndrome, or West Nile virus is similar, without integration, despite differing plasmid backbones or gene inserts. Toxicol Sci 2006; 91(2):610-619.
- 51. Sheets RL, Stein J, Manetz TS, Andrews C, Bailer R, Rathmann J, et al. Toxicological safety evaluation of DNA plasmid vaccines against HIV-1, Ebola, Severe Acute Respiratory Syndrome, or West Nile virus is similar despite differing plasmid backbones or gene-inserts. Toxicol Sci 2006; 91(2):620-630.
- 52. Janetzki S, Panageas KS, Ben-Porat L, Boyer J, Britten CM, Clay TM, Kalos M, Maecker HT, Romero P, Yuan J, Kast WM, Hoos A; Elispot Proficiency Panel of the CVC Immune Assay Working Group. Results and harmonization guidelines from two large-scale international Elispot proficiency panels conducted by the Cancer Vaccine Consortium (CVC/SVI). Cancer Immunol Immunother. 2008 Mar;57(3):303-15. Epub 2007 Aug 25.
- 53. Weber WA, Ott K, Becker K, et al. (2001) Prediction of response to preoperative chemotherapy in adenocarcinomas of the esophagogastric junction by metabolic imaging. J Clin Oncol. 19(12):3058-3065.
- 54. Ott K, Fink U, Becker K, et al. (2003) Prediction of response to preoperative chemotherapy in gastric carcinoma by metabolic imaging: results of a prospective trial. J Clin Oncol. 21(24):4604-4610.
- 55. Weber WA, Petersen V, Schmidt B, et al. (2003) Positron emission tomography in non-small-cell lung cancer: prediction of response to chemotherapy by quantitative assessment of glucose use. J Clin Oncol. 21(14):2651-2657.
- 56. Brun E, Kjellen E, Tennvall J, et al. (2002) FDG PET studies during treatment: prediction of therapy outcome in head and neck squamous cell carcinoma. Head Neck. 24(2):127-135.
- 57. Schwarz JK, Siegel BA, Dehdashti F, Grigsby PW. (2007) Association of Posttherapy Positron Emission Tomography With Tumor Response and Survival in Cervical Carcinoma. JAMA. 298(19):2289-2295.
- 58. Zhao, Qianying, et al. (2013) Prognostic Value of Fluorine-18-Fluorodeoxyglucose Positron Emission Tomography or PET-Computed Tomography in Cervical Cancer: A Meta-Analysis. International journal of gynecological cancer.
- 59. Postow MA, Callahan MK, Barker CA, Yamada Y, Yuan J, et al. (2012) Immunologic correlates of the abscopal effect in a patient with melanoma. N. Engl. J. Med. 366:925–31.
- 60. Prise KM, O'Sullivan JM. (2009) Radiation-induced bystander signalling in cancer therapy. Nat. Rev. Cancer, 9: 351–360.
- 61. Lee Y, Auh SL, Wang Y et al. Therapeutic effects of ablative radiation on local tumor require CD8+ T cells: changing strategies for cancer treatment. Blood 2009;114:589-95.
- 62. Meng, Y., Beckett, M. A., Liang, H., Mauceri, H. J., van Rooijen, N., Cohen, K. S., & Weichselbaum, R. R. (2010). Blockade of tumor necrosis factor α signaling in tumor-associated macrophages as a radiosensitizing strategy. Cancer research, 70(4), 1534-1543.
- 63. Seung SK, Curti BD, Crittenden M et al. Phase 1 study of stereotactic body radiotherapy and interleukin-2--tumor and immunological responses. Sci Transl Med 2012;4:137ra74.
- 64. Grigsby PW, Siegel BA, Dehdashti F, Rader J, Zoberi I. Posttherapy [18F] fluorodeoxyglucose positron emission tomography in carcinoma of the cervix: response and outcome. J Clin Oncol. 2004 Jun 1;22(11):2167-71.
- 65. Grigsby PW, Siegel BA, Dehdashti F, Mutch DG. Posttherapy surveillance monitoring of cervical cancer by FDG-PET. Int J Radiat Oncol Biol Phys. 2003 Mar 15;55(4):907-13.
- 66. Schwarz JK, Siegel BA, Dehdashti F, Grigsby PW. Metabolic response on posttherapy FDG-PET predicts patterns of failure after radiotherapy for cervical cancer. Int J Radiat Oncol Biol Phys. 2012 May 1;83(1):185-90. doi: 10.1016/j.ijrobp.2011.05.053. Epub 2011 Oct 17.

# 13 APPENDICES

# 13.1 Appendix 1: Subject Identification Fax Form

| SCREENING NUMBER: | |
|-----------------------------------------------|----------------------|
| GENDER: | |
| Date of Birth: | |
| Screening Date: | |
| Anticipated Date of Immunotherapy Dose: | |
| Allocation Number (to be completed by Inovio) | Allocation Number: |
| | INO initials: |
| COMMENTS BOX: | |
| SITE PERSONNEL REPORTING: | DATE REPORTED/FAXED: |

# 13.2 Appendix 2: ECOG Performance Status

| ECOG PERFORMANCE STATUS* | |
|---|---|
| Grade | ECOG |
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair |
| 5 | Dead |

<sup>\*</sup> As published in Am. J. Clin. Oncol.:

Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982.

# 13.3 Appendix 3: Standard Chemoradiation Guidelines

Below are standard guidelines for chemoradiation in this patient population. It is highly suggested these guidelines be followed.

#### I. Standard therapy

a. Concurrent chemoradiotherapy

# II. Chemotherapy

- a. Cisplatin
- I. Source and Formulation: Cisplatin is commercially available from Bristol-Myers Oncology and from Pfizer as a dry powder supplied in 10 mg and 50 mg vials, and in aqueous solution in 50 mg and 100 mg vials with 100 mg mannitol and 90 mg sodium chloride; 10 mg/vial. The 10 mg and 50 mg vials should be reconstituted with 10 mL or 50 mL sterile water for injection USP, respectively. Each mL of the resulting solution will contain 1 mg of cisplatin. Reconstitution of powder results in a clear colorless solution when completed as recommended. NOTE: Aluminum reacts with cisplatin causing precipitation formation and loss of potency; therefore, needles or intravenous sets containing aluminum parts that may come in contact with the drug must not be used for the preparation or administration of cisplatin.
- II. Administration: Patients will be pre-hydrated per institutional guidelines. Cisplatin will be dissolved at a concentration of 1 mL of sterile water/mg of drug, and the solution will be administered intravenously over 45-60 minutes. Supportive treatment will be given according to institutional policy.
- III. Storage and Stability: Store at 15° to 20°C. Unopened vials of dry powder are stable for the lot life indicated on the package when stored at room temperature. The aqueous solution should be stored at room temperature and protected from light. The reconstituted solution is stable for 20 hours at room temperature. Do not refrigerate. The cisplatin remaining in the amber vial following initial entry is stable for 28 days protected from light or for 7 days under fluorescent room light. NOTE: Once reconstituted, the solution should be kept at room temperature. If the reconstituted solution is refrigerated, a precipitate will form.
- IV. Adverse Events: Incidence rates of adverse events associated with cisplatin are provided in the product package insert. The following events are expected with the administration of cisplatin:
  - a. Nephrotoxicity: Dose-related and cumulative renal insufficiency is the major dose-limiting adverse events of cisplatin. Renal adverse events have been noted in 28-36% of patients treated with a single dose of 50 mg/m2. It is first noted in the second week after a dose and is manifested as elevated BUN, creatinine, and serum uric acid, or as a decrease in creatinine clearance. Because renal adverse events become more prolonged and severe with repeated

- courses of cisplatin, renal function must return to normal before another dose can be given.
- b. Ototoxicity: Ototoxicity has been observed in up to 31% of patients treated with a single dose of cisplatin 50 mg/m2. It is manifested by tinnitus and/or hearing loss in the high frequency range. Deafness has been reported rarely.
- c. Hematologic Toxicity: Myelosuppression occurs in 25-30% of patients treated with cisplatin. Nadirs in circulating platelets and leukocytes occur between Days 18 and 23 with most patients recovering by Day 39. Thrombocytopenia, anemia, neutropenia, and fever are also possible adverse events.
- d. Gastrointestinal Toxicity: Marked nausea and vomiting occur in almost all patients treated with cisplatin. Diarrhea and anorexia have also been reported.
- e. Neurotoxicity: Neurotoxicity usually characterized by peripheral neuropathies, has been reported. Neuropathy usually occurs after prolonged therapy (4 to 7 months); however, symptoms have been reported after a single dose. Muscle cramps, loss of taste, seizures, autonomic neuropathy, dorsal column myelopathy, and Lhermitte's sign have also been reported.
- f. Ocular Toxicity: Optic neuritis, papilledema, and cerebral blindness have been reported infrequently in patients receiving standard recommended doses of cisplatin. Blurred vision and altered color perception have been reported after the use of regimens with higher doses of cisplatin or greater dose frequency than those recommended in the package insert.
- g. Anaphylactic-like Reactions: Anaphylactic-like reactions have occasionally been reported in patients previously exposed to cisplatin. Symptoms include facial edema, wheezing, tachycardia, and hypotension.
- h. Hepatotoxicity: Transient elevations in liver enzymes, especially SGOT (AST), and bilirubin, have been reported.
- i. Other Toxicities: Other infrequent toxicities that have been reported include cardiac abnormalities, hiccups, elevated serum amylase, rash, alopecia, malaise, and asthenia. Rare cases of local soft tissue adverse events have occurred.
- V. Mechanism of Action: Primarily causes inhibition of DNA synthesis and, to a lesser degree, inhibition of RNA and protein; it has not been shown to be cell cycle specific.
- VI. Pharmaceutical data: Cisplatin (cis-diamminedichloroplatinum II) has the empiric formula N2CL2 PtH6. It is a planar inorganic compound with a molecular weight of 300; soluble in water at a concentration of 1 mg/mL. The (II) nomenclature denotes the active valence state of the platinum. The interatomic distance of the chlorides is 3.3A, which is different from the 5-7A interatomic distance of the classic alkylating agents. Only the cis-isomer is therapeutically active.

- VII. Supply: This drug is commercially available.
- VIII. Duration of administration: Cisplatin 40 mg/m² (80 mg max) should be administered once weekly during external beam RT (5 cycles only). It is recommended that cisplatin be started on day 1 of external beam RT but it is acceptable to give cisplatin on days 1, 2, or 3 of external beam RT. Dose modifications and indications for holding cisplatin are provided below.

#### IX. Dose Modification

- a. Chemotherapy should be held for:
- ANC  $< 500 \text{ /mm}^3$ .
- Platelets  $< 50,000/\text{mm}^3$ .
- Febrile neutropenia or bleeding.
- Persistent (>24 hours) grade 3 or 4 nausea and vomiting.
- Renal Failure (creatinine > 2.0 mg% or creatinine clearance < 50 ml/min).
- b. Cisplatin can be resumed at a dose of 30 mg/m² (60 mg max) after the resolution of:
- Persistent (>24 hours) grade 3 or 4 nausea and vomiting.
- Renal Failure (creatinine > 2.0 mg% or creatinine clearance < 50 ml/min).

#### **III.** Radiation Therapy

Patients should receive pelvic radiation therapy in combination with cisplatin infusion given on a weekly basis for six weeks. The last dose can be given during parametrial boost.

Radiation therapy should be administered to the pelvis with external beam and intracavitary techniques. Radiation therapy may also be administered to the para-aortic nodal chain as clinically indicated when there is clinical and/or imaging evidence of nodal disease in the high common iliac or para-aortic nodal chain. Radiation therapy **must** be completed within 10 weeks of its initiation.

#### **a.** Physical Factors

External beam radiation sources will be linear accelerators which produce megavoltage energy radiation beams. SAD (source-axis distance) 100 cm is required. Low-Dose-Rate (LDR) intracavitary radiation may be delivered by Cesium-137 sources. High-Dose-Rate (HDR) may also be used using an Iridium-192 source.

#### **b.** Simulation and Localization

- i. Simulation should be done in the supine position.
- ii. Recommended contrast and markers are intravenous contrast unless medically contraindicated, oral contrast, bladder contrast, rectal contrast, and a radio-opaque cervical marker at the apex of the vagina. Implanted fiducials are optional.
- iii. A gyne swab with CT wire at the tip should be placed into into the vagina

- iv. A foley catheter should be placed for simulation with both an empty and full bladder. Full bladder is recommend to be achieved through injection 120 cc of 90cc bacteriostatic water and 30 cc of conray through foley into bladder.
- v. Patient should be scanned with both full and empty bladder. Full and empty bladder CT scans should be fused.
- vi. Immobilization should be achieved with custom alpha cradles.
- vii. Imaging should include CT simulation using 2-5mm slice thickness from T10 to 5cm below the ischial tuberosities, or to include the maximal extent of disease.
- viii. Isocenter placement is per the discretion of the treating physicians
- ix. Localization films taken on the simulator and/or treatment machine are necessary in all patients. Polaroid or digital pictures of all treatment portals with the patient in the treatment position are recommended.

# Treatment Plan, Dose Specification and Distribution

- i. Depending on the FIGO stage and radiographic extent of disease, patients should receive radiation therapy to the pelvis, cervix, gross lymph nodes, and if indicated, the paraortic nodal chain.
- ii. The volume irradiated should include the totality of the gross disease locally and regionally, as visualized by CT, PET or MRI scanning, the whole uterus, paracervical, parametrial and uterosacral ligaments as well as the areas of the obturator, hypogastric, external and internal iliac lymph nodes. A margin of 2-3 cm should be given around the gross disease and 1.5-2 cm around involved lymph nodes.
- iii. Patients treated to the whole pelvis +/- paraaortic chain should receive a total dose of 4500 cGy in 25 fractions at 180 cGy/fx, using a four field technique or intensity modulated radiation therapy (IMRT) throughout the entire treatment with all fields treated each day. Gross nodal disease should be treated with either a sequential boost or simultaneous integrated boost per the treating physician and as determined by proximity of organs at risk.
- iv. If overall treatment time for external pelvic RT exceeds 50 days, then reason for the delay must be documented.

#### c. Dose Specification

- 1. Fractionation: Conventional fractionation should consist of one fraction per day, total five fractions per week.
- 2. The pelvis and, if indicated, the para-aortic nodal chain, should be treated at a dose per fraction of 180 cGy per day.
- 3. Sequential or simultaneous integrated boost may be delivered to a maximum of 65Gy in 1.8-2.5Gy per fraction, while maintaining normal tissue constraints.
- 4. Parametrial boost should be delivered sequentially after pelvic/para-aortic radiation therapy to a maximum dose of 65Gy to the sidewall. Point B may be used as the calculation point dose site. The superior border should be reduced to include the true pelvis only as defined as 1cm above the inferior aspect of the sacroiliac joint.

#### **d.** Target Delineation

1. General

Pelvic MRI and/or PET fusion with the simulation scan is recommended to aid target delineation. Fusion should be optimized to match the MRI / PET scan to the treatment position. The Gross Tumor Volume (GTV) and Clinical Target Volume (CTV) and normal tissues will be contoured on all CT slices in which the structures exist. The definition of all volumes will be in accordance with the 1993 ICRU Report #50: Prescribing, Recording and Reporting Photon Beam Therapy (<a href="http://www.icru.org/home/reports/prescribing-recording-and-reporting-photon-beam-therapy-report-50">http://www.icru.org/home/reports/prescribing-recording-and-reporting-photon-beam-therapy-report-50</a>).

#### 2. GTV Delineation

The GTV is defined as all known gross disease determined from radiographic studies, clinical information, physical examination, endoscopic examination, and biopsy results.

#### 3. CTV Delineation

The CTV is defined as the gross tumor plus areas containing potential microscopic disease, including the cervix, uterus (if present), the superior third of the vagina (or half of the vagina, if clinically involved), the parametria, and the regional lymph nodes. CTV delineation should follow reported consensus guidelines [Small W, Mell LK, Creutzberg C, et al. Consensus recommendations for intensity modulated radiation therapy planning for post-operative pelvic radiotherapy in endometrial and cervical cancer. Int J Radiat Oncol Biol Phys. 2008;71:428-34, <a href="http://www.ncbi.nlm.nih.gov/pubmed/18037584">http://www.ncbi.nlm.nih.gov/pubmed/18037584</a> and Lim K, Small W, Portelance L, et al. Consensus guidelines for delineation of clinical target volume for intensity-modulated pelvic radiotherapy for the definitive treatment of cervix cancer <a href="https://www.redjournal.org/article/S0360-3016(09)03587-1/abstract">htt J Radiat Oncol Biol Phys. 2009, <a href="https://www.redjournal.org/article/S0360-3016(09)03587-1/abstract">https://www.redjournal.org/article/S0360-3016(09)03587-1/abstract</a>, accessed March 25, 2014].

For patients with distal one third vaginal involvement, the inguinal nodes should be contoured continuously from the external iliac nodes to 2 cm caudad to the saphenous/femoral junction. For contouring guidelines for patients with inguinal nodal involvement, refer to atlases used to treat anal carcinoma [Myerson RJ, Garofalo MC, et al. Elective clinical target volumes for conformal therapy in anorectal cancer: a radiation therapy oncology group consensus panel contouring atlas. *Int J Radiat Oncol Biol Phys.* 2009;74:824-30, <a href="http://www.ncbi.nlm.nih.gov/pubmed/19117696">http://www.ncbi.nlm.nih.gov/pubmed/19117696</a>, accessed March 25, 2014].

#### 4. PTV Delineation

The Planning Target Volume (PTV) will add a 7-15mm margin around CTV to compensate for treatment setup and internal organ motion. The PTV should be manually or automatically trimmed up to 3 mm from the skin surface, if necessary, to spare skin, provided that the CTV is still included entirely within the PTV.

# e. Normal Tissue Delineation

#### General

Normal tissues should be contoured on the simulation scan. The tissue within the skin surface and outside all other critical normal structures and the PTV is

designated as unspecified tissue. Critical normal tissues for IMRT optimization will consist of the bowel, bladder, rectum, and bone marrow. Femoral heads will be contoured to determine delivered dose but will not be used as a planning constraint.

#### Bowel

The bowel should be contoured beginning from the axial slice situated 1 cm superior to the superior-most slice containing PTV (if bowel is not present at this level, the bowel contour will start from its most superior extent), and will continue to its most inferior extent in the pelvis. Individual loops of bowel should not be contoured separately. Rectum should be contoured separately from bowel.

#### Rectum

The outer rectal wall should be contoured and will be defined from the level of the sigmoid flexure to the anus.

#### Bladder

The outer bladder wall should be contoured, treating the organ as a solid continuous structure.

#### Bone Marrow

The outer bone contour should be delineated and filled in, treating the bone marrow as a solid continuous structure. The regions contoured should include the os coxae, L5 vertebral body, entire sacrum, acetabulae, and proximal femora. The superior extent of the bone marrow contour should be at the level of the superior border of L5 or the iliac crest, whichever is more superior. When the para-aortic nodal chain is treated, the vertebral bodies should be contoured to T12 or the most cephalad vertebral level being treated. The caudal-most extent of the bone marrow contour should be at the level of the ischial tuberosities.

#### Femoral Heads

The outer contours of the femoral heads will be delineated and filled in, treating each as a solid continuous structure. Do not include the femoral neck.

# f. Treatment Planning

#### Field Design

- a. Conventional RT consists of a 4-field "box" arrangement using opposed AP/PA and lateral fields. For conventional RT, it is permissible to use bone landmarks to draw field borders or to use 3-D planning with explicit targeting as outlined above, using customized blocking to encompass the PTV. If bone landmarks are used, use the following portals:
  - Superior border: L4-5
  - Lateral border: 1-2 cm lateral to the border of the true pelvis
  - Inferior border: Obturator foramen or 4 cm inferior to vaginal cuff, whichever is lower
  - Anterior border: line from pubic symphysis to 1 cm anterior to common iliac nodes at L4-5

- Posterior border: draw border posterior to or splitting the sacrum from S1-S4
- Custom blocking to shield femoral heads. Do not block the obturator foramen or within 1 cm of the common iliac nodes
- b. Intensity-modulated radiation therapy plans may include static field arrangements (e.g. 5-9 fields).

#### Target coverage requirements

- The 99% prescription isodose surface will encompass  $\geq$  90% of the PTV.
- > 99% of the PTV will receive > 90% of the prescription dose.
- $\geq$  97% of the PTV will receive  $\geq$  97% of the prescription dose.
- < 1% of PTV will receive > 115% of the prescription dose.
- < 10% of the PTV will receive  $\ge 110\%$  of the prescription dose.
- Dose maximum should occur within the PTV

#### Normal tissue planning goals for IMRT (soft constraints):

- Bowel: volume receiving >45 Gy  $(V_{45}) \le 200$  cc;  $V_{40} < 30\%$ ; maximum dose < 50 Gy
- Rectum:  $V_{45} < 50\%$ ;  $V_{30} < 60\%$ ; maximum dose < 50 Gy
- Bone Marrow:  $V_{10} < 80\%$ ;  $V_{20} < 66\%$
- Bladder:  $V_{45} < 50\%$ ; maximum dose < 50 Gy
- Femoral Head: V<sub>30</sub> < 15%; maximum dose < 50 Gy

# Normal tissue requirements for IMRT (hard constraints):

- Bowel: volume receiving >45 Gy  $(V_{45}) \le 250$  cc; maximum dose < 110%
- Rectum: maximum dose < 110%
- Bone Marrow:  $V_{10} < 90\%$ ;  $V_{20} < 75\%$
- Bladder: maximum dose < 110%
- Femoral Head: maximum dose < 110%

#### Heterogeneity corrections: Heterogeneity corrections should be applied

#### g. External Beam Treatment Modification

Treatment should be held for ANC  $<500/\text{mm}^3$ , platelets  $<20,000~\text{mm}^3$ , febrile neutropenia, or uncontrolled bleeding. No dose reductions are allowed. Treatment will be resumed upon resolution of neutropenia (ANC  $\ge 500/\text{mm}^3$ ), thrombocytopenia (platelets  $\ge 20,000~\text{mm}^3$ ), and febrile neutropenia (temperature <38.0~°C).

#### **h.** Setup Verification

Skeletal imaging (e.g., electronic portal MV or kV imaging or CBCT) should be performed at least weekly to verify setup accuracy. For patients treated with conventional techniques, MV portal verification is recommended at least weekly. Daily on-line imaging (image-guided radiotherapy (IGRT)) is allowed but not required.

#### i. Intracavitary Brachytherapy

The treating physician should select the dose rate to be used for brachytherapy, either HDR or LDR. Orthogonal x-rays, CT, and/or MRI may be used for brachytherapy

**HPV-004** 

Inovio Pharmaceuticals, Inc.

#### planning

# j. Low Dose Rate (LDR) Brachytherapy

Following the completion of external beam RT, the patient will receive 3500-4000 cGy to Point A by intracavitary implant with Cesium-137. The patient may receive this in one or two applications at the discretion of the radiation oncologist. The first insertion should be performed promptly upon completion of external beam irradiation. If two implants are contemplated, the second implant should be completed within three weeks of the completion of external beam irradiation (with total radiation treatment time not to exceed 8 weeks).

# Normal Tissue Constraints

Maximum allowable cumulative doses (external beam + brachytherapy) to normal tissues are (in EQD2,  $\alpha/\beta=3$ ,  $T_{1/2}=1.5$  hours): bladder (ICRU reference point), 85 Gy; rectum (ICRU reference point), 80 Gy; vaginal surface (reference point), 135 Gy. If CT is used for planning it is recommended to keep the maximum bowel dose < 25% of the brachytherapy prescription dose. Every attempt should be made to deliver the full prescription dose, even if the late responding tissues receive a slightly higher dose.

**k.** High Dose Rate (HDR) Brachytherapy -Iridium-192 as the source for HDR brachytherapy.

HDR Schema -

Dose should be prescribed to point A. Permissible dose/fractionation schemes are:

- 5.5 Gy x 6 fractions
- 5.5 Gy x 5 fractions
- 6.0 Gy x 5 fractions
- 6.0 Gy x 6 fractions
- 7.0 Gy x 3 fractions
- 7.0 Gy x 4 fractions
- 7.0 Gy x 5 fractions
- 7.5 Gy x 3 fractions

In general, insertions should be separated by a minimum of 48 hours and no more than 2 insertions should be performed per week. HDR brachytherapy should start at week four of chemoradiation. When HDR brachytherapy begins, at least one insertion should be performed per week with no external beam therapy given on the day of the insertion.

#### Instruments

It is recommended that tandem and ovoids or tandem and ring be used for brachytherapy. A tandem and cylinder or interstitial system is also permissible.

#### Determination of Normal Tissue Tolerance

Maximum allowable cumulative doses (external beam + brachytherapy) to normal tissues are (in EQD2,  $\alpha/\beta=3$ ,  $T_{1/2}=1.5$  hours): bladder (ICRU reference point), 80 Gy; rectum (ICRU reference point), 75 Gy. It is recommended that the rectum and bladder for each fraction receive less than or equal to 70% and 80% of the point A

dose, respectively, if feasible. If CT is used for planning it is recommended to keep the maximum bowel dose < 25% of the brachytherapy prescription dose. Every attempt should be made to deliver the full prescription dose, even if the late responding tissues receive a slightly higher dose.

#### Intracavitary Radiotherapy Dosimetry

The dose to points A and B, the rectal reference point dose, bladder reference point dose, and vaginal surface reference point dose, and central axis isodose curve should be calculated and documented.

Point A: Measure 2 cm along the intrauterine tandem from the cervical os or flange of the tandem and 2 cm laterally in the plane of the intracavitary system.

Point B: Measure 5 cm lateral from a point 2 cm vertically superior to the cervical os or flange of the central tandem along the patients' midline.

Bladder Dose: Calculated at the center (in the superior-inferior plane on AP view) of a contrast-filled balloon of a Foley catheter and closest to the applicator system on a lateral view, as defined by ICRU 38.

Rectal dose: In accordance with ICRU 38, mark the point 0.5 cm posterior to the vaginal surface (as demarcated by the opaque packing) at the midpoint of the applicator system or at the level of the flange if no ovoids are used.

#### Parametrial Boost to Involved Parametrium

All patients with initial parametrial involvement should be considered for a parametrial boost. The radiation oncologist should choose the dose and beam and beam energy to be used to the involved parametrium based on bulk of parametrial disease at presentation, as well as the contribution from intracavitary brachytherapy to the external beam, in order to deliver a minimum cumulative (external beam and brachytherapy) dose to the mid-parametrium, or Point B dose, of 5500 cGy (maximum of 6000 cGy) when using LDR intracavitary brachytherapy or a minimum of 5000 cGy (maximum of 5500 cGy) when using HDR intracavitary brachytherapy. Patients with parametrial involvement at the time of brachytherapy implant should receive a cumulative dose to Point B of no less than 6000 cGy (maximum of 7000 cGy) when using LDR brachytherapy or a minimum of 5500 cGy (maximum of 6500 cGy) with HDR implant.

Maximum parametrial boost shall be 1000 cGy at 180 cGy per fraction given AP/PA daily to mid-plane if unilateral or bilateral parametrial boost is used. The prescription point should be at the center of the unblocked portion of the field. The parametrial boost should be delivered if possible between implant 1 & 2 or immediately after implant 1 if only one implant is used.

The total elapsed time for completion of external whole pelvis, intracavitary RT, and parametrial RT shall not exceed eight to ten weeks.

#### **l.** Radiation Adverse Events

Risks and side effects related to radiation therapy include:

Likely (more than 10%)

• Redness and skin irritation in the treatment area that may result in bleeding and/or infection, which may require hospitalization

- Loss of pubic hair in the treated area, usually temporary
- Tiredness
- Nausea and/or vomiting
- Sterility (inability to bear children) in fertile women
- Sterility (inability to produce children) in men

#### Less Likely (3-9%)

- Diarrhea
- Sores and bleeding from the bowel (these side effects may occur well after treatment and be serious enough to require surgery)
- Narrowing and dryness of the vagina (birth canal) and genital area with painful or difficult intercourse and possibly bleeding
- Development of extra tissue (fibrosis) in the anal canal, which may result in decreased function
- Long-term dryness of the skin
- Inability to have or keep an erection (impotency)
- Hip, pelvic, or sacral fracture
- Build up of fluid in ankles, feet, and/or legs

#### Rare, but serious (less than 2%)

- Narrowing or blockage of the bowel (these side effects may occur well after treatment and be serious enough to require surgery)
- Blockage of the urinary tubes
- Development of an abnormal path or connection between organs (fistulae)
- Skin damage (tissue death), which may result in surgery
- Narrowing of or persistent bleeding in the vagina (birth canal), which may result in surgery

13.4 Appendix 4: Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 dated June 14, 2010

# Common Terminology Criteria for Adverse Events (CTCAE)

# Version 4.0

Published: May 28, 2009 (v4.03: June 14, 2010)

#### U.S.DEPARTMENT OF HEALTH AND HUMAN SERVICES

National Institutes of Health National Cancer Institute

# Common Terminology Criteria for Adverse Events v4.0 (CTCAE)

Publish Date: May 28, 2009

#### **Quick Reference**

The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.

#### **Components and Organization**

#### SOC

System Organ Class, the highest level of the MedDRA hierarchy, is identified by anatomical or physiological system, etiology, or purpose (e.g., SOC Investigations for laboratory test results). CTCAE terms are grouped by MedDRA Primary SOCs. Within each SOC, AEs are listed and accompanied by descriptions of severity (Grade).

#### **CTCAE Terms**

An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may <u>not</u> be considered related to the medical treatment or procedure. An AE is a term that is a unique representation of a specific event used for medical documentation and scientific analyses. Each CTCAE v4.0 term is a MedDRA LLT (Lowest Level Term).

#### **Definitions**

A brief definition is provided to clarify the meaning of each AE term.

#### Grades

Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:

- Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
- Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL\*.
- Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL\*\*.
- Grade 4 Life-threatening consequences; urgent intervention indicated.
- Grade 5 Death related to AE.

A Semi-colon indicates 'or' within the description of the grade.

A single dash (-) indicates a grade is not available.

Not all Grades are appropriate for all AEs. Therefore, some AEs are listed with fewer than five options for Grade selection.

#### Grade 5

Grade 5 (Death) is not appropriate for some AEs and therefore is not an option.

#### Activities of Daily Living (ADL)

\*Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

\*\*Self care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

<sup>†</sup> CTCAE v4.0 incorporates certain elements of the MedDRA terminology. For further details on MedDRA refer to the MedDRA MSSO Web site (http://www.meddramsso.com).

#### CONTENTS

| SOC | Page |
|---------------------------------------------------------------------|------|
| Blood and lymphatic system disorders | 3 |
| Cardiac disorders | 4 |
| Congenital, familial and genetic disorders | 7 |
| Ear and labyrinth disorders | 8 |
| Endocrine disorders | 9 |
| Eye disorders | 10 |
| Gastrointestinal disorders | 12 |
| General disorders and administration site conditions | 22 |
| Hepatobiliary disorders | 24 |
| Immune system disorders | 26 |
| Infections and infestations | 27 |
| Injury, poisoning and procedural complications | 34 |
| Investigations | 41 |
| Metabolism and nutrition disorders | 44 |
| Musculoskeletal and connective tissue disorders | 46 |
| Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 50 |
| Nervous system disorders | 51 |
| Pregnancy, puerperium and perinatal conditions | 56 |
| Psychiatric disorders | 57 |
| Renal and urinary disorders | 59 |
| Reproductive system and breast disorders | 61 |
| Respiratory, thoracic and mediastinal disorders | 65 |
| Skin and subcutaneous tissue disorders | 71 |
| Social circumstances | 75 |
| Surgical and medical procedures | 76 |
| Vascular disorders | 77 |

| | В | lood and lymphatic syste | em disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Anemia | Hemoglobin (Hgb) <lln -="" 10.0<br="">g/dL; <lln -="" -<br="" 6.2="" <lln="" l;="" mmol="">100 g/L</lln></lln> | Hgb <10.0 - 8.0 g/dL; <6.2 - 4.9 mmol/L; <100 - 80g/L | Hgb <8.0 g/dL; <4.9 mmol/L; <80 g/L; transfusion indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by an reduction in the amount on the part of the part, soft systems. | <del>-</del> | = : | ay include pallor of the skin and m | ucous |
| Bone marrow hypocellular | Mildly hypocellular or <=25% reduction from normal cellularity for age | Moderately hypocellular or >25 -<br><50% reduction from normal<br>cellularity for age | Severely hypocellular or >50 -<br><=75% reduction cellularity from<br>normal for age | Aplastic persistent for longer than 2 weeks | Death |
| Definition: A disorder characteriz | ed by the inability of the bone mar | row to produce hematopoietic eler | ments. | | 1 |
| Disseminated intravascular coagulation | - | Laboratory findings with no bleeding | Laboratory findings and bleeding | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by systemic pathological activa<br>s depleted of platelets and coagula | <del>-</del> | which results in clot formation thro | oughout the body. There is an incr | ease in the |
| Febrile neutropenia | - | - | ANC <1000/mm3 with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >=38 degrees C (100.4 degrees F) for more than one hour. | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz degrees F) for more than one ho | ed by an ANC <1000/mm3 and a sur. | single temperature of >38.3 degre | es C (101 degrees F) or a sustain | ed temperature of >=38 degrees C | C (100.4 |
| Hemolysis | Laboratory evidence of<br>hemolysis only (e.g., direct<br>antiglobulin test; DAT; Coombs';<br>schistocytes; decreased<br>haptoglobin) | Evidence of hemolysis and >=2 gm decrease in hemoglobin. | Transfusion or medical intervention indicated (e.g., steroids) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate widespread erythrocyte ce | Il membrane destruction. | T | 1 |
| Hemolytic uremic syndrome | Evidence of RBC destruction (schistocytosis) without clinical consequences | - | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| Definition: A disorder characteriz | ed by a form of thrombotic microal | ngiopathy with renal failure, hemol | ytic anemia, and severe thromboo | cytopenia. | |
| Leukocytosis | - | - | >100,000/mm3 | Clinical manifestations of leucostasis; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate an increased number of wh | nite blood cells in the blood. | T | I |
| Lymph node pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Spleen disorder | Incidental findings (e.g., Howell-Jolly bodies); mild degree of thrombocytosis and leukocytosis | Prophylactic antibiotics indicated | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder of the splee | en. | I | I | T | 1 |
| Thrombotic thrombocytopenic purpura | Evidence of RBC destruction (schistocytosis) without clinical consequences | - | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| | ed by the presence of microangion<br>all disturbances. It is an acute or s | <u>-</u> | cytopenic purpura, fever, renal abr | normalities and neurological abnor | malities such |
| Blood and lymphatic system disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Acute coronary syndrome | - | Symptomatic, progressive angina; cardiac enzymes normal; hemodynamically stable | Symptomatic, unstable angina and/or acute myocardial infarction, cardiac enzymes abnormal, hemodynamically stable | Symptomatic, unstable angina and/or acute myocardial infarction, cardiac enzymes abnormal, hemodynamically unstable | Death |
| | ed by signs and symptoms related unstable angina to myocardial infa | | lium secondary to coronary artery | disease. The clinical presentation | covers a |
| Aortic valve disease | Asymptomatic valvular | Asymptomatic; moderate | Symptomatic; severe | Life-threatening consequences; | Death |
| | thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | regurgitation or stenosis by imaging | regurgitation or stenosis by<br>imaging; symptoms controlled<br>with medical intervention | urgent intervention indicated (e.g., valve replacement, valvuloplasty) | Joan |
| Definition: A disorder characteriz | ed by a defect in aortic valve funct | ion or structure. | | | |
| Asystole | Periods of asystole; non-urgent medical management indicated | - a plactrical pativity. Turnically, this | is accommonical by according of the | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | ed by a dysrhythmia without cardia | | T | 1 | ъ " |
| Atrial fibrillation | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz originates above the ventricles. | ed by a dysrhythmia without disce | rnible P waves and an irregular ve | entricular response due to multiple | reentry circuits. The rhythm distur | bance |
| Atrial flutter | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz atria. | ed by a dysrhythmia with organize | d rhythmic atrial contractions with | a rate of 200-300 beats per minut | e. The rhythm disturbance origina | tes in the |
| Atrioventricular block complete | - | Non-urgent intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with complete | re failure of atrial electrical impulse | conduction through the AV node t | to the ventricles. | ' |
| Atrioventricular block first degree | Asymptomatic, intervention not indicated | Non-urgent intervention indicated | - | - | - |
| | ed by a dysrhythmia with a delay i<br>interval greater than 200 milliseco | · · | tion of an electrical impulse throuç | gh the atrioventricular (AV) node be | eyond 0.2 |
| Cardiac arrest | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by cessation of the pumping fu | nction of the heart. | I | T | T |
| Chest pain - cardiac | Mild pain | Moderate pain; limiting instrumental ADL | Pain at rest; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by substernal discomfort due to | insufficient myocardial oxygenati | on. | _ | |
| Conduction disorder | Mild symptoms; intervention not indicated | Moderate symptoms | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by pathological irregularities in | the cardiac conduction system. | | | |
| Constrictive pericarditis | - | - | Symptomatic heart failure or other cardiac symptoms, responsive to intervention | Refractory heart failure or other poorly controlled cardiac symptoms | Death |
| Definition: A disorder characteriz | ed by a thickened and fibrotic peri | cardial sac; these fibrotic changes | impede normal myocardial function | on by restricting myocardial muscle | e action. |
| Heart failure | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe with symptoms at rest or with minimal activity or exertion; intervention indicated | Life-threatening consequences; urgent intervention indicated (e.g., continuous IV therapy or mechanical hemodynamic support) | Death |
| Definition: A disorder characteriz in the filling pressure. | ed by the inability of the heart to p | ump blood at an adequate volume | to meet tissue metabolic requirer | nents, or, the ability to do so only a | at an elevatior |

| | | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Left ventricular systolic<br>dysfunction | - | - | Symptomatic due to drop in ejection fraction responsive to intervention | Refractory or poorly controlled<br>heart failure due to drop in<br>ejection fraction; intervention<br>such as ventricular assist<br>device, intravenous vasopressor<br>support, or heart transplant<br>indicated | Death |
| | ed by failure of the left ventricle to<br>nea, orthopnea, and other signs ar | | an increase in distending pressure stion and edema. | e and in end-diastolic volume. Clin | ical |
| Mitral valve disease | Asymptomatic valvular<br>thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences; urgent intervention indicated (e.g., valve replacement, valvuloplasty) | Death |
| Definition: A disorder characteriz | ed by a defect in mitral valve funct | tion or structure. | 1 | T | ı |
| Mobitz (type) II atrioventricular<br>block | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with relatively<br>atrioventricular (AV) node to the ve | • | block of an atrial impulse. This is t | he result of intermittent failure of a | trial electrical |
| Mobitz type I | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with a progre<br>on through the atrioventricular (AV | | ior to the blocking of an atrial impu | lse. This is the result of intermitter | nt failure of |
| Myocardial infarction | - | Asymptomatic and cardiac<br>enzymes minimally abnormal<br>and no evidence of ischemic<br>ECG changes | Severe symptoms; cardiac<br>enzymes abnormal;<br>hemodynamically stable; ECG<br>changes consistent with<br>infarction | Life-threatening consequences; hemodynamically unstable | Death |
| Definition: A disorder characteriz | ed by gross necrosis of the myoca | rdium; this is due to an interruptio | n of blood supply to the area. | ' | |
| Myocarditis | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe with symptoms at rest or with minimal activity or exertion; intervention indicated | | Death |
| Definition: A disorder characteriz | ed by inflammation of the muscle | tissue of the heart. | | 1 | Т |
| Palpitations | Mild symptoms; intervention not indicated | Intervention indicated | - | - | - |
| Definition: A disorder characteriz | ed by an unpleasant sensation of | irregular and/or forceful beating of | f the heart. | T | I |
| Paroxysmal atrial tachycardia | Asymptomatic, intervention not indicated | Symptomatic; medical management indicated | IV medication indicated | Life-threatening consequences;<br>incompletely controlled<br>medically; cardioversion<br>indicated | Death |
| Definition: A disorder characteriz originates in the atria. | ed by a dysrhythmia with abrupt o | nset and sudden termination of at | rial contractions with a rate of 150- | -250 beats per minute. The rhythm | disturbance |
| Pericardial effusion | - | Asymptomatic effusion size small to moderate | Effusion with physiologic consequences | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by fluid collection within the per | ricardial sac, usually due to inflam | mation. | T | |
| Pericardial tamponade | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an increase in intrapericardi | | | Ι | |
| Pericarditis | Asymptomatic, ECG or physical findings (e.g., rub) consistent with pericarditis | Symptomatic pericarditis (e.g., chest pain) | Pericarditis with physiologic consequences (e.g., pericardial constriction) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by irritation to the layers of the | pericardium (the protective sac ar | round the heart). | | |

| Cardiac disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pulmonary valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteriz | zed by a defect in pulmonary valve | function or structure. | T | T | 1 |
| Restrictive cardiomyopathy | - | - | Symptomatic heart failure or other cardiac symptoms, responsive to intervention | Refractory heart failure or other poorly controlled cardiac symptoms | Death |
| | zed by an inability of the ventricles | | 1 | | |
| Right ventricular dysfunction | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe symptoms, associated with hypoxemia, right heart failure; oxygen indicated | Life-threatening consequences; urgent intervention indicated (e.g., ventricular assist device); heart transplant indicated | Death |
| | zed by impairment of right ventricul | 1 | | 1 | |
| Sick sinus syndrome | Asymptomatic, intervention not indicated | Non-urgent intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by a dysrhythmia with alternatii | ng periods of bradycardia and atria | al tachycardia accompanied by syr | ncope, fatigue and dizziness. | 1 |
| Sinus bradycardia | Asymptomatic, intervention not indicated | Symptomatic, medical intervention indicated | Severe, medically significant, medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by a dysrhythmia with a heart r | ate less than 60 beats per minute | that originates in the sinus node. | T | 1 |
| Sinus tachycardia | Asymptomatic, intervention not indicated | Symptomatic; non-urgent medical intervention indicated | Urgent medical intervention indicated | - | - |
| Definition: A disorder characteriz | zed by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates in the sinus no | de. | |
| Supraventricular tachycardia | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates above the ven | tricles. | |
| Tricuspid valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| | zed by a defect in tricuspid valve fu | | | | |
| Ventricular arrhythmia | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by a dysrhythmia that originate | s in the ventricles. | | | |
| Ventricular fibrillation | - | - | - | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz ventricles. | zed by a dysrhythmia without disce | rnible QRS complexes due to rapi | d repetitive excitation of myocardi | al fibers without coordinated contra | action of the |
| Ventricular tachycardia | - | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates distal to the bu | indle of His. | |
| Wolff-Parkinson-White<br>syndrome | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically or controlled with procedure | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the presence of an accesso | ry conductive pathway between th | e atria and the ventricles that caus | ses premature ventricular activatio | n. |
| Cardiac disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Congenital, familial and genetic disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Congenital, familial and genetic disorders - Other, specify | • | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Ear and labyrinth dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Ear pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | zed by a sensation of marked disco | mfort in the ear. | | | |
| External ear inflammation | External otitis with erythema or dry desquamation | External otitis with moist<br>desquamation, edema,<br>enhanced cerumen or<br>discharge; tympanic membrane<br>perforation; tympanostomy | External otitis with mastoiditis;<br>stenosis or osteomyelitis;<br>necrosis of soft tissue or bone | Urgent operative intervention indicated | Death |
| Definition: A disorder characterize | zed by inflammation, swelling and r | ·<br>edness to the outer ear and ear ca | anal. | ' | ' |
| External ear pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care | - | - |
| Definition: A disorder characteriz | zed by a sensation of marked disco | mfort in the external ear region. | | | |
| Hearing impaired Definition: A disorder characterize | Adults enrolled on a Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of 15 - 25 dB averaged at 2 contiguous test frequencies in at least one ear. Adults not enrolled in Monitoring Program: subjective change in hearing in the absence of documented hearing loss. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift >20 dB at 8 kHz in at least one ear. | contiguous test frequencies in at least one ear. Adults not enrolled in Monitoring Program: hearing loss but hearing aid or intervention not indicated; limiting instrumental ADL. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift >20 dB at 4 kHz and above in at least one ear. | Adults enrolled in Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of >25 dB averaged at 3 contiguous test frequencies in at least one ear; therapeutic intervention indicated. Adults not enrolled in Monitoring Program: hearing loss with hearing aid or intervention indicated; limiting self care ADL. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): hearing loss sufficient to indicate therapeutic intervention, including hearing aids; threshold shift >20 dB at 3 kHz and above in at least one ear; additional speech-language related services indicated. | Pediatric: Audiologic indication<br>for cochlear implant and<br>additional speech-language<br>related services indicated. | - |
| Middle ear inflammation | Serous otitis | Serous otitis, medical intervention indicated | Mastoiditis; necrosis of canal | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ा<br>zed by inflammation (physiologic re | 1 | 1 | ı <del>-</del> | T. |
| Tinnitus | Mild symptoms; intervention not indicated | · · · · · · | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by noise in the ears, such as rir | nging, buzzing, roaring or clicking. | Г | <u> </u> | |
| Vertigo | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz vertigo). | zed by a sensation as if the externa | al world were revolving around the | patient (objective vertigo) or as if | he himself were revolving in space | e (subjective |
| Vestibular disorder | - | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by dizziness, imbalance, nause | ea, and vision problems. | Т | <u> </u> | ı |
| Ear and labyrinth disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Endocrine disord | lers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Adrenal insufficiency | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death to a disorder |
| | s when the adrenal cortex does not<br>con's disease or primary adrenal ins | | cortisol and in some cases, the no | rmone aldosterone. It may be due | to a disorder |
| Cushingoid | Mild symptoms; intervention not indicated | | Severe symptoms, medical intervention or hospitalization indicated | - | - |
| Definition: A disorder characteriz osteoporosis, usually due to exo | zed by signs and symptoms that regenous corticosteroids. | semble Cushing's disease or sync | frome: buffalo hump obesity, striat | ions, adiposity, hypertension, diab | etes, and |
| Delayed puberty | - | No breast development by age<br>13 yrs for females; testes<br>volume of <3 cc or no Tanner<br>Stage 2 development by age<br>14.5 yrs for males | No breast development by age<br>14 yrs for females; no increase<br>in testes volume or no Tanner<br>Stage 2 by age 16 yrs for<br>males; hormone replacement<br>indicated | - | - |
| Definition: A disorder characteriz | zed by unusually late sexual maturi | ty. | | | |
| Growth accelerated | - | >= +2 SD (standard deviation)<br>above mid parental height or<br>target height | - | - | - |
| Definition: A disorder characterize | zed by greater growth than expecte | ed for age. | 1 | I | 1 |
| Hyperparathyroidism | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder characterize the blood). | zed by an increase in production of | parathyroid hormone by the para | thyroid glands. This results in hype | ercalcemia (abnormally high levels | of calcium in |
| Hyperthyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thyroid suppression therapy indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by excessive levels of thyroid h | ormone in the body. Common car | uses include an overactive thyroid | gland or thyroid hormone overdos | e. |
| Hypoparathyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; medical intervention or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by a decrease in production of | parathyroid hormone by the parat | hyroid glands. | | |
| Hypothyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thyroid replacement indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by a decrease in production of | | and.<br>T | | |
| Precocious puberty | Physical signs of puberty with<br>no biochemical markers for<br>females <8 years and males <9<br>years | Physical signs and biochemical markers of puberty for females <8 years and males <9 years | - | - | - |
| Definition: A disorder characteriz 9 for boys. | zed by unusually early developmen | t of secondary sexual features; th | e onset of sexual maturation begir | ns usually before age 8 for girls an | d before age |
| Virilization | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder characteriz | zed by inappropriate masculinization | n occurring in a female or prepub | ertal male. | | |
| Endocrine disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Eye disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Blurred vision | Intervention not indicated | Symptomatic; limiting instrumental ADL | Limiting self care ADL | - | - |
| | erized by visual perception of u | | C | Dii: | |
| Cataract Definition: A disorder characte | Asymptomatic; clinical or diagnostic observations only; intervention not indicated erized by partial or complete op | Symptomatic; moderate decrease in visual acuity (20/40 or better) | Symptomatic with marked decrease in visual acuity (worse than 20/40 but better than 20/200); operative intervention indicated (e.g., cataract surgery) one or both eyes. This results in | Blindness (20/200 or worse) in the affected eye a decrease in visual acuity an | d eventual blindness if |
| untreated. | 1 | 1 | <b>.</b> | | 1 |
| Conjunctivitis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; topical intervention indicated (e.g., antibiotics); limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder characte | erized by inflammation, swelling | g and redness to the conjunctiv | a of the eye. | | |
| Corneal ulcer | - | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Limiting self care ADL;<br>declining vision (worse than<br>20/40 but better than 20/200) | Perforation or blindness<br>(20/200 or worse) in the<br>affected eye | - |
| Definition: A disorder characte | erized by an area of epithelial ti | ssue loss on the surface of the | cornea. It is associated with in | flammatory cells in the cornea | and anterior chamber. |
| Dry eye | Asymptomatic; clinical or diagnostic observations only; mild symptoms relieved by lubricants | Symptomatic; multiple<br>agents indicated; limiting<br>instrumental ADL | Decrease in visual acuity<br>(<20/40); limiting self care<br>ADL | - | - |
| Definition: A disorder characte | erized by dryness of the cornea | and conjunctiva. | T | | ı |
| Extraocular muscle paresis | Asymptomatic; clinical or diagnostic observations only | Symptomatic; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characte | erized by incomplete paralysis o | of an extraocular muscle. | T | T | T |
| Eye pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characte | erized by a sensation of marked | d discomfort in the eye. | Γ | | |
| Eyelid function disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; nonoperative intervention indicated; limiting instrumental ADL | Limiting self care ADL;<br>operative intervention<br>indicated | - | - |
| Definition: A disorder characte | erized by impaired eyelid function | on. | Τ | <u> </u> | Г |
| Flashing lights | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder characte | erized by a sudden or brief burs | st of light. | Γ | | |
| Floaters | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder characte | | | ots are shadows of opaque cell | | or or lens. |
| Glaucoma | Elevated intraocular<br>pressure (EIOP) with single<br>topical agent for intervention;<br>no visual field deficit | EIOP causing early visual<br>field deficits; multiple topical<br>or oral agents indicated;<br>limiting instrumental ADL | EIOP causing marked visual<br>field deficits (e.g., involving<br>both superior and inferior<br>visual fields); operative<br>intervention indicated;<br>limiting self care ADL | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | erized by an increase in pressu | re in the eyeball due to obstruc | ction of the aqueous humor out | low. | |
| Keratitis | - | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Decline in vision (worse than<br>20/40 but better than<br>20/200); limiting self care<br>ADL | Perforation or blindness<br>(20/200 or worse) in the<br>affected eye | - |
| Definition: A disorder characte | erized by inflammation to the co | ornea of the eye. | Γ | | Г |
| Night blindness | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | erized by an inability to see clea | arly in dim light. | | | |

| | | Eye dis | sorders | | |
|---|---|---|---|---|---|
| | | · | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Optic nerve disorder | Asymptomatic; clinical or diagnostic observations only erized by involvement of the op | eye (20/40 or better) | eye (worse than 20/40 but<br>better than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| | 1 | · · | Marked visual field defect | Plindness (20/200 or worse) | |
| Papilledema | Asymptomatic; no visual field defects | vision; visual field defect<br>present sparing the central<br>20 degrees | (worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | erized by swelling around the o | ptic disc. | | | |
| Photophobia | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder characte | erized by fear and avoidance of | light. | 1 | 1 | |
| Retinal detachment | Asymptomatic | Exudative and visual acuity<br>20/40 or better | Rhegmatogenous or<br>exudative detachment;<br>operative intervention<br>indicated; decline in vision<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | erized by the separation of the i | nner retina layers from the unc | lerlying pigment epithelium. | | _ |
| Retinal tear | - | Laser therapy or pneumopexy indicated | Vitroretinal surgical repair indicated | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | erized by a small laceration of t | he retina, this occurs when the | vitreous separates from the re | tina. Symptoms include flashes | and floaters. |
| Retinal vascular disorder | - | Topical medication indicated | Intravitreal medication; operative intervention indicated | - | - |
| Definition: A disorder characte | erized by pathological retinal blo | ood vessels that adversely affe | cts vision. | | |
| Retinopathy | Asymptomatic; clinical or diagnostic observations only | Symptomatic with moderate decrease in visual acuity (20/40 or better); limiting instrumental ADL | Symptomatic with marked decrease in visual acuity (worse than 20/40); disabling; limiting self care ADL | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder involving | g the retina. | ' | ' | ' | ' |
| Scleral disorder | Asymptomatic; clinical or diagnostic observations only | Symptomatic, limiting instrumental ADL; moderate decrease in visual acuity (20/40 or better) | Symptomatic, limiting self care ADL; marked decrease in visual acuity (worse than 20/40) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | erized by involvement of the sol | era of the eye. | | | |
| Uveitis | Asymptomatic; clinical or diagnostic observations only | Anterior uveitis; medical intervention indicated | Posterior or pan-uveitis | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | erized by inflammation to the uv | yea of the eye. | | | |
| Vitreous hemorrhage | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only | Symptomatic; limiting instrumental ADL | Limiting self care ADL;<br>vitrectomy indicated | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | erized by blood extravasation in | to the vitreous humor. | | | I |
| Watering eyes | Intervention not indicated | Intervention indicated | Operative intervention indicated | - | - |
| Definition: A disorder of exces | ssive tearing in the eyes; it can | be caused by overproduction o | of tears or impaired drainage of | the tear duct. | |
| Eye disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental<br>ADL | Severe or medically<br>significant but not<br>immediately sight-<br>threatening; hospitalization<br>or prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care<br>ADL | Sight-threatening<br>consequences; urgent<br>intervention indicated;<br>blindness (20/200 or worse)<br>in the affected eye | - |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal distension | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe discomfort; limiting self care ADL | - | - |
| | rized by swelling of the abdomen. | A | 0 ' | | |
| Abdominal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | rized by a sensation of marked disco | omfort in the abdominal region. | T | | |
| Anal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | between the opening in the anal | canal to the perianal skin. | | |
| Anal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | 1 | | C | | D 41- |
| Anal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by inflammation of the mucous | membrane of the anus. | T | | 1 |
| Anal necrosis | - | - | TPN or hospitalization indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by a necrotic process occurring | i i | | | |
| Anal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | rized by a sensation of marked disco | omfort in the anal region. | T | T | |
| Anal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; non-<br>emergent operative intervention<br>indicated; TPN or hospitalization<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by a narrowing of the lumen of | the anal canal. | _ | | |
| Anal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the anal ca | nal. | |
| Ascites | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by accumulation of serous or h | emorrhagic fluid in the peritoneal | cavity. | | |
| Bloating | No change in bowel function or oral intake | Symptomatic, decreased oral intake; change in bowel function | - | - | - |
| Definition: A disorder character | rized by subject-reported feeling of u | incomfortable fullness of the abdo | men. | | |
| Cecal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by bleeding from the cecum. | | | | |
| Cheilitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; intervention indicated | - | - |
| D C ''' A I' I I I | rized by inflammation of the lip. | | | | |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | Г | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Colitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood in stool | Severe abdominal pain; change in bowel habits; medical intervention indicated; peritoneal signs | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inflammation of the colon. | | _ | | |
| Colonic fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function | Severely altered GI function;<br>bowel rest, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | between the large intestine and a | another organ or anatomic site. | | |
| Colonic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the colon. | | T | | |
| Colonic obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Hospitalization indicated;<br>elective operative intervention<br>indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | erized by blockage of the normal flow | | | Life threatening con | Doot!- |
| Colonic perforation | | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by a rupture in the colonic wall. | 0 1 11 101 | 0 1 11 1016 11 | lee ii e | Б " |
| Colonic stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by a narrowing of the lumen of | the colon. | | • | , |
| Colonic ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a circumscribed, inflammato | ry and necrotic erosive lesion on t | the mucosal surface of the colon. | | |
| Constipation | Occasional or intermittent<br>symptoms; occasional use of<br>stool softeners, laxatives,<br>dietary modification, or enema | Persistent symptoms with regular use of laxatives or enemas; limiting instrumental ADL | Obstipation with manual evacuation indicated; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by irregular and infrequent or d | ifficult evacuation of the bowels. | | | |
| Dental caries | One or more dental caries, not involving the root | Dental caries involving the root | Dental caries resulting in pulpitis<br>or periapical abscess or<br>resulting in tooth loss | - | - |
| | erized by the decay of a tooth, in whic | | 1 | | |
| Diarrhea | Increase of <4 stools per day<br>over baseline; mild increase in<br>ostomy output compared to<br>baseline | Increase of 4 - 6 stools per day<br>over baseline; moderate<br>increase in ostomy output<br>compared to baseline | Increase of >=7 stools per day<br>over baseline; incontinence;<br>hospitalization indicated; severe<br>increase in ostomy output<br>compared to baseline; limiting<br>self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by frequent and watery bowel n | novements. | I | Г | |
| Dry mouth | Symptomatic (e.g., dry or thick saliva) without significant dietary alteration; unstimulated saliva flow >0.2 ml/min | Moderate symptoms; oral intake alterations (e.g., copious water, other lubricants, diet limited to purees and/or soft, moist foods); unstimulated saliva 0.1 to 0.2 ml/min | Inability to adequately aliment orally; tube feeding or TPN indicated; unstimulated saliva <0.1 ml/min | - | - |
| | 1 | oral cavity. | 1 | I | 1 |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Duodenal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the duodenum and anot | ther organ or anatomic site. | _ | |
| Duodenal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the duodenun | 1.<br>I | Т | T | |
| Duodenal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Hospitalization or elective operative intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by blockage of the normal flow | of stomach contents through the c | duodenum. | _ | |
| Duodenal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the duodenal wa | all. | T | | |
| Duodenal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the duodenum. | | | |
| Duodenal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a circumscribed, inflammato | ry and necrotic erosive lesion on t | he mucosal surface of the duoder | nal wall. | |
| Dyspepsia | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; surgical intervention indicated | - | - |
| Definition: A disorder characteriz heartburn, nausea and vomiting. | ed by an uncomfortable, often pair | nful feeling in the stomach, resultir | ng from impaired digestion. Sympt | oms include burning stomach, blo | ating, |
| Dysphagia | Symptomatic, able to eat regular diet | Symptomatic and altered eating/swallowing | Severely altered<br>eating/swallowing; tube feeding<br>or TPN or hospitalization<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by difficulty in swallowing. | | | | |
| Enterocolitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood in stool | Severe or persistent abdominal pain; fever; ileus; peritoneal signs | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the small an | d large intestines. | T | | |
| Enterovesical fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; noninvasive intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the urinary bladder and | the intestine. | 1 | 1 |
| Esophageal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the esophagus and ano | ther organ or anatomic site. | 1 | 1 |
| Esophageal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the esophagu | S. | | | |

| | | Gastrointestinal dis | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Esophageal necrosis | - | - | Inability to aliment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | in the esophageal wall. | _ | | |
| Esophageal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by blockage of the normal flow | of the contents in the esophagus | | | |
| Esophageal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by a sensation of marked disco | omfort in the esophageal region. | | | |
| Esophageal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by a rupture in the wall of the e | sophagus. | | | |
| Esophageal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by a narrowing of the lumen of | the esophagus. | | | |
| Esophageal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the esopha | geal wall. | |
| Esophageal varices<br>hemorrhage | - | Self-limited; intervention not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by bleeding from esophageal v | rarices. | T | Т | |
| Esophagitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered eating/swallowing; oral supplements indicated | Severely altered<br>eating/swallowing; tube feeding,<br>TPN or hospitalization indicated | | Death |
| | zed by inflammation of the esopha | 1 | | | |
| Fecal incontinence | Occasional use of pads required | Daily use of pads required | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteri | zed by inability to control the escap | e of stool from the rectum. | | | |
| Flatulence | Mild symptoms; intervention not indicated | Moderate; persistent;<br>psychosocial sequelae | - | - | - |
| Definition: A disorder characteri | zed by a state of excessive gas in t | the alimentary canal. | T | T | |
| Gastric fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>bowel rest; tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | between the stomach and anoth | ner organ or anatomic site. | | |
| Gastric hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by bleeding from the gastric wa | all. | | | |
| Gastric necrosis | - | - | Inability to aliment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Gastric perforation Definition: A disorder characterize | -<br>ed by a rupture in the stomach wa | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Gastric stenosis | Asymptomatic; clinical or | Symptomatic; altered GI | Soverely altered Cl function: | Life threatening consequences: | Dooth |
| Gastric stenosis | diagnostic observations only; intervention not indicated | function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the stomach. | | | |
| Gastric ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; medical intervention<br>indicated; limiting instrumental<br>ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | 1 | ſ | the mucosal surface of the stomac | | |
| Gastritis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; medical intervention indicated | Severely altered eating or<br>gastric function; TPN or<br>hospitalization indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | ed by inflammation of the stomach | l. | T | | |
| Gastroesophageal reflux disease | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; surgical intervention indicated | - | - |
| | ed by reflux of the gastric and/or d<br>result in injury to the esophageal m | | sophagus. It is chronic in nature ar<br>urn and acid indigestion. | nd usually caused by incompetend | e of the lower |
| Gastrointestinal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between any part of the gastroin | testinal system and another organ | or anatomic site. | |
| Gastrointestinal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characterize | ed by a sensation of marked disco | mfort in the gastrointestinal region | 1. | | |
| Gastroparesis | Mild nausea, early satiety and<br>bloating, able to maintain caloric<br>intake on regular diet | Moderate symptoms; able to maintain nutrition with dietary and lifestyle modifications; may need pharmacologic intervention | Weight loss; refractory to medical intervention; unable to maintain nutrition orally | - | - |
| Definition: A disorder characteriz | ed by an incomplete paralysis of th | ne muscles of the stomach wall re | sulting in delayed emptying of the | gastric contents into the small inte | estine. |
| Gingival pain | Mild pain | Moderate pain interfering with oral intake | Severe pain; inability to aliment orally | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | mfort in the gingival region. | | | |
| Hemorrhoidal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the hemorrho | ids. | T | T | |
| Hemorrhoids | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; banding or medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | - | - |
| Definition: A disorder characteriz | ed by the presence of dilated vein: | s in the rectum and surrounding a | rea. | ı | 1 |
| lleal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the ileum and another o | organ or anatomic site. | Г | 1 |
| lleal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the ileal wall. | | | | |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | T |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| lleal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | ed by blockage of the normal flow | | um.<br>T | | |
| lleal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the ileal wall. | | | | |
| Ileal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the ileum. | | | |
| lleal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the ileum. | 1 | 1 |
| lleus | - | Symptomatic; altered GI function; bowel rest indicated | Severely altered GI function;<br>TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by failure of the ileum to transp | | | | |
| Intra-abdominal hemorrhage | - | Medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding in the abdominal c | avity. | | | |
| Jejunal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | ,<br>n between the jejunum and anothe | r organ or anatomic site. | • | , |
| Jejunal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the jejunal wa | ıll. | • | • | , |
| Jejunal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by blockage of the normal flow | of the intestinal contents in the jej | unum. | | |
| Jejunal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the jejunal wall. | | | | |
| Jejunal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the jejunum. | | | |
| Jejunal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the jejunun | 1. | 1 |
| Lip pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort of the lip. | | | |

| | | Gastrointestinal dis | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| ower gastrointestinal.<br>emorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by bleeding from the lower gas | trointestinal tract (small intestine, | large intestine, and anus). | 1 | |
| Malabsorption | - | Altered diet; oral intervention indicated | Inability to aliment adequately; TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by inadequate absorption of nu | | | 1 | |
| Mucositis oral | Asymptomatic or mild symptoms; intervention not indicated | Moderate pain; not interfering with oral intake; modified diet indicated | Severe pain; interfering with oral intake | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by inflammation of the oral muc | cosal. | 1 | T | |
| Nausea | Loss of appetite without alteration in eating habits | Oral intake decreased without significant weight loss, dehydration or malnutrition | Inadequate oral caloric or fluid intake; tube feeding, TPN, or hospitalization indicated | - | - |
| | rized by a queasy sensation and/or t | 1 | T | | |
| Obstruction gastric | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | rized by blockage of the normal flow | | T | | |
| Oral cavity fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | n between the oral cavity and ano | ther organ or anatomic site. | 1 | |
| Oral dysesthesia | Mild discomfort; not interfering with oral intake | Moderate pain; interfering with oral intake | Disabling pain; tube feeding or TPN indicated | - | - |
| | rized by a burning or tingling sensati | | | | L |
| Oral hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by bleeding from the mouth. | T | 1 | T | |
| Oral pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| | rized by a sensation of marked disco | 1 | | | |
| Pancreatic duct stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by a narrowing of the lumen of | the pancreatic duct. | | | |
| Pancreatic fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | n between the pancreas and anoth | ner organ or anatomic site. | T | |
| Pancreatic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by bleeding from the pancreas. | | 1 | _ | |
| Pancreatic necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | rized by a necrotic process occurring | 1 | | <u> </u> | |
| Pancreatitis | - | Enzyme elevation or radiologic findings only | Severe pain; vomiting; medical intervention indicated (e.g., analgesia, nutritional support) | Life-threatening consequences; urgent intervention indicated | Death |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | ed by inflammation of the pancrea | s. | 1 | T | |
| Periodontal disease | Gingival recession or gingivitis;<br>limited bleeding on probing; mild<br>local bone loss | Moderate gingival recession or<br>gingivitis; multiple sites of<br>bleeding on probing; moderate<br>bone loss | Spontaneous bleeding; severe bone loss with or without tooth loss; osteonecrosis of maxilla or mandible | - | - |
| Definition: A disorder in the gingi | ival tissue around the teeth. | | | T | |
| Peritoneal necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | red by a necrotic process occurring | in the peritoneum. | 1 | T | |
| Proctitis | Rectal discomfort, intervention not indicated | Symptoms (e.g., rectal<br>discomfort, passing blood or<br>mucus); medical intervention<br>indicated; limiting instrumental<br>ADL | Severe symptoms; fecal<br>urgency or stool incontinence;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the rectum. | | | | |
| Rectal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the rectum and another | organ or anatomic site. | | |
| Rectal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the rectal wall | and discharged from the anus. | 1 | T | |
| Rectal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent operative intervention indicated | Death |
| | ted by inflammation of the mucous | membrane of the rectum. | | | |
| Rectal necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | red by a necrotic process occurring | in the rectal wall. | | | |
| Rectal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | red by blockage of the normal flow | of the intestinal contents in the re | ctum. | T | |
| Rectal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| | red by a sensation of marked disco | _ | | <u> </u> | |
| Rectal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ted by a rupture in the rectal wall. | | 1 | | |
| Rectal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the rectum. | | 1 | |
| Rectal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function (e.g. altered dietary<br>habits, vomiting, diarrhea) | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a circumscribed, inflammato | ry and necrotic erosive lesion on | the mucosal surface of the rectum | · | • |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Retroperitoneal hemorrhage | -<br>ed by bleeding from the retroperite | Self-limited; intervention indicated | Transfusion, medical, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | | | | Lie ii i | Б " |
| Salivary duct inflammation | Slightly thickened saliva; slightly altered taste (e.g., metallic) | Thick, ropy, sticky saliva;<br>markedly altered taste;<br>alteration in diet indicated;<br>secretion-induced symptoms;<br>limiting instrumental ADL | Acute salivary gland necrosis;<br>severe secretion-induced<br>symptoms (e.g., thick saliva/oral<br>secretions or gagging); tube<br>feeding or TPN indicated;<br>limiting self care ADL; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the salivary | duct. | | | |
| Salivary gland fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; tube feeding indicated | Severely altered GI function;<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between a salivary gland and an | other organ or anatomic site. | | |
| Small intestinal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe pain; interfering with oral intake; tube feeding, TPN or hospitalization indicated; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the mucous | membrane of the small intestine. | | | |
| Small intestinal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by blockage of the normal flow | of the intestinal contents. | | | |
| Small intestinal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the small intesti | ne wall. | | | |
| Small intestinal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the small intestine. | | | |
| Small intestine ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a circumscribed, inflammato | ry and necrotic erosive lesion on t | the mucosal surface of the small in | ntestine. | |
| Stomach pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the stomach. | I | T | 1 |
| ooth development disorder | Asymptomatic; hypoplasia of tooth or enamel | Impairment correctable with oral surgery | Maldevelopment with impairment not surgically correctable; disabling | - | - |
| Definition: A disorder characteriz | ed by a pathological process of the | e teeth occurring during tooth deve | elopment. | T | 1 |
| ooth discoloration | Surface stains | - | - | - | - |
| Definition: A disorder characteriz | ed by a change in tooth hue or tint | i. | | | 1 |
| oothache | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | ı | • | | ' |

| 1 | 2 | Grade | | | | | | | |
|---|---|---|---|---|--|--|--|--|--|
| 1 | 2 | | Grade | | | | | | |
| | = | 3 | 4 | 5 | | | | | |
| - | - | Symptomatic (e.g., abdominal pain, fever, change in bowel habits with ileus); peritoneal signs | Life-threatening consequences; urgent operative intervention indicated | Death | | | | | |
| ed by inflammation of the cecum. | | | | | | | | | |
| Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death | | | | | |
| ed by bleeding from the upper gas | trointestinal tract (oral cavity, pha | rynx, esophagus, and stomach). | | | | | | | |
| 1 - 2 episodes (separated by 5 minutes) in 24 hrs | 3 - 5 episodes (separated by 5 minutes) in 24 hrs | >=6 episodes (separated by 5 minutes) in 24 hrs; tube feeding, TPN or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death | | | | | |
| ed by the reflexive act of ejecting t | he contents of the stomach throug | gh the mouth. | | | | | | | |
| Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death | | | | | |
| | Mild; intervention not indicated ed by bleeding from the upper gas 1 - 2 episodes (separated by 5 minutes) in 24 hrs ed by the reflexive act of ejecting to the symptomatic or mild symptoms; clinical or diagnostic observations only; intervention | Mild; intervention not indicated Moderate symptoms; medical intervention or minor cauterization indicated ed by bleeding from the upper gastrointestinal tract (oral cavity, pharmal 1 - 2 episodes (separated by 5 minutes) in 24 hrs 3 - 5 episodes (separated by 5 minutes) in 24 hrs ed by the reflexive act of ejecting the contents of the stomach through the symptomatic or mild symptoms; clinical or diagnostic observations only; intervention indicated; limiting age- | signs and by inflammation of the cecum. Mild; intervention not indicated intervention or minor cauterization indicated ed by bleeding from the upper gastrointestinal tract (oral cavity, pharynx, esophagus, and stomach). 1 - 2 episodes (separated by 5 minutes) in 24 hrs 3 - 5 episodes (separated by 5 minutes) in 24 hrs 3 - 5 episodes (separated by 5 minutes) in 24 hrs 3 - 6 episodes (separated by 5 minutes) in 24 hrs; tube feeding, TPN or hospitalization indicated ed by the reflexive act of ejecting the contents of the stomach through the mouth. Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated instrumental ADL signs Transfusion, radiologic, endoscopic, or elective operative intervention indicated See episodes (separated by 5 minutes) in 24 hrs; tube feeding, TPN or hospitalization indicated Severe or medically significant but not immediately lifethreatening; hospitalization or prolongation of existing | signs Signs | | | | | |
| | | | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Chills | Mild sensation of cold;<br>shivering; chattering of teeth | Moderate tremor of the entire body; narcotics indicated | Severe or prolonged, not responsive to narcotics | - | - |
| Definition: A disorder charact | erized by a sensation of cold that often | n marks a physiologic response to | sweating after a fever. | _ | |
| Death neonatal | - | - | - | - | Death |
| Definition: A disorder charact | erized by cessation of life occurring du | uring the first 28 days of life. | | | |
| Death NOS | - | - | - | - | Death |
| Definition: A cessation of life | that cannot be attributed to a CTCAE | term associated with Grade 5. | | | |
| Edema face | Localized facial edema | Moderate localized facial edema; limiting instrumental ADL | Severe swelling; limiting self care ADL | - | - |
| Definition: A disorder charact | erized by swelling due to excessive flu | uid accumulation in facial tissues. | _ | | |
| Edema limbs | 5 - 10% inter-limb discrepancy in volume or circumference at point of greatest visible difference; swelling or obscuration of anatomic architecture on close inspection | >10 - 30% inter-limb<br>discrepancy in volume or<br>circumference at point of<br>greatest visible difference;<br>readily apparent obscuration of<br>anatomic architecture;<br>obliteration of skin folds; readily<br>apparent deviation from normal<br>anatomic contour; limiting<br>instrumental ADL | >30% inter-limb discrepancy in<br>volume; gross deviation from<br>normal anatomic contour;<br>limiting self care ADL | - | - |
| Definition: A disorder charact | erized by swelling due to excessive flu | uid accumulation in the upper or lo | wer extremities. | • | , |
| Edema trunk | Swelling or obscuration of anatomic architecture on close inspection | Readily apparent obscuration of anatomic architecture; obliteration of skin folds; readily apparent deviation from normal anatomic contour; limiting instrumental ADL | anatomic contour; limiting self care ADL | - | - |
| | erized by swelling due to excessive flu | | | | |
| acial pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder charact | erized by a sensation of marked disco | mfort in the face. | 1 | 1 | 1 |
| Fatigue | Fatigue relieved by rest | Fatigue not relieved by rest;<br>limiting instrumental ADL | Fatigue not relieved by rest, limiting self care ADL | - | - |
| Definition: A disorder charact | erized by a state of generalized weak | ness with a pronounced inability to | summon sufficient energy to acc | omplish daily activities. | 1 |
| Fever | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) | >40.0 degrees C (>104.0 degrees F) for <=24 hrs | >40.0 degrees C (>104.0 degrees F) for >24 hrs | Death |
| | erized by elevation of the body's temp | | | | |
| lu like symptoms | Mild flu-like symptoms present | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder charact ough. | erized by a group of symptoms similar | to those observed in patients with | n the flu. It includes fever, chills, b | ody aches, malaise, loss of appeti | ite and dry |
| Sait disturbance | Mild change in gait (e.g., wide-<br>based, limping or hobbling) | Moderate change in gait (e.g., wide-based, limping or hobbling); assistive device indicated; limiting instrumental ADL | Disabling; limiting self care ADL | - | - |
| Definition: A disorder charact | erized by walking difficulties. | | | | |
| Hypothermia | - | 35 - >32 degrees C; 95 - >89.6 degrees F | 32 - >28 degrees C; 89.6 -<br>>82.4 degrees F | <=28 degrees C; 82.4 degrees<br>F; life-threatening<br>consequences (e.g., coma,<br>hypotension, pulmonary edema,<br>acidemia, ventricular fibrillation) | Death |

| | Conoral | disorders and administra | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| nfusion related reaction | Mild transient reaction; infusion | Therapy or infusion interruption | Prolonged (e.g., not rapidly | Life-threatening consequences; | Death |
| Thusion related reaction | interruption not indicated; | indicated but responds promptly | responsive to symptomatic | urgent intervention indicated | Death |
| | intervention not indicated | to symptomatic treatment (e.g., | medication and/or brief | argoni microminan maicatea | |
| | | antihistamines, NSAIDS, | interruption of infusion); | | |
| | | narcotics, IV fluids); prophylactic | | | |
| | | medications indicated for <=24 | following initial improvement; | | |
| | | hrs | hospitalization indicated for | | |
| | | | clinical sequelae | | |
| Definition: Δ disorder characteria | ।<br>zed by adverse reaction to the infus | ion of pharmacological or hiologic | 1 | | l |
| | Led by adverse reaction to the linus | | | | D45 |
| nfusion site extravasation | - | Erythema with associated | Ulceration or necrosis; severe | Life-threatening consequences; | Death |
| | | symptoms (e.g., edema, pain, | tissue damage; operative | urgent intervention indicated | |
| | | induration, phlebitis) | intervention indicated | | |
| | zed by leakage of a pharmacologic | <del>-</del> | nfusion site into the surrounding ti | ssue. Signs and symptoms include | e induratio |
| rythema, swelling, burning sens | sation and marked discomfort at the | e infusion site. | | | 1 |
| njection site reaction | Tenderness with or without | Pain; lipodystrophy; edema; | Ulceration or necrosis; severe | Life-threatening consequences; | Death |
| | associated symptoms (e.g., | phlebitis | tissue damage; operative | urgent intervention indicated | |
| | warmth, erythema, itching) | | intervention indicated | | |
| Definition: A disorder characteriz | ed by an intense adverse reaction | (usually immunologic) developing | at the site of an injection. | | |
| rritability | Mild; easily consolable | Moderate; limiting instrumental | Severe abnormal or excessive | - | - |
| | | ADL; increased attention | response; limiting self care ADL; | | |
| | | indicated | inconsolable | | |
| Definition: A disorder characteria | red by an abnormal responsivenes | ı<br>e to etimuli or physiological arous: | l<br>al: may be in response to pain frig | t<br>ht a drug an emotional situation ( | ı<br>or a medic |
| condition. | ed by all abilionnal responsivenes | s to stillfull of physiological arouse | ai, may be in response to pain, mg | ni, a drug, an emotional situation ( | Ji a medic |
| ocalized edema | Localized to dependent areas, | Moderate localized edema and | Severe localized edema and | | |
| ocalized edema | | | | - | - |
| | no disability or functional impairment | intervention indicated; limiting instrumental ADL | intervention indicated; limiting self care ADL | | |
| | | ı | 1 | | 1 |
| Definition: A disorder characteriz | zed by swelling due to excessive flu | uid accumulation at a specific anal | omic site. | | |
| Malaise | Uneasiness or lack of well being | | - | - | - |
| | | being; limiting instrumental ADL | | | |
| Definition: A disorder characteriz | zed by a feeling of general discomf | ort or uneasiness, an out-of-sorts | feeling. | | |
| Multi-organ failure | - | - | Shock with azotemia and acid- | Life-threatening consequences | Death |
| | | | base disturbances; significant | (e.g., vasopressor dependent | |
| | | | coagulation abnormalities | and oliguric or anuric or | |
| | | | | ischemic colitis or lactic | |
| | | | | acidosis) | |
| Definition: A disorder characteriz | zed by progressive deterioration of | the lungs, liver, kidnev and clotting | mechanisms. | | |
| leck edema | Asymptomatic localized neck | Moderate neck edema; slight | Generalized neck edema (e.g., | _ | |
| took edema | edema | obliteration of anatomic | difficulty in turning neck); | | |
| | edema | landmarks; limiting instrumental | limiting self care ADL | | |
| | | ADL | limiting sen care ADL | | |
| | | IADL | I | | l |
| N-fi-iki A didlki- | | | | | |
| | zed by swelling due to an accumula | | | | |
| Definition: A disorder characteriz | red by swelling due to an accumula | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| Non-cardiac chest pain | Mild pain | Moderate pain; limiting instrumental ADL | | - | - |
| Non-cardiac chest pain | T | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care | - | - |
| Non-cardiac chest pain Definition: A disorder characteriz | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care | - | - |
| lon-cardiac chest pain<br>Definition: A disorder characteriz | Mild pain ted by discomfort in the chest unrel | Moderate pain; limiting instrumental ADL lated to a heart disorder. | Severe pain; limiting self care<br>ADL | - | - |
| lon-cardiac chest pain<br>Pefinition: A disorder characteriz | Mild pain ted by discomfort in the chest unrel | Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL Severe pain; limiting self care | - | - |
| lon-cardiac chest pain<br>refinition: A disorder characteriz<br>rain<br>refinition: A disorder characteriz | Mild pain eed by discomfort in the chest unrel | Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL Severe pain; limiting self care | - | - Death |
| on-cardiac chest pain efinition: A disorder characteriz ain efinition: A disorder characteriz udden death NOS | Mild pain ted by discomfort in the chest unrel Mild pain ted by the sensation of marked disc | Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. | Severe pain; limiting self care ADL Severe pain; limiting self care ADL | - | - Death |
| lon-cardiac chest pain Definition: A disorder characteriz Pain Definition: A disorder characteriz Budden death NOS Definition: An unexpected cessa | Mild pain red by discomfort in the chest unrel Mild pain red by the sensation of marked disc - tion of life that cannot be attributed | Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. - to a CTCAE term associated with | Severe pain; limiting self care ADL Severe pain; limiting self care ADL - Grade 5. | Life threatesing and | 1 |
| lon-cardiac chest pain Definition: A disorder characteriz Pain Definition: A disorder characteriz Budden death NOS Definition: An unexpected cessa General disorders and | Mild pain red by discomfort in the chest unrel Mild pain red by the sensation of marked disc - tion of life that cannot be attributed Asymptomatic or mild | Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. - to a CTCAE term associated with Moderate; minimal, local or | Severe pain; limiting self care ADL Severe pain; limiting self care ADL - Grade 5. Severe or medically significant | - Life-threatening consequences; | - Death |
| Jon-cardiac chest pain Definition: A disorder characterized in Definition: A disorder characterized death NOS Definition: An unexpected cessary of the conditions of the condi | Mild pain red by discomfort in the chest unrel Mild pain red by the sensation of marked disc tion of life that cannot be attributed Asymptomatic or mild symptoms; clinical or diagnostic | Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. - Ito a CTCAE term associated with Moderate; minimal, local or noninvasive intervention | Severe pain; limiting self care ADL Severe pain; limiting self care ADL - Grade 5. Severe or medically significant but not immediately life- | - Life-threatening consequences; urgent intervention indicated | 1 |
| Non-cardiac chest pain Definition: A disorder characteriz Pain Definition: A disorder characteriz Budden death NOS Definition: An unexpected cessa General disorders and administration site conditions - | Mild pain ted by discomfort in the chest unrel Mild pain ted by the sensation of marked disc tion of life that cannot be attributed Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention | Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. I to a CTCAE term associated with Moderate; minimal, local or noninvasive intervention indicated; limiting age- | Severe pain; limiting self care ADL Severe pain; limiting self care ADL - Grade 5. Severe or medically significant but not immediately lifethreatening; hospitalization or | | 1 |
| Non-cardiac chest pain Definition: A disorder characteriz Pain Definition: A disorder characteriz Sudden death NOS | Mild pain red by discomfort in the chest unrel Mild pain red by the sensation of marked disc tion of life that cannot be attributed Asymptomatic or mild symptoms; clinical or diagnostic | Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. - Ito a CTCAE term associated with Moderate; minimal, local or noninvasive intervention | Severe pain; limiting self care ADL Severe pain; limiting self care ADL - Grade 5. Severe or medically significant but not immediately life- | | 1 |
| Non-cardiac chest pain Definition: A disorder characteriz Pain Definition: A disorder characteriz Sudden death NOS Definition: An unexpected cessa General disorders and administration site conditions - | Mild pain ted by discomfort in the chest unrel Mild pain ted by the sensation of marked disc tion of life that cannot be attributed Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention | Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. I to a CTCAE term associated with Moderate; minimal, local or noninvasive intervention indicated; limiting age- | Severe pain; limiting self care ADL Severe pain; limiting self care ADL - Grade 5. Severe or medically significant but not immediately lifethreatening; hospitalization or | | 1 |

| | | Hepatobiliary diso | rders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Bile duct stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; IV fluids indicated <24<br>hrs | Severely altered GI function;<br>radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the bile duct. | T | T | |
| Biliary fistula | - | Symptomatic and intervention not indicated | Severely altered GI function;<br>TPN indicated; endoscopic<br>intervention indicated; elective<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the bile ducts and anoth | ner organ or anatomic site. | <b>.</b> | |
| Cholecystitis | - | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation involving the g | allbladder. It may be associated w | vith the presence of gallstones. | • | , |
| Gallbladder fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Symptomatic or severely altered<br>GI function; TPN indicated;<br>radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the gallbladder and and | ther organ or anatomic site. | T | |
| Gallbladder necrosis | - | - | - | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the gallbladder. | | | |
| Gallbladder obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; IV fluids indicated <24<br>hrs | Symptomatic and severely<br>altered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by blockage of the normal flow | of the contents of the gallbladder. | T | I | |
| Gallbladder pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the gallbladder region. | T | T | |
| Gallbladder perforation | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the gallbladder | wall. | 1 | T | |
| Hepatic failure | - | - | Asterixis; mild encephalopathy; limiting self care ADL | Moderate to severe encephalopathy; coma; life-threatening consequences | Death |
| | | etabolize chemicals in the body. La | aboratory test results reveal abnor | rmal plasma levels of ammonia, bi | lirubin, lactic |
| dehydrogenase, and alkaline pho | | O | Towns for the Control of the Control | 1 15- 41 | D" |
| Hepatic hemorrhage | Mild; intervention not indicated | Symptomatic; medical intervention indicated | Transfusion indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the liver. | | | Ī | <u> </u> |
| Hepatic necrosis | - | - | - | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the hepatic parenchyma. | 1 | <b>.</b> | |
| Hepatic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the liver region. | | | |
| Perforation bile duct | - | - | Radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the wall of the e | xtrahepatic or intrahepatic bile du | ct. | | |

| Hepatobiliary disorders | | | | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Portal hypertension | - | Decreased portal vein flow | Reversal/retrograde portal vein flow; associated with varices and/or ascites | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an increase in blood pressu | re in the portal venous system. | | | |
| Portal vein thrombosis | - | Intervention not indicated | Medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the formation of a thrombus | (blood clot) in the portal vein. | • | | |
| Hepatobiliary disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Immune system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Allergic reaction | Transient flushing or rash, drug<br>fever <38 degrees C (<100.4<br>degrees F); intervention not<br>indicated | Intervention or infusion interruption indicated; responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics); prophylactic medications indicated for <=24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an adverse local or general | response from exposure to an alle | ergen.<br>I | T | |
| Anaphylaxis | - | - | Symptomatic bronchospasm,<br>with or without urticaria;<br>parenteral intervention<br>indicated; allergy-related<br>edema/angioedema;<br>hypotension | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an acute inflammatory react<br>presents with breathing difficulty, dia | <del>-</del> | | <del>-</del> | ypersensitivi |
| Autoimmune disorder | Asymptomatic; serologic or other evidence of autoimmune reaction, with normal organ function; intervention not indicated | Evidence of autoimmune reaction involving a non-essential organ or function (e.g., hypothyroidism) | Autoimmune reactions involving major organ (e.g., colitis, anemia, myocarditis, kidney) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder resulting fr tissue constituents. | om loss of function or tissue destru | iction of an organ or multiple orga | ns, arising from humoral or cellula | r immune responses of the individe | ual to his ow |
| Cytokine release syndrome | Mild reaction; infusion interruption not indicated; intervention not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for <=24 hrs | following initial improvement;<br>hospitalization indicated for<br>clinical sequelae (e.g., renal<br>impairment, pulmonary<br>infiltrates) | Life-threatening consequences; pressor or ventilatory support indicated | Death |
| Definition: A disorder characterize | zed by nausea, headache, tachyca | rdia, hypotension, rash, and shorti | ness of breath; it is caused by the | release of cytokines from the cells | i. |
| Serum sickness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate arthralgia; fever, rash, urticaria, antihistamines indicated | Severe arthralgia or arthritis;<br>extensive rash; steroids or IV<br>fluids indicated | Life-threatening consequences; pressor or ventilatory support indicated | Death |
| | zed by a delayed-type hypersensitive foreign antigen. Symptoms include | = : | | | - |
| Immune system disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | 1 |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process involv | ving the abdominal cavity. | | | |
| Anorectal infection | Localized; local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process invol | ving the anal area and the rectum. | 1 | 1 | 1 |
| Appendicitis | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by acute inflammation to the v | ermiform appendix caused by a pa | athogenic agent. | | |
| | -<br>erized by acute inflammation to the v | | | | Death<br>the |
| appendiceal wall. The append | diceal wall rupture causes the release | e of inflammatory and bacterial cor | tents from the appendiceal lumen | into the abdominal cavity. | |
| Arteritis infective | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process involv | ving an artery. | | | |
| Biliary tract infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process involv | ving the biliary tract. | | • | |
| Bladder infection | - | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process involv | ving the bladder. | | | |
| Bone infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | erized by an infectious process invol | ving the bones. | 1 | 1 | |
| Breast infection Definition: A disorder character | erized by an infectious process involv | Local infection with moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | Severe infection; axillary<br>adenitis; IV antibacterial,<br>antifungal, or antiviral<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Bronchial infection | | Moderate symptoms; oral | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| bionamia medion | | intervention indicated (e.g., antibiotic, antifungal, antiviral) | antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | urgent intervention indicated | Deam |
| Definition: A disorder character | erized by an infectious process involv | ving the bronchi. | | | |
| Catheter related infection | - | Localized; local intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | erized by an infectious process that a | arises secondary to catheter use. | | | 1 |
| Cecal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| Infections and infestations | | | | | |
|---|---|---|---|---|---|
| | | | Grade | Т | I |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterize | ed by an infectious process i | nvolving the cecum. | | | |
| Cervicitis infection Definition: A disorder characterize | ad by an infectious process is | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by an infectious process i | | n | | - · |
| Conjunctivitis infective | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process i | nvolving the conjunctiva. Clinical manif | estations include pink or red color | in the eyes. | |
| Corneal infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process i | nvolving the cornea. | 1 | | |
| Cranial nerve infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process i | nvolving a cranial nerve. | 1 | <u> </u> | |
| Device related infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process i | nvolving the use of a medical device. | | | |
| Duodenal infection | - | Moderate symptoms; medical intervention indicated (e.g., oral antibiotics) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process i | nvolving the duodenum. | | | |
| Encephalitis infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>severe changes in mental<br>status; self-limited seizure<br>activity; focal neurologic<br>abnormalities | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process i | nvolving the brain tissue. | | | |
| Encephalomyelitis infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process i | nvolving the brain and spinal cord tissu | es. | | |
| Endocarditis infective | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process i | nvolving the endocardial layer of the he | eart. | | |
| | | Local intervention indicated | Systemic intervention or | Blindness (20/200 or worse) | |

| Infections and infestations | | | | | |
|---|---|---|---|---|---|
| | | T | Grade | Г | 1 |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Enterocolitis infectious | - | Passage of >3 unformed stools<br>per 24 hrs or duration of illness<br>>48 hrs; moderate abdominal<br>pain | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated;<br>profuse watery diarrhea with | Life-threatening consequences; urgent intervention indicated | Death |
| | | | signs of hypovolemia; bloody<br>diarrhea; fever; severe<br>abdominal pain; hospitalization<br>indicated | | |
| Definition: A disorder characteriz | zed by an infectious process involv | ing the small and large intestines. | 1 | | |
| Esophageal infection | - | Local intervention indicated (e.g., oral antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ing the esophagus. | _ | | |
| Eye infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated;<br>enucleation | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ing the eye. | | | 1 |
| Gallbladder infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ing the gallbladder. | | | |
| Gum infection | Local therapy indicated (swish and swallow) | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ing the gums. | | | |
| Hepatic infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ing the liver. | ' | • | , |
| Hepatitis viral | Asymptomatic, treatment not indicated | - | Symptomatic liver dysfunction;<br>fibrosis by biopsy; compensated<br>cirrhosis; reactivation of chronic<br>hepatitis | Decompensated liver function<br>(e.g., ascites, coagulopathy,<br>encephalopathy, coma) | Death |
| Definition: A disorder characteriz | zed by a viral pathologic process in | volving the liver parenchyma. | | | |
| Infective myositis | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ing the skeletal muscles. | | | |
| Joint infection | - | Localized; local intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral); needle aspiration indicated (single or multiple) | Arthroscopic intervention indicated (e.g., drainage) or arthrotomy (e.g., open surgical drainage) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ing a joint. | | | |
| Kidney infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ।<br>zed by an infectious process involv | 1 | 1 . | 1 | I . |

| Infections and infestations | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Laryngitis | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an inflammatory process | involving the larynx. | _ | 1 | |
| Lip infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder charac | terized by an infectious process invo | olving the lips. | _ | 1 | |
| Lung infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an infectious process invo | olving the lungs. | T | | |
| Lymph gland infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an infectious process invo | olving the lymph nodes. | I | | |
| Mediastinal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an infectious process invo | olving the mediastinum. | T | | |
| Meningitis | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated; focal<br>neurologic deficit | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | terized by acute inflammation of the | meninges of the brain and/or spinal | cord. | • | , |
| Mucosal infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an infectious process invo | olving a mucosal surface. | ' | • | , |
| Nail infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder charac | terized by an infectious process invo | olving the nail. | T | 1 | |
| Otitis externa | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | | olving the outer ear and ear canal. C | · | ive water exposure (swimmer's ea | r infection) |
| Otitis media | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an infectious process invo | olving the middle ear. | · | · | |
| Ovarian infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | 1 | i i | 1 | İ | 1 |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pancreas infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involvi | ing the pancreas. | 1 | 1 | |
| Papulopustular rash | Papules and/or pustules covering <10% BSA, which may or may not be associated with symptoms of pruritus or tenderness | Papules and/or pustules covering 10-30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self-care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| | zed by an eruption consisting of pa | | | | o, and upper |
| Paronychia | s rash does not present with whiteh Nail fold edema or erythema; disruption of the cuticle | Localized intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral); nail fold edema or erythema with pain; associated with discharge or nail plate separation; limiting instrumental ADL | Surgical intervention or IV antibiotics indicated; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by an infectious process involving | ing the soft tissues around the nai | l.<br>I | T | |
| Pelvic infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involvi | ing the pelvic cavity. | T | T | |
| Penile infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involvi | ing the penis. | 1 | 1 | |
| Periorbital infection | -<br>ized by an infectious process involvi | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Peripheral nerve infection | Zed by all lillections process lilvolvi | Localized; local intervention | IV antibiotic, antifungal, or | Life threatening consequences: | Death |
| | zed by an infectious process involvi | indicated (e.g., topical antibiotic, antifungal, or antiviral) | antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Peritoneal infection | | | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| r entonear infection | | | antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involvi | ing the peritoneum. | | _ | |
| Pharyngitis | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by inflammation of the throat. | 1 | 1 | 1 | 1 |
| Phlebitis infective | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterize of the infected vein. | zed by an infectious process involv | ing the vein. Clinical manifestation | is include erythema, marked disco | mfort, swelling, and induration alo | ng the course |
| Pleural infection | - led by an infectious process involved | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an infectious process involv | | N/ | | D4b |
| Prostate infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an infectious process involv | ing the prostate gland. | T | 1 | |
| Rash pustular | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder characterize | red by a circumscribed and elevate | ed skin lesion filled with pus. | | | |
| Rhinitis infective | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | - | - | - |
| | zed by an infectious process involv | ing the nasal mucosal. | T | T | 1 |
| Salivary gland infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an infectious process involv | ing the salivary gland. | • | | |
| Scrotal infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an infectious process involv | ing the scrotum. | | | |
| Sepsis | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the presence of pathogenic | microorganisms in the blood stream | m that cause a rapidly progressin | g systemic reaction that may lead | to shock. |
| Sinusitis | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | red by an infectious process involv | ing the mucous membranes of the | paranasal sinuses. | T | |
| Skin infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | red by an infectious process involv | ing the skin. | Т | Т | |
| Small intestine infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ing the small intestine. | | | |
| Soft tissue infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by an infectious process involv | ing soft tissues. | • | 1 | 1 |
| Splenic infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| | Infections and infestations | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the spleen. | | | |
| Stoma site infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing a stoma (surgically created op | ening on the surface of the body). | | |
| Tooth infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involving | ing a tooth. | Т | T | |
| Tracheitis | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the trachea. | T | T | |
| Upper respiratory infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the upper respiratory tract (nos | se, paranasal sinuses, pharynx, la | rynx, or trachea). | 1 |
| Urethral infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the urethra. | | | |
| Urinary tract infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the urinary tract, most commo | nly the bladder and the urethra. | | |
| Uterine infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the endometrium. It may exten | d to the myometrium and parame | trial tissues. | |
| Vaginal infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the vagina. | | | |
| Vulval infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the vulva. | | | |
| Wound infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the wound. | T | T | |
| Infections and infestations -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Injury | , poisoning and procedu | ral complications | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Ankle fracture | Mild; non-surgical intervention indicated | Limiting instrumental ADL; operative intervention indicated | Limiting self care ADL; elective surgery indicated | - | - |
| Definition: A finding of damage to affected leg and foot. | the ankle joint characterized by a | a break in the continuity of the ank | le bone. Symptoms include marke | d discomfort, swelling and difficult | moving the |
| Aortic injury | - | - | Severe symptoms; limiting self care ADL; disabling; repair or revision indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | the aorta. | T | T | T | |
| Arterial injury | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic (e.g., claudication); repair or revision not indicated | Severe symptoms; limiting self<br>care ADL; disabling; repair or<br>revision indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | an artery. | 1 | T | | |
| Biliary anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | f bile due to breakdown of a biliary | anastomosis (surgical connection | of two separate anatomic structu | res). | |
| Bladder anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | furine due to breakdown of a blad | der anastomosis (surgical connec | tion of two separate anatomic stru | ctures). | 1 |
| Bruising | Localized or in a dependent area | Generalized | - | - | - |
| Definition: A finding of injury of th | e soft tissues or bone characterize | ed by leakage of blood into surrou | nding tissues. | | |
| Burn | Minimal symptoms; intervention not indicated | Medical intervention; minimal debridement indicated | Moderate to major debridement or reconstruction indicated | Life-threatening consequences | Death |
| <u> </u> | ntegrity to the anatomic site of an a<br>depends on the length and intensi | | an be caused by exposure to cher<br>sion of treatment. | nicals, direct heat, electricity, flame | es and |
| Dermatitis radiation | Faint erythema or dry desquamation | Moderate to brisk erythema;<br>patchy moist desquamation,<br>mostly confined to skin folds<br>and creases; moderate edema | Moist desquamation in areas<br>other than skin folds and<br>creases; bleeding induced by<br>minor trauma or abrasion | Life-threatening consequences;<br>skin necrosis or ulceration of full<br>thickness dermis; spontaneous<br>bleeding from involved site; skin<br>graft indicated | Death |
| Definition: A finding of cutaneous | inflammatory reaction occurring a | as a result of exposure to biologica | ally effective levels of ionizing radia | ation. | |
| Esophageal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of an esophagea | l anastomosis (surgical connection | of two separate anatomic structu | res). | 1 |
| Fall | Minor with no resultant injuries; intervention not indicated | Symptomatic; noninvasive intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding of sudden me | ovement downward, usually result | ing in injury. | T | | |
| Fallopian tube anastomotic leak | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a fallopian tub | e anastomosis (surgical connectio | n of two separate anatomic structu | ıres). | |
| Fallopian tube perforation | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., organ resection) | Death |
| Definition: A finding of rupture of | the fallopian tube wall. | | | | |
| Fracture | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic but non-displaced; immobilization indicated | Severe symptoms; displaced or open wound with bone exposure; disabling; operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of traumatic | injury to the bone in which the con | tinuity of the bone is broken. | , | | • |

| | , | , poisoning and procedu | | | |
|---|---|---|---|---|---|
| | | | Grade | | 1 |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| astric anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | observations only; intervention not indicated | intervention indicated | endoscopic or elective operative | urgent operative intervention indicated | |
| 6 W A 6 W 60 A | 1 | | intervention indicated | Indicated | 1 |
| efinition: A finding of leakage d | ue to breakdown of a gastric anas | 1 | o separate anatomic structures). | | |
| astrointestinal anastomotic | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| eak | observations only; intervention | intervention indicated | endoscopic or elective operative | urgent operative intervention | |
| | not indicated | | intervention indicated | indicated | l |
| efinition: A finding of leakage d | ue to breakdown of a gastrointesti | nal anastomosis (surgical connect | tion of two separate anatomic struc | ctures). | |
| Gastrointestinal stoma necrosis | - | Superficial necrosis; | Severe symptoms; | Life-threatening consequences; | Death |
| | | intervention not indicated | hospitalization or elective | urgent intervention indicated | |
| | | | operative intervention indicated | | |
| efinition: A finding of a necrotic | process occurring in the gastroint | estinal tract stoma. | 1 | | |
| lip fracture | - | Hairline fracture; mild pain; | Severe pain; hospitalization or | Life-threatening consequences; | - |
| | | limiting instrumental ADL; non- | intervention indicated for pain | symptoms associated with | |
| | | surgical intervention indicated | control (e.g., traction); operative | neurovascular compromise | |
| | | | intervention indicated | | ļ |
| Definition: A finding of traumatic | injury to the hip in which the contin | nuity of either the femoral head, fe | moral neck, intertrochanteric or su | btrochanteric regions is broken. | |
| njury to carotid artery | - | - | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| | | | care ADL (e.g., transient | urgent intervention indicated | |
| | | | cerebral ischemia); repair or | | |
| | | | revision indicated | | l |
| efinition: A finding of damage to | o the carotid artery. | T | 1 | | 1 |
| njury to inferior vena cava | - | - | - | Life-threatening consequences; | Death |
| | | | | urgent intervention indicated | |
| Definition: A finding of damage to | o the inferior vena cava. | | 1 | | |
| njury to jugular vein | - | - | Symptomatic limiting self care | Life-threatening consequences; | Death |
| | | | ADL; disabling; repair or | urgent intervention indicated | |
| | | | revision indicated | | |
| Definition: A finding of damage to | o the jugular vein. | | | | |
| njury to superior vena cava | Asymptomatic diagnostic | Symptomatic; repair or revision | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| | finding; intervention not | not indicated | care ADL; disabling; repair or | evidence of end organ damage; | |
| | | | | evidence of end organi damage, | |
| | indicated | | revision indicated | urgent operative intervention | |
| | indicated | | revision indicated | | |
| Definition: A finding of damage to | | | revision indicated | urgent operative intervention | |
| | | Symptomatic; medical | revision indicated Severe symptoms; radiologic, | urgent operative intervention | Death |
| | o the superior vena cava. | Symptomatic; medical intervention indicated | | urgent operative intervention indicated | Death |
| | o the superior vena cava. Asymptomatic diagnostic | * ' | Severe symptoms; radiologic, | urgent operative intervention indicated Life-threatening consequences; | Death |
| ntestinal stoma leak | o the superior vena cava. Asymptomatic diagnostic observations only; intervention | intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention | Death |
| ntestinal stoma leak | Asymptomatic diagnostic observations only; intervention not indicated | intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated | |
| ntestinal stoma leak<br>Definition: A finding of leakage o | Asymptomatic diagnostic observations only; intervention not indicated | intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention | Death |
| ntestinal stoma leak<br>Definition: A finding of leakage o | Asymptomatic diagnostic observations only; intervention not indicated | intervention indicated (surgically created opening on the Self-limited; intervention not | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; | |
| ntestinal stoma leak<br>Definition: A finding of leakage o | Asymptomatic diagnostic observations only; intervention not indicated | intervention indicated (surgically created opening on the Self-limited; intervention not | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention | |
| ntestinal stoma leak<br>Definition: A finding of leakage o<br>ntestinal stoma obstruction | Asymptomatic diagnostic observations only; intervention not indicated | intervention indicated (surgically created opening on the Self-limited; intervention not indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention | |
| ntestinal stoma leak Definition: A finding of leakage o ntestinal stoma obstruction Definition: A finding of blockage | Asymptomatic diagnostic observations only; intervention not indicated f contents from an intestinal stoma - | intervention indicated (surgically created opening on the Self-limited; intervention not indicated of the intestinal stoma. | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative intervention indicated | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated | Death |
| ntestinal stoma leak Definition: A finding of leakage on testinal stoma obstruction Definition: A finding of blockage | Asymptomatic diagnostic observations only; intervention not indicated f contents from an intestinal stoma | intervention indicated (surgically created opening on the Self-limited; intervention not indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative intervention indicated Severe bleeding; transfusion | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; | |
| ntestinal stoma leak Definition: A finding of leakage on testinal stoma obstruction Definition: A finding of blockage | Asymptomatic diagnostic observations only; intervention not indicated f contents from an intestinal stoma - of the normal flow of the contents Minimal bleeding identified on | intervention indicated (surgically created opening on the Self-limited; intervention not indicated of the intestinal stoma. Moderate bleeding; medical | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative intervention indicated | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated | Death |
| ntestinal stoma leak Definition: A finding of leakage on testinal stoma obstruction Definition: A finding of blockage | Asymptomatic diagnostic observations only; intervention not indicated f contents from an intestinal stoma - of the normal flow of the contents Minimal bleeding identified on clinical exam; intervention not | intervention indicated (surgically created opening on the Self-limited; intervention not indicated of the intestinal stoma. Moderate bleeding; medical | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative intervention indicated Severe bleeding; transfusion indicated; radiologic or | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; | Death |
| Definition: A finding of leakage on testinal stoma obstruction Definition: A finding of blockage of the stoma site bleeding | Asymptomatic diagnostic observations only; intervention not indicated f contents from an intestinal stome - of the normal flow of the contents Minimal bleeding identified on clinical exam; intervention not indicated | intervention indicated (surgically created opening on the Self-limited; intervention not indicated of the intestinal stoma. Moderate bleeding; medical | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative intervention indicated Severe bleeding; transfusion indicated; radiologic or endoscopic intervention | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; | Death |
| Definition: A finding of leakage on testinal stoma obstruction Definition: A finding of blockage on testinal stoma site bleeding Definition: A finding of blood leak | Asymptomatic diagnostic observations only; intervention not indicated f contents from an intestinal stoma - of the normal flow of the contents Minimal bleeding identified on clinical exam; intervention not indicated | intervention indicated (surgically created opening on the Self-limited; intervention not indicated of the intestinal stoma. Moderate bleeding; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative intervention indicated Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of leakage on testinal stoma obstruction Definition: A finding of blockage ontestinal stoma site bleeding Definition: A finding of blood leak | Asymptomatic diagnostic observations only; intervention not indicated f contents from an intestinal stoma - of the normal flow of the contents Minimal bleeding identified on clinical exam; intervention not indicated rage from the intestinal stoma. Primary repair of injured | intervention indicated (surgically created opening on the Self-limited; intervention not indicated of the intestinal stoma. Moderate bleeding; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative intervention indicated Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated Complete resection or | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of leakage on testinal stoma obstruction Definition: A finding of blockage on testinal stoma site bleeding Definition: A finding of blood leak | Asymptomatic diagnostic observations only; intervention not indicated f contents from an intestinal stoma - of the normal flow of the contents Minimal bleeding identified on clinical exam; intervention not indicated | intervention indicated (surgically created opening on the Self-limited; intervention not indicated of the intestinal stoma. Moderate bleeding; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative intervention indicated Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of leakage on testinal stoma obstruction Definition: A finding of blockage on testinal stoma site bleeding Definition: A finding of blood leak | Asymptomatic diagnostic observations only; intervention not indicated f contents from an intestinal stoma - of the normal flow of the contents Minimal bleeding identified on clinical exam; intervention not indicated rage from the intestinal stoma. Primary repair of injured | intervention indicated (surgically created opening on the Self-limited; intervention not indicated of the intestinal stoma. Moderate bleeding; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative intervention indicated Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated Complete resection or reconstruction of injured | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of leakage on testinal stoma obstruction Definition: A finding of blockage ontestinal stoma site bleeding Definition: A finding of blood leak ontraoperative arterial injury | Asymptomatic diagnostic observations only; intervention not indicated f contents from an intestinal stoma - of the normal flow of the contents Minimal bleeding identified on clinical exam; intervention not indicated age from the intestinal stoma. Primary repair of injured organ/structure indicated | intervention indicated (surgically created opening on the Self-limited; intervention not indicated of the intestinal stoma. Moderate bleeding; medical intervention indicated Partial resection of injured organ/structure indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative intervention indicated Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated Complete resection or reconstruction of injured organ/structure indicated; | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of leakage of intestinal stoma obstruction Definition: A finding of blockage intestinal stoma site bleeding Definition: A finding of blood leak intraoperative arterial injury | Asymptomatic diagnostic observations only; intervention not indicated f contents from an intestinal stoma - of the normal flow of the contents Minimal bleeding identified on clinical exam; intervention not indicated rage from the intestinal stoma. Primary repair of injured organ/structure indicated o an artery during a surgical proce | intervention indicated (surgically created opening on the Self-limited; intervention not indicated of the intestinal stoma. Moderate bleeding; medical intervention indicated Partial resection of injured organ/structure indicated dure. | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative intervention indicated Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated Complete resection or reconstruction of injured organ/structure indicated; disabling | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death Death |
| Definition: A finding of leakage of intestinal stoma obstruction Definition: A finding of blockage intestinal stoma site bleeding Definition: A finding of blood leak intraoperative arterial injury | Asymptomatic diagnostic observations only; intervention not indicated f contents from an intestinal stoma - of the normal flow of the contents Minimal bleeding identified on clinical exam; intervention not indicated rage from the intestinal stoma. Primary repair of injured organ/structure indicated o an artery during a surgical proce | intervention indicated (surgically created opening on the Self-limited; intervention not indicated of the intestinal stoma. Moderate bleeding; medical intervention indicated Partial resection of injured organ/structure indicated dure. Partial resection of injured | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative intervention indicated Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated Complete resection or reconstruction of injured organ/structure indicated; disabling Complete resection or | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of leakage on testinal stoma obstruction Definition: A finding of blockage ontestinal stoma site bleeding Definition: A finding of blood leak ontraoperative arterial injury | Asymptomatic diagnostic observations only; intervention not indicated f contents from an intestinal stoma - of the normal flow of the contents Minimal bleeding identified on clinical exam; intervention not indicated rage from the intestinal stoma. Primary repair of injured organ/structure indicated o an artery during a surgical proce | intervention indicated (surgically created opening on the Self-limited; intervention not indicated of the intestinal stoma. Moderate bleeding; medical intervention indicated Partial resection of injured organ/structure indicated dure. | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated e surface of the body). Severe symptoms; IV fluids, tube feeding, or TPN indicated >=24 hrs; elective operative intervention indicated Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated Complete resection or reconstruction of injured organ/structure indicated; disabling | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death Death |

| Injury, poisoning and procedural complications | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A finding of damage to | the breast parenchyma during a | surgical procedure. | 1 | | |
| Intraoperative cardiac injury | the heart during a surgical pressure | - | Primary repair of injured organ/structure indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | the heart during a surgical proce | | | | <b>.</b> |
| Intraoperative ear injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection of injured organ/structure indicated; disabling (e.g., impaired hearing; impaired balance) | Life-threatening consequences; urgent intervention indicated | Death |
| | the ear during a surgical procedu | | | | |
| Intraoperative endocrine injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the endocrine gland during a sur | gical procedure. | | | |
| Intraoperative gastrointestinal injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the gastrointestinal system durin | g a surgical procedure. | | | |
| Intraoperative head and neck injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the head and neck during a surg | ical procedure. | | | |
| Intraoperative hemorrhage | - | - | Postoperative radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of uncontrolle | ed bleeding during a surgical proc | edure. | | | |
| Intraoperative hepatobiliary injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the hepatic parenchyma and/or l | piliary tract during a surgical pro | cedure. | | |
| Intraoperative musculoskeletal injury Definition: A finding of damage to | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Intraoperative neurological | Primary repair of injured | Partial resection of injured | Complete resection or | Life threatening consequences: | Death |
| injury | organ/structure indicated | organ/structure indicated | reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| - | the nervous system during a sur | - | O-market " | Life there to | D" |
| Intraoperative ocular injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the eye during a surgical proced | | 1 | | |
| Intraoperative renal injury | Primary repair of injured organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the kidney during a surgical proc | edure. | • | • | • |
| Intraoperative reproductive tract injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |

| | Injury | , poisoning and procedu | ral complications | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A finding of damage to | the reproductive organs during a | surgical procedure. | | | 1 |
| Intraoperative respiratory injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the respiratory system during a s | surgical procedure. | T | T | |
| Intraoperative skin injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the skin during a surgical proced | ure. | | | |
| Intraoperative splenic injury | - | Primary repair of injured organ/structure indicated | Resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | the spleen during a surgical prod | | | | Ι |
| Intraoperative urinary injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | the urinary system during a surg | | | | I |
| Intraoperative venous injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | a vein during a surgical procedu | e. | _ | | |
| Kidney anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | f urine due to breakdown of a kidn | ey anastomosis (surgical connecti | on of two separate anatomic struc | tures). | |
| Large intestinal anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of an anastomos | is (surgical connection of two sepa | arate anatomic structures) in the la | rge intestine. | |
| Pancreatic anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a pancreatic a | nastomosis (surgical connection o | f two separate anatomic structures | s). | |
| Pharyngeal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | | · - | of two separate anatomic structure | 1 | D .: |
| Postoperative hemorrhage | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; radiologic,<br>endoscopic, or operative<br>intervention indicated | Transfusion indicated of >=2 units (10 cc/kg for pediatrics) pRBCs beyond protocol specification; urgent radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of bleeding of | occurring after a surgical procedure | e.<br>T | T | T | |
| Postoperative thoracic procedure complication | - | Extubated within 24 - 72 hrs postoperatively | Extubated >72 hrs<br>postoperatively, but before<br>tracheostomy indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A finding of a previous | sly undocumented problem that oc | | T | T | |
| Prolapse of intestinal stoma | Asymptomatic; reducible | Recurrent after manual<br>reduction; local irritation or stool<br>leakage; difficulty to fit<br>appliance; limiting instrumental<br>ADL | Severe symptoms; elective operative intervention indicated; limiting self care ADL | Life-threatening consequences; urgent operative intervention indicated | Death |

| | Injury | , poisoning and procedu | ral complications | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A finding of protrusion | of the intestinal stoma (surgically | created opening on the surface of | the body) above the abdominal su | urface. | 1 |
| Prolapse of urostomy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Local care or maintenance;<br>minor revision indicated | Dysfunctional stoma; elective operative intervention or major stomal revision indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of displacem | ent of the urostomy. | 1 | T | T | 1 |
| Radiation recall reaction<br>(dermatologic) | Faint erythema or dry<br>desquamation | Moderate to brisk erythema;<br>patchy moist desquamation,<br>mostly confined to skin folds<br>and creases; moderate edema | Moist desquamation in areas<br>other than skin folds and<br>creases; bleeding induced by<br>minor trauma or abrasion | Life-threatening consequences;<br>skin necrosis or ulceration of full<br>thickness dermis; spontaneous<br>bleeding from involved site; skin<br>graft indicated | Death |
| Definition: A finding of acute skir | inflammatory reaction caused by | drugs, especially chemotherapeut | ic agents, for weeks or months fol | lowing radiotherapy. The inflamma | atory reaction |
| is confined to the previously irrac | diated skin and the symptoms disa | ppear after the removal of the pha | rmaceutical agent. | T | 1 |
| Rectal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a rectal anasto | pmosis (surgical connection of two | separate anatomic structures). | _ | |
| Seroma | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; simple aspiration indicated | Symptomatic, elective radiologic or operative intervention indicated | - | - |
| Definition: A finding of tumor-like | collection of serum in the tissues. | T | Τ | T | |
| Small intestinal anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of an anastomos | is (surgical connection of two sepa | arate anatomic structures) in the si | mall bowel. | 1 |
| Spermatic cord anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a spermatic co | ord anastomosis (surgical connecti | on of two separate anatomic struc | tures). | 1 |
| Spinal fracture | Mild back pain; nonprescription analgesics indicated | Moderate back pain;<br>prescription analgesics<br>indicated; limiting instrumental<br>ADL | Severe back pain;<br>hospitalization or intervention<br>indicated for pain control (e.g.,<br>vertebroplasty); limiting self care<br>ADL; disability | Life-threatening consequences; symptoms associated with neurovascular compromise | Death |
| Definition: A finding of traumatic | injury to the spine in which the cor | ntinuity of a vertebral bone is broke | en. | • | , |
| Stenosis of gastrointestinal stoma | - | Symptomatic; IV fluids indicated <24 hrs; manual dilation at bedside | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of narrowing | of the gastrointestinal stoma (surg | gically created opening on the surf | ace of the body). | <u> </u> | 1 |
| Stomal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| | red by a circumscribed, inflammato | ory and necrotic erosive lesion on t | the jejunal mucosal surface close t | to the anastomosis site following a | |
| gastroenterostomy procedure. | No. 111 P. 11 P. 11 | M 1 / 11 / 11 / 11 / 11 / 11 | 0 11 11 11 11 11 | | D # |
| Tracheal hemorrhage | Minimal bleeding identified on clinical or diagnostic exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of bleeding f | rom the trachea. | Т | Т | Т | |
| Tracheal obstruction | Partial asymptomatic<br>obstruction on examination<br>(e.g., visual, radiologic or<br>endoscopic) | Symptomatic (e.g., noisy airway breathing), no respiratory distress; medical intervention indicated (e.g., steroids); limiting instrumental ADL | Stridor; radiologic or endoscopic intervention indicated (e.g., stent, laser); limiting self care ADL | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A finding of blockage | of the lumen of the trachea. | | | | |

| Injury, poisoning and procedural complications | | | | | |
|---|---|---|---|---|---|
| Grade Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Tracheostomy site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of blood leak | age from the tracheostomy site. | _ | _ | | |
| Ureteric anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a ureteral ana | stomosis (surgical connection of tw | vo separate anatomic structures). | I | |
| Urethral anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a urethral ana | stomosis (surgical connection of tw | vo separate anatomic structures). | 1 | |
| Urostomy leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | f contents from a urostomy. | | | | |
| Urostomy obstruction | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; dilation or endoscopic repair or stent placement indicated | Altered organ function (e.g.,<br>sepsis or hydronephrosis, or<br>renal dysfunction); elective<br>operative intervention indicated | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A finding of blockage | of the urostomy. | | | | |
| Urostomy site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of bleeding for | rom the urostomy site. | ' | • | • | • |
| Urostomy stenosis | - | Symptomatic but no<br>hydronephrosis, no sepsis or no<br>renal dysfunction; dilation or<br>endoscopic repair or stent<br>placement indicated | Symptomatic (e.g.,<br>hydronephrosis, or renal<br>dysfunction); elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of narrowing | of the opening of a urostomy. | 1. | 1 | ı | 1 |
| Uterine anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a uterine anas | tomosis (surgical connection of tw | o separate anatomic structures). | | |
| Uterine perforation | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the uterine wall. | | | | |
| Vaginal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a vaginal anas | tomosis (surgical connection of tw | o separate anatomic structures). | | |
| Vas deferens anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a vas deferens | s anastomosis (surgical connection | of two separate anatomic structu | res). | |
| /ascular access complication | - | Device dislodgement, blockage, leak, or malposition; device replacement indicated | Deep vein or cardiac<br>thrombosis; intervention<br>indicated (e.g., anticoagulation,<br>lysis, filter, invasive procedure) | Embolic event including pulmonary embolism or life-threatening thrombus | Death |
| | I. | I | 1 ,,ass procedure) | I | 1 |

| | Injury | , poisoning and procedu | ral complications | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Venous injury Definition: A finding of damage t | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic (e.g., claudication); repair or revision not indicated | Severe symptoms; limiting self care ADL; repair or revision indicated; disabling | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Wound complication | Incisional separation of <=25% | Incisional separation >25% of | Hernia without evidence of | Hernia with evidence of | Death |
| would complication | of wound, no deeper than superficial fascia | wound; local care indicated | strangulation; fascial<br>disruption/dehiscence; primary<br>wound closure or revision by | strangulation; major<br>reconstruction flap, grafting,<br>resection, or amputation<br>indicated | Death |
| Definition: A finding of developm | ent of a new problem at the site of | an existing wound. | | | |
| Wound dehiscence | Incisional separation of <=25% of wound, no deeper than superficial fascia | Incisional separation >25% of<br>wound with local care;<br>asymptomatic hernia or<br>symptomatic hernia without<br>evidence of strangulation | without evisceration; primary wound closure or revision by operative intervention indicated | Life-threatening consequences; symptomatic hernia with evidence of strangulation; fascial disruption with evisceration; major reconstruction flap, grafting, resection, or amputation indicated | Death |
| Definition: A finding of separatio | n of the approximated margins of a | surgical wound. | | | |
| Wrist fracture | Mild; non-surgical intervention indicated | Limiting instrumental ADL; operative intervention indicated | Limiting self care ADL; elective surgery indicated | - | - |
| Definition: A finding of traumatic | injury to the wrist joint in which the | continuity of a wrist bone is broke | en. | | |
| Injury, poisoning and procedural<br>complications - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Investigations | 5 | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Activated partial thromboplastin ime prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage | - | - |
| | y test result in which the partial th<br>may occur in a variety of disease | = | reater than the control value. As a related to treatment. | possible indicator of coagulopat | hy, a prolonge |
| Alanine aminotransferase | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| | l<br>oratory test results that indicate a | l<br>n increase in the level of alanine a | I<br>minotransferase (ALT or SGPT) ir | I<br>n the blood specimen. | |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of alkaline p | phosphatase in a blood specimen. | | |
| Aspartate aminotransferase<br>ncreased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | increase in the level of aspartate | aminotransferase (AST or SGOT | i) in a blood specimen. | 1 |
| Blood antidiuretic hormone<br>abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | ।<br>bnormal levels of antidiuretic horm | none in the blood specimen. | I | 1 |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | '<br>n abnormally high level of bilirubin | in the blood. Excess bilirubin is as | ssociated with jaundice. | 1 |
| Blood corticotrophin decreased | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | ,<br>n decrease in levels of corticotropl | hin in a blood specimen. | ' | ' |
| Blood gonadotrophin abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of gonadotrophin h | ormone in a blood specimen. | | |
| Blood prolactin abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | ।<br>bnormal levels of prolactin hormor | ı<br>ne in a blood specimen. | I | ! |
| Carbon monoxide diffusing | 3 - 5 units below LLN; for follow- | 6 - 8 units below LLN; for follow- | Asymptomatic decrease of >8 | - | - |
| capacity decreased | up, a decrease of 3 - 5 units<br>(ml/min/mm Hg) below the<br>baseline value | up, an asymptomatic decrease<br>of >5 - 8 units (ml/min/mm Hg)<br>below the baseline value | units drop; >5 units drop along<br>with the presence of pulmonary<br>symptoms (e.g. , >Grade 2<br>hypoxia or >Grade 2 or higher<br>dyspnea) | | |
| Definition: A finding based on lun | g function test results that indicate | a decrease in the lung capacity | to absorb carbon monoxide. | T | |
| Cardiac troponin I increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer | - | - |
| | t which indicates increased levels | of cardiac troponin I in a biologica | 1 | | |
| Cardiac troponin T increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer | - | - |
| Definition: A laboratory test result | t which indicates increased levels | of cardiac troponin T in a biologica | al specimen. | • | • |
| CD4 lymphocytes decreased | <lln -="" 0.5="" 500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200 - 50/mm3; <0.2 x 0.05 -<br>10e9 /L | <50/mm3; <0.05 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of CD4 lymph | nocytes in a blood specimen. | • | • |
| Cholesterol high | - | >300 - 400 mg/dL; >7.75 - 10.34 mmol/L | 1 | >500 mg/dL; >12.92 mmol/L | - |
| Definition: A finding based on lab | i<br>oratory test results that indicate hi | igher than normal levels of cholest | 1 | ·<br>I | <u>'</u> |
| CPK increased | >ULN - 2.5 x ULN | >2.5 x ULN - 5 x ULN | >5 x ULN - 10 x ULN | >10 x ULN | - |

| | | Investigations | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Creatinine increased | >1 - 1.5 x baseline; >ULN - 1.5 | >1.5 - 3.0 x baseline; >1.5 - 3.0 | >3.0 baseline; >3.0 - 6.0 x ULN | >6.0 x ULN | - |
| Definition: A finding based on lab | x ULN | x ULN | ialasiaal anasiman | | 1 |
| | oratory test results that indicate in | | | | |
| Ejection fraction decreased | - | Resting ejection fraction (EF) 50 - 40%; 10 - 19% drop from baseline | Resting ejection fraction (EF) 39 - 20%; >20% drop from baseline | | - |
| Definition: The percentage compount contraction. | uted when the amount of blood ejલ | ected during a ventricular contracti | on of the heart is compared to the | amount that was present prior to | the |
| Electrocardiogram QT corrected interval prolonged | | QTc 481 - 500 ms | ' | QTc >= 501 or >60 ms change<br>from baseline and Torsade de<br>pointes or polymorphic<br>ventricular tachycardia or<br>signs/symptoms of serious<br>arrhythmia | - |
| | dysrhythmia characterized by an a | bnormally long corrected Q1 inter | | | |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 - 0.25 x LLN or 50 - <75% decrease from baseline | <0.25 x LLN or 75% decrease<br>from baseline or absolute value<br><50 mg/dL | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of fibrinogen i | n a blood specimen. | | |
| Forced expiratory volume decreased | FEV1% (percentages of<br>observed FEV1 and FVC<br>related to their respective<br>predicted values) 99 - 70%<br>predicted | FEV1 60 - 69% | 50 - 59% | <= 49% | - |
| Definition: A finding based on tes | t results that indicate a relative de | crease in the fraction of the forced | l vital capacity that is exhaled in a | specific number of seconds. | |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate hi | gher than normal levels of the enz | yme gamma-glutamyltransferase | '<br>in the blood specimen. GGT (gam | ima- |
| glutamyltransferase ) catalyzes th | ne transfer of a gamma glutamyl g | roup from a gamma glutamyl pept | ide to another peptide, amino acid | s or water. | |
| Growth hormone abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate al | onormal levels of growth hormone | in a biological specimen. | | |
| Haptoglobin decreased | <lln< td=""><td>-</td><td>-</td><td>-</td><td>-</td></lln<> | - | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of haptoglobir | n in a blood specimen. | | |
| Hemoglobin increased | Increase in >0 - 2 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | Increase in >2 - 4 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | Increase in >4 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | - | - |
| Definition: A finding based on lab | oratory test results that indicate in | creased levels of hemoglobin in a | biological specimen. | | |
| INR increased | >1 - 1.5 x ULN; >1 - 1.5 times<br>above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN; >1.5 - 2.5<br>times above baseline if on<br>anticoagulation | >2.5 x ULN; >2.5 times above baseline if on anticoagulation | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the ratio of the patier | t's prothrombin time to a control s | ample in the blood. | |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of lipase in | a biological specimen. | | |
| Lymphocyte count decreased | <lln -="" 0.8="" 800="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <800 - 500/mm3; <0.8 - 0.5 x<br>10e9 /L | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200/mm3; <0.2 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of lymphocyte | es in a blood specimen. | | 1 |
| Lymphocyte count increased | - | >4000/mm3 - 20,000/mm3 | >20,000/mm3 | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n abnormal increase in the numbe | r of lymphocytes in the blood, effu | sions or bone marrow. | |
| Neutrophil count decreased | <lln -="" 1.5="" 1500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <1500 - 1000/mm3; <1.5 - 1.0 x<br>10e9 /L | <1000 - 500/mm3; <1.0 - 0.5 x<br>10e9 /L | <500/mm3; <0.5 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of neutrophils | s in a blood specimen. | | |
| Pancreatic enzymes decreased | <lln and="" asymptomatic<="" td=""><td>Increase in stool frequency, bulk, or odor; steatorrhea</td><td>Sequelae of absorption deficiency</td><td>-</td><td>-</td></lln> | Increase in stool frequency, bulk, or odor; steatorrhea | Sequelae of absorption deficiency | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of pancreatic | enzymes in a biological specimen. | | |

| | | Investigations | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Platelet count decreased | <lln -="" 10e9="" 75,000="" 75.0="" <lln="" l<="" mm3;="" td="" x=""><td>&lt;75,000 - 50,000/mm3; &lt;75.0 - 50.0 x 10e9 /L</td><td>&lt;50,000 - 25,000/mm3; &lt;50.0 - 25.0 x 10e9 /L</td><td>&lt;25,000/mm3; &lt;25.0 x 10e9 /L</td><td>-</td></lln> | <75,000 - 50,000/mm3; <75.0 - 50.0 x 10e9 /L | <50,000 - 25,000/mm3; <50.0 - 25.0 x 10e9 /L | <25,000/mm3; <25.0 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of platelets in | a blood specimen. | | |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate ar | n increase in the levels of amylase | in a serum specimen. | | |
| Urine output decreased | - | - | Oliguria (<80 ml in 8 hr) | Anuria (<240 ml in 24 hr) | - |
| Definition: A finding based on tes | t results that indicate urine produc | tion is less relative to previous ou | tput. | | |
| Vital capacity abnormal | 90 - 75% of predicted value | <75 - 50% of predicted value;<br>limiting instrumental ADL | <50% of predicted value;<br>limiting self care ADL | - | - |
| Definition: A finding based on pu value. | lmonary function test results that ir | ndicate an abnormal vital capacity | (amount of exhaled after a maxim | num inhalation) when compared to | the predicted |
| Weight gain | 5 - <10% from baseline | 10 - <20% from baseline | >=20% from baseline | - | - |
| Definition: A finding characterize | d by an increase in overall body we | eight; for pediatrics, greater than t | he baseline growth curve. | | • |
| Weight loss | 5 to <10% from baseline; intervention not indicated | 10 - <20% from baseline;<br>nutritional support indicated | >=20% from baseline; tube feeding or TPN indicated | - | - |
| Definition: A finding characterize | d by a decrease in overall body we | eight; for pediatrics, less than the b | paseline growth curve. | | |
| White blood cell decreased | <lln -="" 3.0="" 3000="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <3000 - 2000/mm3; <3.0 - 2.0 x<br>10e9 /L | <2000 - 1000/mm3; <2.0 - 1.0 x<br>10e9 /L | <1000/mm3; <1.0 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate ar | n decrease in number of white blo | od cells in a blood specimen. | | |
| Investigations - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Metabolism and nutrition | n disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 | Life-threatening consequences | Death |
| Definition: A disorder characteriz | ted by abnormally high acidity (high | h hydrogen-ion concentration) of t | he blood and other body tissues. | Τ | |
| Alcohol intolerance | - | Present | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz<br>vomiting, indigestion and headac | ted by an increase in sensitivity to thes. | the adverse effects of alcohol, whi | ich can include nasal congestion, s | skin flushes, heart dysrhythmias, r | nausea, |
| Alkalosis | pH >normal, but <=7.5 | - | pH >7.5 | Life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by abnormally high alkalinity (lo | ow hydrogen-ion concentration) of | the blood and other body tissues. | , | 1 |
| Anorexia | Loss of appetite without alteration in eating habits | Oral intake altered without significant weight loss or malnutrition; oral nutritional supplements indicated | Associated with significant weight loss or malnutrition (e.g., inadequate oral caloric and/or fluid intake); tube feeding or TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a loss of appetite. | I | T | T | |
| Dehydration | Increased oral fluids indicated;<br>dry mucous membranes;<br>diminished skin turgor | IV fluids indicated <24 hrs | IV fluids or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by excessive loss of water from | the body. It is usually caused by | severe diarrhea, vomiting or diaph | noresis. | |
| Glucose intolerance | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; dietary<br>modification or oral agent<br>indicated | Severe symptoms; insulin indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an inability to properly metal | bolize glucose. | | | |
| Hypercalcemia | Corrected serum calcium of >ULN - 11.5 mg/dL; >ULN - 2.9 mmol/L; lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 - 13.5 mg/dL; >3.1 - 3.4 mmol/L; lonized calcium >1.6 - 1.8 mmol/L; hospitalization indicated | Corrected serum calcium of >13.5 mg/dL; >3.4 mmol/L; lonized calcium >1.8 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate an elevation in the concen | tration of calcium (corrected for all | oumin) in blood. | |
| Hyperglycemia | Fasting glucose value >ULN -<br>160 mg/dL; Fasting glucose<br>value >ULN - 8.9 mmol/L | Fasting glucose value >160 -<br>250 mg/dL; Fasting glucose<br>value >8.9 - 13.9 mmol/L | >250 - 500 mg/dL; >13.9 - 27.8<br>mmol/L; hospitalization<br>indicated | >500 mg/dL; >27.8 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder characteriz<br>intolerance. | ed by laboratory test results that ir | ndicate an elevation in the concen | tration of blood sugar. It is usually | an indication of diabetes mellitus | or glucose |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L;<br>hospitalization indicated | >7.0 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz the use of diuretic drugs. | ed by laboratory test results that in | ndicate an elevation in the concen | tration of potassium in the blood; a | associated with kidney failure or so | ometimes with |
| Hypermagnesemia | >ULN - 3.0 mg/dL; >ULN - 1.23<br>mmol/L | - | >3.0 - 8.0 mg/dL; >1.23 - 3.30<br>mmol/L | >8.0 mg/dL; >3.30 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate an elevation in the concen | tration of magnesium in the blood | | |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L;<br>hospitalization indicated | >160 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate an elevation in the concen | tration of sodium in the blood. | T | |
| Hypertriglyceridemia | 150 mg/dL - 300 mg/dL; 1.71<br>mmol/L - 3.42 mmol/L | >300 mg/dL - 500 mg/dL; >3.42<br>mmol/L - 5.7 mmol/L | >500 mg/dL - 1000 mg/dL; >5.7<br>mmol/L - 11.4 mmol/L | >1000 mg/dL; >11.4 mmol/L;<br>life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate an elevation in the concen | tration of triglyceride concentration | n in the blood. | |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L)<br>without physiologic<br>consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences | >10 mg/dL; >0.59 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate an elevation in the concen | tration of uric acid. | 1 | 1 |
| Hypoalbuminemia | <lln -="" 3="" 30="" <lln="" dl;="" g="" l<="" td=""><td>&lt;3 - 2 g/dL; &lt;30 - 20 g/L</td><td>&lt;2 g/dL; &lt;20 g/L</td><td>Life-threatening consequences; urgent intervention indicated</td><td>Death</td></lln> | <3 - 2 g/dL; <30 - 20 g/L | <2 g/dL; <20 g/L | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate a low concentration of albu | ımin in the blood. | | |

| | | Metabolism and nutrition | n disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypocalcemia | Corrected serum calcium of<br><lln -="" 2.0<br="" 8.0="" <lln="" dl;="" mg="">mmol/L; lonized calcium <lln -<br="">1.0 mmol/L</lln></lln> | Corrected serum calcium of<br><8.0 - 7.0 mg/dL; <2.0 - 1.75<br>mmol/L; lonized calcium <1.0 -<br>0.9 mmol/L; symptomatic | Corrected serum calcium of<br><7.0 - 6.0 mg/dL; <1.75 - 1.5<br>mmol/L; lonized calcium <0.9 -<br>0.8 mmol/L; hospitalization<br>indicated | Corrected serum calcium of <6.0 mg/dL; <1.5 mmol/L; lonized calcium <0.8 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterization | zed by laboratory test results that ir | ndicate a low concentration of calc | ium (corrected for albumin) in the | blood. | |
| Hypoglycemia | <lln -="" 3.0="" 55="" <lln="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;55 - 40 mg/dL; &lt;3.0 - 2.2<br/>mmol/L</td><td>&lt;40 - 30 mg/dL; &lt;2.2 - 1.7<br/>mmol/L</td><td>&lt;30 mg/dL; &lt;1.7 mmol/L; life-<br/>threatening consequences;<br/>seizures</td><td>Death</td></lln> | <55 - 40 mg/dL; <3.0 - 2.2<br>mmol/L | <40 - 30 mg/dL; <2.2 - 1.7<br>mmol/L | <30 mg/dL; <1.7 mmol/L; life-<br>threatening consequences;<br>seizures | Death |
| Definition: A disorder characterize | red by laboratory test results that in | ndicate a low concentration of gluc | ose in the blood. | | |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" l;<br="" mmol="">symptomatic; intervention<br/>indicated</lln></td><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <lln -="" 3.0="" l;<br="" mmol="">symptomatic; intervention<br/>indicated</lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated | <2.5 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize | zed by laboratory test results that ir | ndicate a low concentration of pota | ssium in the blood. | | |
| Hypomagnesemia | <lln -="" 0.5="" 1.2="" <lln="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL; &lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 - 0.7 mg/dL; &lt;0.4 - 0.3<br/>mmol/L</td><td>&lt;0.7 mg/dL; &lt;0.3 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <1.2 - 0.9 mg/dL; <0.5 - 0.4 mmol/L | <0.9 - 0.7 mg/dL; <0.4 - 0.3<br>mmol/L | <0.7 mg/dL; <0.3 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize | red by laboratory test results that in | ndicate a low concentration of mag | nesium in the blood. | | |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 - 120 mmol/L</td><td>&lt;120 mmol/L; life-threatening consequences</td><td>Death</td></lln> | - | <130 - 120 mmol/L | <120 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize | zed by laboratory test results that ir | ndicate a low concentration of sodi | um in the blood. | | |
| Hypophosphatemia | <lln -="" 0.8="" 2.5="" <lln="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL; &lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 - 1.0 mg/dL; &lt;0.6 - 0.3 mmol/L</td><td>&lt;1.0 mg/dL; &lt;0.3 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <2.5 - 2.0 mg/dL; <0.8 - 0.6 mmol/L | <2.0 - 1.0 mg/dL; <0.6 - 0.3 mmol/L | <1.0 mg/dL; <0.3 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate a low concentration of pho- | sphates in the blood. | | |
| Iron overload | - | Moderate symptoms; intervention not indicated | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by accumulation of iron in the ti | ssues. | | | 1 |
| Obesity | - | BMI 25 - 29.9 kg/m2 | BMI 30 - 39.9 kg/m2 | BMI >=40 kg/m2 | - |
| Definition: A disorder characterization | zed by having a high amount of boo | dy fat. | | 1 | 1 |
| Tumor lysis syndrome | - | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by metabolic abnormalities that | result from a spontaneous or the | apy-related cytolysis of tumor cell | S. | 1 |
| Metabolism and nutrition<br>disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Musculoskeletal and connective tissue disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| bdominal soft tissue necrosis | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other invasive intervention indicated (e.g. tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ।<br>ed by a necrotic process occurrino | | 1 | ı | II. |
| Arthralgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in a joint. | 1 | 1 | |
| Arthritis | Mild pain with inflammation, erythema, or joint swelling | Moderate pain associated with<br>signs of inflammation,<br>erythema, or joint swelling;<br>limiting instrumental ADL | Severe pain associated with<br>signs of inflammation,<br>erythema, or joint swelling;<br>irreversible joint damage;<br>disabling; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by inflammation involving a joir | nt. | | | |
| Avascular necrosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by necrotic changes in the bon<br>d the destruction of the bone struc | • | od supply. Most often affecting the | epiphysis of the long bones, the n | ecrotic |
| Back pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n in the back region. | | | |
| Bone pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n in the bones. | T | 1 | 1 |
| Buttock pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n in the buttocks. | | 1 | |
| Chest wall pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n in the chest wall region. | I | T | |
| Exostosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by non-neoplastic overgrowth | of bone. | | | |
| Fibrosis deep connective tissue | Mild induration, able to move skin parallel to plane (sliding) and perpendicular to skin (pinching up) | Moderate induration, able to slide skin, unable to pinch skin; limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting joint<br>or orifice movement (e.g.<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| | ed by fibrotic degeneration of the | 1 | | | |
| Flank pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n on the lateral side of the body in | the region below the ribs and abo | ove the hip. | |
| Generalized muscle weakness | Symptomatic; weakness perceived by patient but not evident on physical exam | Symptomatic; weakness evident on physical exam; weakness limiting instrumental ADL | Weakness limiting self care<br>ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | of muscles in multiple anatomic sit | es. | • | |
| Growth suppression | Reduction in growth velocity by 10 - 29% ideally measured over the period of a year | Reduction in growth velocity by 30 - 49% ideally measured over the period of a year or 0 - 49% reduction in growth from the baseline growth curve | Reduction in growth velocity of >=50% ideally measured over the period of a year | - | - |
| | ed by of stature that is smaller tha | - | • | • | |

| Musculoskeletal and connective tissue disorders | | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Head soft tissue necrosis | - | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the soft tissues of the head. | | | |
| Joint effusion | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated; disabling | - | - |
| Definition: A disorder characteriz | ed by excessive fluid in a joint, usu | ually as a result of joint inflammation | on. | | |
| Joint range of motion decreased | <=25% loss of ROM (range of<br>motion); decreased ROM<br>limiting athletic activity | >25 - 50% decrease in ROM;<br>limiting instrumental ADL | >50% decrease in ROM; limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a decrease in joint flexibility | of any joint. | | | |
| Joint range of motion decreased<br>cervical spine | Mild restriction of rotation or flexion between 60 - 70 degrees | Rotation <60 degrees to right or left; <60 degrees of flexion | Ankylosed/fused over multiple segments with no C-spine rotation | - | - |
| Definition: A disorder characteriz | ed by a decrease in flexibility of a | cervical spine joint. | T | | |
| Joint range of motion decreased umbar spine | Stiffness; difficulty bending to<br>the floor to pick up a very light<br>object but able to do athletic<br>activity | Pain with range of motion<br>(ROM) in lumbar spine; requires<br>a reaching aid to pick up a very<br>light object from the floor | <50% lumbar spine flexion;<br>associated with symptoms of<br>ankylosis or fused over multiple<br>segments with no L-spine | - | - |
| Dofinition, A dispardor above starin | ad by a degreese in flevibility of a | lumbar anina isint | flexion (e.g., unable to reach to<br>floor to pick up a very light<br>object) | | |
| | ed by a decrease in flexibility of a | Moderate accentuation; limiting | Source accontraction: anarotive | | |
| Kyphosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | instrumental ADL | Severe accentuation; operative intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by an abnormal increase in the | curvature of the thoracic portion of | of the spine. | T | |
| Lordosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate accentuation; limiting instrumental ADL | Severe accentuation; operative intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by an abnormal increase in the | curvature of the lumbar portion of | the spine. | | |
| Muscle weakness left-sided | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | '<br>If the muscles on the left side of th | e body. | ' | ' |
| Muscle weakness lower limb | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the lower limb muscles. | <b>.</b> | 1 | |
| Muscle weakness right-sided | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the muscles on the right side of t | the body. | <b>.</b> | |
| Muscle weakness trunk | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the trunk muscles. | | : | • |
| Muscle weakness upper limb | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |

| Musculoskeletal and connective tissue disorders Grade | | | | | |
|---|---|---|---|---|---|
| A.L | 4 | | Grade | | _ |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Musculoskeletal deformity | Cosmetically and functionally insignificant hypoplasia | Deformity, hypoplasia, or<br>asymmetry able to be<br>remediated by prosthesis (e.g., | Significant deformity,<br>hypoplasia, or asymmetry,<br>unable to be remediated by | - | - |
| | | shoe insert) or covered by clothing | prosthesis or covered by clothing; disabling | | |
| Definition: A disorder characteriz | zed by of a malformation of the mu | sculoskeletal system. | | | |
| Myalgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | zed by marked discomfort sensatio | n originating from a muscle or gro | up of muscles. | | |
| Myositis | Mild pain | Moderate pain associated with weakness; pain limiting instrumental ADL | Pain associated with severe weakness; limiting self care ADL | - | - |
| Definition: A disorder characteris | ।<br>zed by inflammation involving the s | 1 | /\DE | | l |
| Neck pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care | - | - |
| Definition: A disorder characteriz | zed by marked discomfort sensatio | n in the neck area. | ! | I | ı |
| Neck soft tissue necrosis | - | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteris | ା<br>zed by a necrotic process occurrinç | 1 | or graning) | | l |
| | | | Sovere symptoms: limiting self | Life threatening consequences: | Death |
| Osteonecrosis of jaw | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Deam |
| Definition: A disorder characteriz | zed by a necrotic process occurring | in the bone of the mandible. | | | |
| Osteoporosis | Radiologic evidence of osteoporosis or Bone Mineral Density (BMD) t-score -1 to -2.5 (osteopenia); no loss of height or intervention indicated | BMD t-score <-2.5; loss of<br>height <2 cm; anti-osteoporotic<br>therapy indicated; limiting<br>instrumental ADL | Loss of height >=2 cm;<br>hospitalization indicated; limiting<br>self care ADL | - | - |
| Definition: A disorder characterize composition), resulting in increase | zed by reduced bone mass, with a | decrease in cortical thickness and | in the number and size of the trab | eculae of cancellous bone (but no | rmal chemi |
| Pain in extremity | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by marked discomfort sensatio | n in the upper or lower extremities | i. | | |
| Pelvic soft tissue necrosis | - | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by a necrotic process occurring | in the soft tissues of the pelvis. | | | |
| Scoliosis | <20 degrees; clinically undetectable | >20 - 45 degrees; visible by<br>forward flexion; limiting<br>instrumental ADL | >45 degrees; scapular<br>prominence in forward flexion;<br>operative intervention indicated;<br>limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ा<br>zed by a malformed, lateral curvatu | re of the spine. | ,9 | 1 | T. |
| Soft tissue necrosis lower limb | - | Local wound care; medical intervention indicated (e.g., dressings or topical | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap | Life-threatening consequences; urgent intervention indicated | Death |
| | | medications) | or grafting) | | |
| | zed by a necrotic process occurring | | 1 | | |
| Soft tissue necrosis upper limb | - | Local wound care; medical intervention indicated (e.g., | Operative debridement or other invasive intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | | dressings or topical medications) | (e.g., tissue reconstruction, flap or grafting) | | |

| | Musculoskeletal and connective tissue disorders | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Superficial soft tissue fibrosis | Mild induration, able to move | Moderate induration, able to | Severe induration; unable to | Generalized; associated with | Death |
| | skin parallel to plane (sliding) | slide skin, unable to pinch skin; | slide or pinch skin; limiting joint | signs or symptoms of impaired | |
| | and perpendicular to skin | limiting instrumental ADL | or orifice movement (e.g., | breathing or feeding | |
| | (pinching up) | | mouth, anus); limiting self care | | |
| | | | ADL | | |
| Definition: A disorder characteriz | ed by fibrotic degeneration of the | superficial soft tissues. | | | |
| Trismus | Decreased ROM (range of | Decreased ROM requiring small | Decreased ROM with inability to | - | - |
| | motion) without impaired eating | bites, soft foods or purees | adequately aliment or hydrate | | |
| | | | orally | | |
| Definition: A disorder characteriz | ed by lack of ability to open the mo | outh fully due to a decrease in the | range of motion of the muscles of | mastication. | |
| Unequal limb length | Mild length discrepancy <2 cm | Moderate length discrepancy 2 - | Severe length discrepancy >5 | - | - |
| | | 5 cm; shoe lift indicated; limiting | cm; limiting self care ADL; | | |
| | | instrumental ADL | disabling; operative intervention | | |
| | | | indicated | | |
| Definition: A disorder characteriz | ed by of a discrepancy between th | e lengths of the lower or upper ex | tremities. | | |
| Musculoskeletal and connective | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| tissue disorder - Other, specify | symptoms; clinical or diagnostic | noninvasive intervention | but not immediately life- | urgent intervention indicated | |
| | observations only; intervention | indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| | | | disabling; limiting self care ADL | | |

| | Neopiasms benig | n, maiignant and unspe | cified (incl cysts and poly | /ps) | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| _eukemia secondary to<br>oncology chemotherapy | - | - | - | Present | Death |
| Definition: A disorder characteriz | ed by leukemia arising as a result | of the mutagenic effect of chemo | therapy agents. | | |
| Myelodysplastic syndrome | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by insufficiently healthy hemata | apoietic cell production by the bon | e marrow. | | |
| Treatment related secondary | - | - | Non life-threatening secondary | Acute life-threatening secondary | Death |
| malignancy | | | malignancy | malignancy; blast crisis in leukemia | |
| Definition: A disorder characteriz | ed by development of a malignand | cy most probably as a result of tre | atment for a previously existing ma | alignancy. | |
| Tumor pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort from a ne | eoplasm that may be pressing on | a nerve, blocking blood vessels, ir | flamed or fractured from metastas | is. |
| Neoplasms benign, malignant and unspecified (incl cysts and | Asymptomatic or mild symptoms; clinical or diagnostic | Moderate; minimal, local or noninvasive intervention | Severe or medically significant but not immediately life- | Life-threatening consequences; urgent intervention indicated | Death |
| polyps) - Other, specify | observations only; intervention not indicated | indicated; limiting age-<br>appropriate instrumental ADL | threatening; hospitalization or prolongation of existing hospitalization indicated; | | |
| | | | disabling; limiting self care ADL | | |

| Nervous system disorders | | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abducens nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by involvement of the abducen | s nerve (sixth cranial nerve). | | | |
| Accessory nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by involvement of the accessor | y nerve (eleventh cranial nerve). | _ | | |
| Acoustic nerve disorder NOS | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by involvement of the acoustic | nerve (eighth cranial nerve). | T | | |
| kathisia | Mild restlessness or increased motor activity | Moderate restlessness or increased motor activity; limiting instrumental ADL | Severe restlessness or increased motor activity; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by an uncomfortable feeling of | inner restlessness and inability to | stay still; this is a side effect of so | me psychotropic drugs. | |
| Amnesia | Mild; transient memory loss | Moderate; short term memory loss; limiting instrumental ADL | Severe; long term memory loss; limiting self care ADL | - | - |
| | zed by systematic and extensive lo | ss of memory. | V-il | | |
| Aphonia | - | - | Voicelessness; unable to speak | - | - |
| Definition: A disorder characteri<br>Arachnoiditis | zed by the inability to speak. It may Mild symptoms | Moderate symptoms; limiting | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| | | instrumental ADL | care ADL | urgent intervention indicated | 1 |
| | zed by inflammation of the arachno | | 1 | | |
| Ataxia | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; mechanical assistance indicated | - | - |
| Definition: A disorder characteri | zed by lack of coordination of musc | ·<br>le movements resulting in the imp | ·<br>airment or inability to perform volu | ntary activities. | • |
| Brachial plexopathy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by regional paresthesia of the l | rachial plexus, marked discomfor | t and muscle weakness, and limite | ed movement in the arm or hand. | |
| Central nervous system<br>necrosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms;<br>corticosteroids indicated | Severe symptoms; medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | in the brain and/or spinal cord. | Т | Т | |
| Cerebrospinal fluid leakage | Post-craniotomy: asymptomatic;<br>Post-lumbar puncture: transient<br>headache; postural care<br>indicated | Post-craniotomy: moderate<br>symptoms; medical intervention<br>indicated; Post-lumbar<br>puncture: persistent moderate<br>symptoms; blood patch<br>indicated | Severe symptoms; medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by loss of cerebrospinal fluid in | to the surrounding tissues. | | | |
| Cognitive disturbance | Mild cognitive disability; not interfering with work/school/life performance; specialized educational services/devices not indicated | Moderate cognitive disability;<br>interfering with work/school/life<br>performance but capable of<br>independent living; specialized<br>resources on part time basis<br>indicated | Severe cognitive disability;<br>significant impairment of<br>work/school/life performance | - | - |
| Definition: A disorder characteri | zed by a conspicuous change in co | gnitive function. | | • | • |
| Concentration impairment | Mild inattention or decreased level of concentration | Moderate impairment in attention or decreased level of concentration; limiting instrumental ADL | Severe impairment in attention<br>or decreased level of<br>concentration; limiting self care<br>ADL | - | - |
| | 1 | I . | 1 | I | 1 |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Depressed level of consciousness | Decreased level of alertness | Sedation; slow response to stimuli; limiting instrumental ADL | Difficult to arouse | Life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by a decrease in ability to perce | eive and respond. | T | T | |
| Dizziness | Mild unsteadiness or sensation of movement | Moderate unsteadiness or sensation of movement; limiting instrumental ADL | Severe unsteadiness or sensation of movement; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a disturbing sensation of ligh | ntheadedness, unsteadiness, gidd | liness, spinning or rocking. | • | , |
| Dysarthria | Mild slurred speech | Moderate impairment of articulation or slurred speech | Severe impairment of articulation or slurred speech | - | - |
| Definition: A disorder characteriz | ed by slow and slurred speech res | ulting from an inability to coordina | te the muscles used in speech. | T | |
| Dysesthesia | Mild sensory alteration | Moderate sensory alteration;<br>limiting instrumental ADL | Severe sensory alteration;<br>limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by distortion of sensory percep | | 1 | <u> </u> | |
| Dysgeusia | Altered taste but no change in diet | Altered taste with change in diet (e.g., oral supplements); noxious or unpleasant taste; loss of taste | - | - | - |
| Definition: A disorder characteriz | ed by abnormal sensual experienc | e with the taste of foodstuffs; it ca | n be related to a decrease in the | sense of smell. | |
| Dysphasia | Awareness of receptive or expressive characteristics; not impairing ability to communicate | Moderate receptive or expressive characteristics; impairing ability to communicate spontaneously | Severe receptive or expressive characteristics; impairing ability to read, write or communicate intelligibly | - | - |
| Definition: A disorder characteriz | ed by impairment of verbal commu | unication skills, often resulting from | n brain damage. | T | |
| Edema cerebral | - | - | - | Life-threatening consequences; urgent intervention indicated | - |
| | ed by swelling due to an excessive | | | | |
| Encephalopathy | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a pathologic process involvi | | <u> </u> | I | I |
| Extrapyramidal disorder | Mild involuntary movements | Moderate involuntary movements; limiting instrumental ADL | Severe involuntary movements or torticollis; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by abnormal, repetitive, involur | tary muscle movements, frenzied | speech and extreme restlessness | <b>5.</b> | |
| Facial muscle weakness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the facial muscles. | | | |
| Facial nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by involvement of the facial ner | rve (seventh cranial nerve). | 1 | <b>.</b> | 1 |
| Glossopharyngeal nerve<br>disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by involvement of the glossoph | aryngeal nerve (ninth cranial nerv | e). | <b>.</b> | 1 |
| Headache | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | mfort in various parts of the head, | , not confined to the area of distrib | ution of any nerve. | |
| Hydrocephalus | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms;<br>intervention not indicated | Severe symptoms or neurological deficit; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal increase of cer | rebrospinal fluid in the ventricles o | f the brain. | <b>.</b> | |
| Hypersomnia | Mild increased need for sleep | Moderate increased need for sleep | Severe increased need for sleep | - | - |
| Definition: A disorder characteriz | ed by characterized by excessive | sleepiness during the daytime. | | | |

| Nervous system disorders | | | | | |
|---|---|---|---|---|---|
| | | T | Grade | T | 1 |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypoglossal nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder character | ized by involvement of the hypoglos | sal nerve (twelfth cranial nerve). | | | |
| Intracranial hemorrhage | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Ventriculostomy, ICP<br>monitoring, intraventricular<br>thrombolysis, or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by bleeding from the cranium. | | | | |
| schemia cerebrovascular | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms | - | - | - |
| Definition: A disorder character<br>damage. | ized by a decrease or absence of bl | ood supply to the brain caused by | obstruction (thrombosis or embol | ism) of an artery resulting in neuro | logical |
| Vth nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| | ized by involvement of the trochlear | T , | | | |
| ethargy | Mild symptoms; reduced alertness and awareness | Moderate symptoms; limiting instrumental ADL | - | - | - |
| Definition: A disorder character | ized by a decrease in consciousnes | s characterized by mental and phy | ysical inertness. | 1 | 1 |
| Leukoencephalopathy | Asymptomatic; small focal T2/FLAIR hyperintensities; involving periventricular white matter or <1/3 of susceptible areas of cerebrum +/- mild increase in subarachnoid space (SAS) and/or mild ventriculomegaly | Moderate symptoms; focal T2/FLAIR hyperintensities, involving periventricular white matter extending into centrum semiovale or involving 1/3 to 2/3 of susceptible areas of cerebrum +/- moderate increase in SAS and/or moderate ventriculomegaly | Severe symptoms; extensive T2/FLAIR hyperintensities, involving periventricular white matter involving 2/3 or more of susceptible areas of cerebrum +/- moderate to severe increase in SAS and/or moderate to severe ventriculomegaly | Life-threatening consequences; extensive T2/FLAIR hyperintensities, involving periventricular white matter involving most of susceptible areas of cerebrum +/- moderate to severe increase in SAS and/or moderate to severe ventriculomegaly | Death |
| Definition: A disorder character | ized by diffuse reactive astrocytosis | | ।<br>:i without inflammation | , , | 1 |
| Memory impairment | Mild memory impairment | Moderate memory impairment; | Severe memory impairment; limiting self care ADL | - | - |
| Definition: A disorder character | ized by a deterioration in memory fu | - | | 1 | I |
| Meningismus | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ।<br>ized by neck stiffness, headache, ai | ı | 1 | angone miles remain maneacea | l |
| Movements involuntary | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder character | ized by uncontrolled and purposeles | ss movements. | 1 | ı | 1 |
| Myelitis | Asymptomatic; mild signs (e.g., Babinski's reflex or Lhermitte's sign) | Moderate weakness or sensory loss; limiting instrumental ADL | Severe weakness or sensory loss; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | ized by inflammation involving the s | 1 | 1 | marked discomfort and incontiner | ice. |
| Neuralgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | ized by intense painful sensation ald | ong a nerve or group of nerves. | T | 1 | |
| Nystagmus | - | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder character | ized by involuntary movements of th | ne eyeballs. | T | | |
| Oculomotor nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder character | ized by involvement of the oculomo | tor nerve (third cranial nerve). | T | ı | |
| Olfactory nerve disorder | - | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder character | ized by involvement of the olfactory | nerve (first cranial nerve). | | | |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Paresthesia | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz are experienced in the absence of | | ensory neurons resulting in abnorr | mal cutaneous sensations of tingli | ng, numbness, pressure, cold, and | warmth that |
| Peripheral motor neuropathy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; assistive device indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz Peripheral sensory neuropathy | ed by inflammation or degeneration Asymptomatic; loss of deep tendon reflexes or paresthesia | n of the peripheral motor nerves. Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation or degeneratio | n of the peripheral sensory nerves | S. | T | |
| Phantom pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort related to | o a limb or an organ that is remove | ed from or is not physically part of | the body. | |
| Presyncope | - | Present (e.g., near fainting) | - | - | - |
| Definition: A disorder characteriz | ed by an episode of lightheadedne | ess and dizziness which may prec | ede an episode of syncope. | <b>.</b> | |
| Pyramidal tract syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by dysfunction of the corticospi<br>and a decrease in fine motor coord | | l cord. Symptoms include an incre | ease in the muscle tone in the lowe | er extremities, |
| Radiculitis | Mild symptoms | Moderate symptoms; limiting instrumental ADL; medical intervention indicated | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz connecting nerve root. | ed by inflammation involving a ner | ve root. Patients experience mark | ed discomfort radiating along a ne | rve path because of spinal pressu | re on the |
| Recurrent laryngeal nerve palsy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord injection) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by paralysis of the recurrent lar | yngeal nerve. | | | |
| Reversible posterior leukoencephalopathy syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; abnormal imaging studies; limiting instrumental ADL | Severe symptoms; very<br>abnormal imaging studies;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | | = | | indings of posterior leukoencephal<br>s an acute or subacute reversible o | · · |
| Seizure | Brief partial seizure; no loss of consciousness | Brief generalized seizure | Multiple seizures despite medical intervention | Life-threatening; prolonged repetitive seizures | Death |
| Definition: A disorder characteriz | ed by a sudden, involuntary skelet | al muscular contractions of cerebi | ral or brain stem origin. | T | |
| Sinus pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort in the fac | ce, between the eyes, or upper tee | eth originating from the sinuses. | I | |
| Somnolence | Mild but more than usual drowsiness or sleepiness | Moderate sedation; limiting instrumental ADL | Obtundation or stupor | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by characterized by excessive | sleepiness and drowsiness. | T | T | |
| Spasticity | Mild or slight increase in muscle tone | Moderate increase in muscle<br>tone and increase in resistance<br>through range of motion | Severe increase in muscle tone and increase in resistance through range of motion | Life-threatening; unable to move active or passive range of motion | Death |
| Definition: A disorder characteriz disturbances. | ed by increased involuntary muscl | | 1 | ।<br>It results in gait, movement, and s <sub>l</sub> | peech |
| Stroke | Asymptomatic or mild neurologic deficit; radiographic findings only | Moderate neurologic deficit | Severe neurologic deficit | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a sudden loss of sensory fu | nction due to an intracranial vascu | ılar event. | | |
| Syncope | - | - | Fainting; orthostatic collapse | - | - |
| Definition: A disorder characteriz | ed by spontaneous loss of conscio | ousness caused by insufficient blo | od supply to the brain. | | |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Transient ischemic attacks | Mild neurologic deficit with or without imaging confirmation | Moderate neurologic deficit with or without imaging confirmation | - | - | - |
| Definition: A disorder character | zed by a brief attack (less than 24 h | nours) of cerebral dysfunction of v | ascular origin, with no persistent n | eurological deficit. | |
| Tremor | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder character | zed by the uncontrolled shaking mo | vement of the whole body or indiv | vidual parts. | T | |
| Trigeminal nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder character | zed by involvement of the trigemina | l nerve (fifth cranial nerve). | | | |
| Vagus nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | zed by involvement of the vagus ne | rve (tenth cranial nerve). | • | • | |
| Vasovagal reaction | - | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character increase in the stimulation of th | zed by a sudden drop of the blood per vagus nerve. | oressure, bradycardia, and periph | eral vasodilation that may lead to l | oss of consciousness. It results fro | om an |
| Nervous system disorders - | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| Other, specify | symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | noninvasive intervention indicated; limiting age-appropriate instrumental ADL | but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | urgent intervention indicated | |
| | | | disabling; limiting self care ADL | | |

| | Pregna | ancy, puerperium and pe | rinatal conditions | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Fetal death | - | - | - | - | Fetal loss at<br>any<br>gestational<br>age |
| | ed by death in utero; failure of the | product of conception to show ev | idence of respiration, heartbeat, or | definite movement of a voluntary | muscle after |
| expulsion from the uterus, withou | it possibility of resuscitation. | | 1 | 1 | |
| Fetal growth retardation | - | <10% percentile of weight for gestational age | <5% percentile of weight for gestational age | <1% percentile of weight for gestational age | - |
| Definition: A disorder characteriz | ed by inhibition of fetal growth res | ulting in the inability of the fetus to | achieve its potential weight. | | |
| Premature delivery | Delivery of a liveborn infant at >34 to 37 weeks gestation | Delivery of a liveborn infant at >28 to 34 weeks gestation | Delivery of a liveborn infant at 24 to 28 weeks gestation | Delivery of a liveborn infant at 24 weeks of gestation or less | - |
| Definition: A disorder characteriz gestation. | ed by delivery of a viable infant be | fore the normal end of gestation. | Typically, viability is achievable be | tween the twentieth and thirty-sev | enth week of |
| Unintended pregnancy | - | - | Unintended pregnancy | - | - |
| Definition: A disorder characteriz | ed by an unexpected pregnancy a | t the time of conception. | | • | |
| Pregnancy, puerperium and perinatal conditions - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate, local or noninvasive intervention indicated; limiting instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Psychiatric disor | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Agitation | Mild mood alteration | Moderate mood alteration | not indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by a state of restlessness asso | 1 | irritability and tension. | | |
| Anorgasmia | Inability to achieve orgasm not adversely affecting relationship | Inability to achieve orgasm adversely affecting relationship | - | - | - |
| Definition: A disorder characte | erized by an inability to achieve orgas | m. | T | Т | 1 |
| Anxiety | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization not indicated | Life-threatening; hospitalization indicated | Death |
| Definition: A disorder characte<br>stimulus. | erized by apprehension of danger and | d dread accompanied by restlessn | ess, tension, tachycardia, and dys | pnea unattached to a clearly ident | ifiable |
| Confusion | Mild disorientation | Moderate disorientation; limiting instrumental ADL | Severe disorientation; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by a lack of clear and orderly t | nought and behavior. | | | |
| Delayed orgasm | Delay in achieving orgasm not adversely affecting relationship | Delay in achieving orgasm adversely affecting relationship | - | - | - |
| Definition: A disorder characte | erized by sexual dysfunction characte | rized by a delay in climax. | 1 | | 1 |
| Delirium | Mild acute confusional state | Moderate and acute confusional state; limiting instrumental ADL | Severe and acute confusional state; limiting self care ADL; hospitalization indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder character<br>reversible condition. | erized by the acute and sudden devel | opment of confusion, illusions, mo | ovement changes, inattentiveness, | agitation, and hallucinations. Usu | ally, it is a |
| Delusions | - | Moderate delusional symptoms | Severe delusional symptoms;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by false personal beliefs held o | ontrary to reality, despite contradi | ctory evidence and common sense | ·<br>∋. | |
| Depression | Mild depressive symptoms | Moderate depressive symptoms; limiting instrumental ADL | Severe depressive symptoms;<br>limiting self care ADL;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by melancholic feelings of grie | or unhappiness. | | | |
| Euphoria | Mild mood elevation | Moderate mood elevation | Severe mood elevation (e.g., hypomania) | - | - |
| Definition: A disorder characte | erized by an exaggerated feeling of w | ell-being which is disproportionate | e to events and stimuli. | | |
| Hallucinations | Mild hallucinations (e.g., perceptual distortions) | Moderate hallucinations | Severe hallucinations;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by a false sensory perception i | n the absence of an external stimu | ılus. | | |
| Insomnia | Mild difficulty falling asleep,<br>staying asleep or waking up<br>early | Moderate difficulty falling asleep, staying asleep or waking up early | Severe difficulty in falling asleep, staying asleep or waking up early | - | - |
| Definition: A disorder characte | erized by difficulty in falling asleep an | d/or remaining asleep. | | | |
| Libido decreased | Decrease in sexual interest not adversely affecting relationship | Decrease in sexual interest adversely affecting relationship | - | - | - |
| Definition: A disorder characte | erized by a decrease in sexual desire | | | | |
| Libido increased | Mild increase in sexual interest<br>not adversely affecting<br>relationship | Moderate increase in sexual interest adversely affecting relationship | Severe increase in sexual interest leading to dangerous behavior | - | - |
| Definition: A disorder characte | erized by an increase in sexual desire | ). | | | |
| Mania | Mild manic symptoms (e.g., elevated mood, rapid thoughts, rapid speech, decreased need for sleep) | Moderate manic symptoms<br>(e.g., relationship and work<br>difficulties; poor hygiene) | Severe manic symptoms (e.g., hypomania; major sexual or financial indiscretions); hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by excitement of psychotic pro | portions manifested by mental and | physical hyperactivity, disorganiz | ation of behavior and elevation of | mood. |
| Personality change | Mild personality change | Moderate personality change | Severe personality change;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| | | Psychiatric disord | ders | | | | | |
|---|---|---|---|---|---|--|--|--|
| | Grade | | | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 | | | |
| Definition: A disorder characteriz | ed by a conspicuous change in a ր | person's behavior and thinking. | | | | | | |
| Psychosis | Mild psychotic symptoms | Moderate psychotic symptoms<br>(e.g., disorganized speech;<br>impaired reality testing) | Severe psychotic symptoms<br>(e.g., paranoid; extreme<br>disorganization); hospitalization<br>not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death | | | |
| Definition: A disorder characteriz tumor. | ed by personality change, impaired | d functioning, and loss of touch wi | th reality. It may be a manifestatio | n of schizophrenia, bipolar disorde | er or brain | | | |
| Restlessness | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - | | | |
| Definition: A disorder characteriz | ed by an inability to rest, relax or b | pe still. | | | | | | |
| Suicidal ideation | Increased thoughts of death but no wish to kill oneself | Suicidal ideation with no specific plan or intent | Specific plan to commit suicide<br>without serious intent to die<br>which may not require<br>hospitalization | Specific plan to commit suicide with serious intent to die which requires hospitalization | - | | | |
| Definition: A disorder characteriz | ed by thoughts of taking one's owr | n life. | | | | | | |
| Suicide attempt | - | - | Suicide attempt or gesture without intent to die which may not require hospitalization | Suicide attempt with intent to die which requires hospitalization | Death | | | |
| Definition: A disorder characteriz | ed by self-inflicted harm in an atte | mpt to end one's own life. | | | | | | |
| Psychiatric disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; disabling; limiting<br>self care ADL | Life-threatening consequences;<br>hospitalization or urgent<br>intervention indicated | Death | | | |

| mg/dL; creabove bas Definition: A disorder characterized by the acauses (ureteral or bladder outflow obstruction and the perforation are perforation and the perforation are perforation and the perforation are perforation and the perforation are perforation. A disorder characterized by a sudden to the perforation are perforation and the perforation and the perforation and the perforation and the perforation and the perforation are perforation and the perforation | cute loss of renal function). Inture in the bladder wall on not indicated dden and involuntary continuated Glomerular Rate) or CrCl eclearance) <lln -="" 60="" 73="" ecatinine="" m2="" or="" proteinuriant;="" urine="">0.5 cual and usually permanuloic hematuria; minimal in frequency, urgency, rinocturia; new onset</lln> | Extraperitoneal perforation, indwelling catheter indicated Antispasmodics indicated ontraction of the bladder wall. eGFR or CrCl 59 - 30 ml/min/1.73 m2 eent loss of kidney function resultii Moderate hematuria; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental | Intraperitoneal perforation; elective radiologic, endoscopic or operative intervention indicated Hospitalization indicated eGFR or CrCl 29 - 15 ml/min/1.73 m2 | dialysis indicated Iney), renal (kidney damage) and public threatening consequences; organ failure; urgent operative intervention indicated | Death Death Death Death |
|---|---|---|---|---|---|
| Acute kidney injury Creatinine mg/dL; creation above bas Definition: A disorder characterized by the acauses (ureteral or bladder outflow obstruction and the perforation are perforation and the perforation are perforation and the perforation are perforation and the perforation are perforation. A disorder characterized by a rup Definition: A disorder characterized by a sudden perforation and perforation are perforation and perforation and perforation and perforation are perforationally as a perforation and perforation an | e level increase of >0.3 eatinine 1.5 - 2.0 x seline cute loss of renal funct ion). eture in the bladder wall on not indicated dden and involuntary co timated Glomerular Rate) or CrCl e clearance) <lln -="" 60="" 73="" eatinine="" m2="" or="" proteinuria="" t;="" urine="">0.5 ual and usually perman oic hematuria; minimal in frequency, urgency, r nocturia; new onset</lln> | Creatinine 2 - 3 x above baseline ion and is traditionally classified a Extraperitoneal perforation, indwelling catheter indicated Antispasmodics indicated ontraction of the bladder wall. eGFR or CrCl 59 - 30 ml/min/1.73 m2 ment loss of kidney function resulting the maturia; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental | Creatinine >3 x baseline or >4.0 mg/dL; hospitalization indicated as pre-renal (low blood flow into kid as pre-renal (low blood flow indicated) Hospitalization indicated eGFR or CrCl 29 - 15 ml/min/1.73 m2 Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative | Life-threatening consequences; dialysis indicated Iney), renal (kidney damage) and public threatening consequences; organ failure; urgent operative intervention indicated - eGFR or CrCl <15 ml/min/1.73 m2; dialysis or renal transplant indicated Life-threatening consequences; urgent radiologic or operative | Death Death - Death |
| mg/dL; creabove base Definition: A disorder characterized by the actauses (ureteral or bladder outflow obstructions) Definition: A disorder characterized by a rup Bladder spasm Intervention Definition: A disorder characterized by a sudder spasm Intervention (creatinine ml/min/1.7 2+ presen protein/creatinine ml/min/composition (creatinine ml/min/composition) Definition: A disorder characterized by gradual displaying of inconting ml/min/composition (creatinine ml/min/composition) Definition: A disorder characterized by gradual displaying of inconting displaying of inconting displaying of inconting displaying displaying output displaying displaying output displaying displaying output displaying displayin | eatinine 1.5 - 2.0 x seline cute loss of renal funct ion). Seline cute loss of renal funct ion). Seline cuter in the bladder wall cuter in the bla | Extraperitoneal perforation, indwelling catheter indicated Antispasmodics indicated ontraction of the bladder wall. eGFR or CrCl 59 - 30 ml/min/1.73 m2 eent loss of kidney function resultii Moderate hematuria; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental | mg/dL; hospitalization indicated as pre-renal (low blood flow into kid as pre-renal (low blood flow into kid as pre-renal (low blood flow into kid as pre-renal (low blood flow into kid lintraperitoneal perforation; elective radiologic, endoscopic or operative intervention indicated Hospitalization indicated eGFR or CrCl 29 - 15 ml/min/1.73 m2 Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative | dialysis indicated Iney), renal (kidney damage) and public threatening consequences; organ failure; urgent operative intervention indicated | Death Death |
| Definition: A disorder characterized by a rup Bladder spasm Intervention Definition: A disorder characterized by a sud Chronic kidney disease eGFR (est Filtration Filtration Filtration: A disorder characterized by gradue Definition: A disorder characterized by gradue Definition: A disorder characterized by gradue Definition: A disorder characterized by gradue Definition: A disorder characterized by gradue Definition: A disorder characterized by increase in dysuria, or of incontinuate displays a display of the displays and displays the displays and displays the displays and displays the displays and displays the displays t | on). Sture in the bladder wall on not indicated dden and involuntary continuated Glomerular (Rate) or CrCl (Ra | Extraperitoneal perforation, indwelling catheter indicated Antispasmodics indicated ontraction of the bladder wall. eGFR or CrCl 59 - 30 ml/min/1.73 m2 ment loss of kidney function resulting the maturia; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental | Intraperitoneal perforation; elective radiologic, endoscopic or operative intervention indicated Hospitalization indicated eGFR or CrCl 29 - 15 ml/min/1.73 m2 Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative | Life-threatening consequences; organ failure; urgent operative intervention indicated - eGFR or CrCl <15 ml/min/1.73 m2; dialysis or renal transplant indicated Life-threatening consequences; urgent radiologic or operative | Death - Death |
| Definition: A disorder characterized by a rup Bladder spasm Intervention Definition: A disorder characterized by a sud Chronic kidney disease eGFR (est Filtration F (creatinine ml/min/1.7 2+ presen protein/cre Definition: A disorder characterized by gradu Cystitis noninfective Microscop increase in dysuria, or of incontin Definition: A disorder characterized by inflan Hematuria Asymptom diagnostic intervention | on not indicated dden and involuntary co timated Glomerular Rate) or CrCl e clearance) <lln -="" 60="" 73="" eatinine="" m2="" or="" proteinuria="" t;="" urine="">0.5 ual and usually perman oic hematuria; minimal n frequency, urgency, r nocturia; new onset</lln> | Antispasmodics indicated Antispasmodics indicated Ontraction of the bladder wall. eGFR or CrCl 59 - 30 ml/min/1.73 m2 Hent loss of kidney function resulting Moderate hematuria; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental | elective radiologic, endoscopic or operative intervention indicated Hospitalization indicated eGFR or CrCl 29 - 15 ml/min/1.73 m2 Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative | organ failure; urgent operative intervention indicated - eGFR or CrCl <15 ml/min/1.73 m2; dialysis or renal transplant indicated Life-threatening consequences; urgent radiologic or operative | - Death |
| Bladder spasm Definition: A disorder characterized by a sud Chronic kidney disease Chronic kidney disease GFR (est Filtration F (creatinine ml/min/1.7 2+ presen protein/cre Definition: A disorder characterized by gradu Cystitis noninfective Microscop increase in dysuria, or of incontin Definition: A disorder characterized by inflan Hematuria Asymptom diagnostic intervention | on not indicated dden and involuntary co timated Glomerular Rate) or CrCl e clearance) <lln -="" 60="" 73="" eatinine="" m2="" or="" proteinuria="" t;="" urine="">0.5 ual and usually perman oic hematuria; minimal n frequency, urgency, r nocturia; new onset</lln> | Antispasmodics indicated ontraction of the bladder wall. eGFR or CrCl 59 - 30 ml/min/1.73 m2 ent loss of kidney function resulting the maturia; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental | eGFR or CrCl 29 - 15 ml/min/1.73 m2 ng in renal failure. Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative | eGFR or CrCl <15 ml/min/1.73 m2; dialysis or renal transplant indicated Life-threatening consequences; urgent radiologic or operative | |
| Definition: A disorder characterized by a sud- Chronic kidney disease eGFR (est Filtration F (creatinine ml/min/1.7 2+ presen protein/cre Definition: A disorder characterized by gradu Cystitis noninfective Microscop increase ir dysuria, or of incontin Definition: A disorder characterized by inflan Hematuria Asymptom diagnostic interventio | dden and involuntary continuated Glomerular Rate) or CrCl e clearance) <lln -="" 60="" 73="" eatinine="" m2="" or="" proteinuria="" tt;="" urine="">0.5 ual and usually perman pic hematuria; minimal in frequency, urgency, r nocturia; new onset</lln> | eGFR or CrCl 59 - 30 ml/min/1.73 m2 ent loss of kidney function resulting the maturia; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental | eGFR or CrCl 29 - 15 ml/min/1.73 m2 ng in renal failure. Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative | eGFR or CrCl <15 ml/min/1.73 m2; dialysis or renal transplant indicated Life-threatening consequences; urgent radiologic or operative | |
| Chronic kidney disease eGFR (est Filtration F (creatinine ml/min/1.7 2+ presen protein/cre Definition: A disorder characterized by gradu dysuria, or of incontin Definition: A disorder characterized by inflantematuria Asymptom diagnostic intervention | timated Glomerular Rate) or CrCl e clearance) <lln -="" 60="" 73="" eatinine="" m2="" or="" proteinuria="" t;="" urine="">0.5 ual and usually perman oic hematuria; minimal n frequency, urgency, r nocturia; new onset</lln> | eGFR or CrCl 59 - 30 ml/min/1.73 m2 ent loss of kidney function resulting the state of kidney function resulting the state of kidney function resulting the state of kidney function resulting the state of kidney function in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental | ml/min/1.73 m2 ng in renal failure. Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative | m2; dialysis or renal transplant indicated Life-threatening consequences; urgent radiologic or operative | |
| Filtration F (creatinine ml/min/1.7 2+ presen protein/cre Definition: A disorder characterized by gradu Cystitis noninfective Microscop increase in dysuria, or of incontin Definition: A disorder characterized by inflantematuria Asymptom diagnostic intervention | Rate) or CrCl e clearance) <lln -="" 60="" 73="" eatinine="" m2="" or="" proteinuria="" t;="" urine="">0.5 ual and usually perman oic hematuria; minimal n frequency, urgency, r nocturia; new onset</lln> | ml/min/1.73 m2 ment loss of kidney function resulting the maturia; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental | ml/min/1.73 m2 ng in renal failure. Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative | m2; dialysis or renal transplant indicated Life-threatening consequences; urgent radiologic or operative | |
| Cystitis noninfective Microscop increase ir dysuria, or of incontin Definition: A disorder characterized by inflan Hematuria Asymptom diagnostic intervention | oic hematuria; minimal<br>n frequency, urgency,<br>r nocturia; new onset | Moderate hematuria; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative | urgent radiologic or operative | Death |
| increase in dysuria, or of inconting properties. Definition: A disorder characterized by inflant diagnostic interventions. | n frequency, urgency,<br>r nocturia; new onset | increase in frequency, urgency,<br>dysuria, nocturia or<br>incontinence; urinary catheter<br>placement or bladder irrigation<br>indicated; limiting instrumental | medications or hospitalization indicated; elective endoscopic, radiologic or operative | urgent radiologic or operative | Death |
| diagnostic | | ADL | | | |
| diagnostic<br>interventio | nmation of the bladder | which is not caused by an infection | on of the urinary tract. | | |
| Definition: A disorder characterized by labora | natic; clinical or<br>c observations only;<br>on not indicated | Symptomatic; urinary catheter or bladder irrigation indicated; limiting instrumental ADL | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated; limiting self care ADL | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| | atory test results that ir | ndicate blood in the urine. | | | |
| diagnostic | natic; clinical or<br>cobservations only;<br>on not indicated | - | - | - | - |
| Definition: A disorder characterized by labor | atory test results that ir | ndicate the presence of free hemo | oglobin in the urine. | | |
| Proteinuria 1+ protein <1.0 g/24 | uria; urinary protein<br>hrs | Adults: 2+ proteinuria; urinary<br>protein 1.0 - 3.4 g/24 hrs;<br>Pediatric: urine P/C<br>(Protein/Creatinine) ratio 0.5 -<br>1.9 | Adults: urinary protein >=3.5 g/24 hrs;<br>Pediatric: urine P/C >1.9 | - | - |
| Definition: A disorder characterized by labor | atory test results that ir | ndicate the presence of excessive | protein in the urine. It is predomin | antly albumin, but also globulin. | |
| symptoms<br>nonprescr<br>indicated | natic or mild<br>s; occasional use of<br>iption analgesics | Symptomatic; oral antiemetics indicated; around the clock nonprescription analgesics or any oral narcotic analgesics indicated | Hospitalization indicated; IV intervention (e.g., analgesics, antiemetics); elective endoscopic or radiologic intervention indicated | Life-threatening consequences; urgent radiologic, endoscopic or operative intervention indicated | Death |
| Definition: A disorder characterized by the fo | - | | | | |
| Renal colic Mild pain r<br>activity; no<br>medication | not interfering with | Moderate pain; limiting instrumental ADL; prescription medication indicated | Hospitalization indicated;<br>limiting self care ADL | - | - |

| Renal and urinary disorders | | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Renal hemorrhage | Mild symptoms; intervention not indicated | Analgesics and hematocrit monitoring indicated | Transfusion, radiation, or<br>hospitalization indicated;<br>elective radiologic, endoscopic<br>or operative intervention<br>indicated | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| | ed by bleeding from the kidney. | | | | |
| Jrinary fistula | - | Noninvasive intervention indicated; urinary or suprapubic catheter placement indicated | Limiting self care ADL; elective radiologic, endoscopic or operative intervention indicated; permanent urinary diversion indicated | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between any part of the urinary s | system and another organ or anato | omic site. | |
| Urinary frequency | Present | Limiting instrumental ADL; medical management indicated | - | - | - |
| Definition: A disorder characteriz | ed by urination at short intervals. | | T | | |
| Urinary incontinence | Occasional (e.g., with coughing, sneezing, etc.), pads not indicated | Spontaneous; pads indicated;<br>limiting instrumental ADL | Intervention indicated (e.g., clamp, collagen injections); operative intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by inability to control the flow o | f urine from the bladder. | | | |
| Urinary retention | Urinary, suprapubic or intermittent catheter placement not indicated; able to void with some residual | Placement of urinary,<br>suprapubic or intermittent<br>catheter placement indicated;<br>medication indicated | Elective operative or radiologic<br>intervention indicated;<br>substantial loss of affected<br>kidney function or mass | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by accumulation of urine within | the bladder because of the inabili | ity to urinate. | | |
| Urinary tract obstruction | Asymptomatic; clinical or diagnostic observations only | Symptomatic but no<br>hydronephrosis, sepsis or renal<br>dysfunction; urethral dilation,<br>urinary or suprapubic catheter<br>indicated | Symptomatic and altered organ function (e.g., hydronephrosis, or renal dysfunction); elective radiologic, endoscopic or operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by blockage of the normal flow | of contents of the urinary tract. | | | |
| Jrinary tract pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | mfort in the urinary tract. | T | | |
| Jrinary urgency | Present | Limiting instrumental ADL;<br>medical management indicated | - | - | - |
| Definition: A disorder characteriz | ed by a sudden compelling urge to | urinate. | T | | |
| Irine discoloration | Present | - | - | - | - |
| Definition: A disorder characteriz | ed by a change in the color of the | urine. | T | T | |
| Renal and urinary disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate, local or noninvasive intervention indicated; limiting instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |

| | Rep | productive system and be | | | |
|---|---|---|---|---|---|
| | | | Grade | | I |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Azoospermia | - | - | Absence of sperm in ejaculate | - | - |
| Definition: A disorder characteri | zed by laboratory test results that in | ndicate complete absence of speri | matozoa in the semen. | | |
| Breast atrophy | Minimal asymmetry; minimal atrophy | Moderate asymmetry; moderate atrophy | Asymmetry >1/3 of breast volume; severe atrophy | - | - |
| Definition: A disorder characteri | zed by underdevelopment of the bro | east. | | | |
| Breast pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensation | n in the breast region. | | | |
| Dysmenorrhea | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by abnormally painful abdomina | al cramps during menses. | | | |
| Dyspareunia | Mild discomfort or pain<br>associated with vaginal<br>penetration; discomfort relieved<br>with use of vaginal lubricants or<br>estrogen | Moderate discomfort or pain<br>associated with vaginal<br>penetration; discomfort or pain<br>partially relieved with use of<br>vaginal lubricants or estrogen | Severe discomfort or pain<br>associated with vaginal<br>penetration; discomfort or pain<br>unrelieved by vaginal lubricants<br>or estrogen | - | - |
| Definition: A disorder characteri | zed by painful or difficult coitus. | | | | |
| Ejaculation disorder | Diminished ejaculation | Anejaculation or retrograde ejaculation | - | - | - |
| Definition: A disorder characteri | zed by problems related to ejaculat | ion. This category includes prema | ture, delayed, retrograde and pain | ıful ejaculation. | |
| Erectile dysfunction | Decrease in erectile function<br>(frequency or rigidity of<br>erections) but intervention not<br>indicated (e.g., medication or<br>use of mechanical device,<br>penile pump) | Decrease in erectile function (frequency/rigidity of erections), erectile intervention indicated, (e.g., medication or mechanical devices such as penile pump) | Decrease in erectile function (frequency/rigidity of erections) but erectile intervention not helpful (e.g., medication or mechanical devices such as penile pump); placement of a permanent penile prosthesis indicated (not previously present) | | |
| Definition: A disorder characteri | zed by the persistent or recurrent ir | ,<br>nability to achieve or to maintain a | n erection during sexual activity. | • | , |
| Fallopian tube obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteri | zed by blockage of the normal flow | of the contents in the fallopian tub | e. | _ | |
| Fallopian tube stenosis | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., organ resection) | Death |
| Definition: A disorder characteri | zed by a narrowing of the fallopian | tube lumen. | T | 1 | 1 |
| Female genital tract fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | n between a female reproductive s | ystem organ and another organ or | r anatomic site. | T |
| Feminization acquired | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder characteri | zed by the development of seconda | ary female sex characteristics in m | ales due to extrinsic factors. | | |
| Genital edema | Mild swelling or obscuration of anatomic architecture on close inspection | Readily apparent obscuration of<br>anatomic architecture;<br>obliteration of skin folds; readily<br>apparent deviation from normal<br>anatomic contour | Lymphorrhea; gross deviation<br>from normal anatomic contour;<br>limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by swelling due to an excessive | e accumulation of fluid in the genit | als. | | |
| Gynecomastia | Asymptomatic breast enlargement | Symptomatic (e.g., pain or psychosocial impact) | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteri | zed by excessive development of the | ne breasts in males. | | | |
| Hematosalpinx | Minimal bleeding identified on imaging study or laparoscopy; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| | Rep | productive system and b | reast disorders | | |
|---|---|---|---|---|---|
| | | T | Grade | Г | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characte | rized by the presence of blood in a fa | allopian tube.<br>I | <u> </u> | | |
| Irregular menstruation | Intermittent menses with skipped menses for no more than 1 to 3 months | Intermittent menses with skipped menses for more than 4 to 6 months | Persistent amenorrhea for more than 6 months | - | - |
| Definition: A disorder characte | rized by irregular cycle or duration of | menses. | Τ | | |
| Lactation disorder | Mild changes in lactation, not<br>significantly affecting production<br>or expression of breast milk | Changes in lactation,<br>significantly affecting breast<br>production or expression of<br>breast milk | - | - | - |
| Definition: A disorder characte | rized by disturbances of milk secretic | on. It is not necessarily related to p | pregnancy that is observed in fema | ales and can be observed in males | S. |
| Menorrhagia | Mild; iron supplements indicated | Moderate symptoms; medical intervention indicated (e.g., hormones) | Severe; transfusion indicated;<br>surgical intervention indicated<br>(e.g., hysterectomy) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by abnormally heavy vaginal bl | eeding during menses. | _ | | |
| Nipple deformity | Asymptomatic; asymmetry with slight retraction and/or thickening of the nipple areolar complex | Symptomatic; asymmetry of<br>nipple areolar complex with<br>moderate retraction and/or<br>thickening of the nipple areolar<br>complex | - | - | - |
| Definition: A disorder characte | rized by a malformation of the nipple | | _ | | |
| Oligospermia | Sperm concentration >48 million/mL or motility >68% | Sperm concentration 13 - 48 million/mL or motility 32 - 68% | Sperm concentration <13<br>million/mL or motility <32% | - | - |
| Definition: A disorder characte | rized by a decrease in the number of | f spermatozoa in the semen. | T | Т | |
| Ovarian hemorrhage | Minimal bleeding identified on imaging study or laproscopy; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the ovary. | | T | ı | 1 |
| Ovarian rupture | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by tearing or disruption of the c | varian tissue. | • | • | • |
| Ovulation pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characte ovarian follicle. | rized by marked discomfort sensatio | n in one side of the abdomen betv | veen menstrual cycles, around the | time of the discharge of the ovum | from the |
| Pelvic floor muscle weakness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic, not interfering with bladder, bowel, or vaginal function; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a reduction in the strength o | f the muscles of the pelvic floor. | | | |
| Pelvic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characte | rized by marked discomfort sensatio | n in the pelvis. | | | |
| Penile pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characte | rized by marked discomfort sensatio | n in the penis. | | | |
| Perineal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | omfort in the area between the ger | ital organs and the anus. | | |
| Premature menopause | - | - | Present | - | - |
| Definition: A disorder characte | rized by ovarian failure before the ag | ge of 40. Symptoms include hot fla | shes, night sweats, mood swings | and a decrease in sex drive. | |
| Prostatic hemorrhage | Minimal bleeding identified on<br>imaging study; intervention not<br>indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| | Rep | productive system and b | reast disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | ed by bleeding from the prostate of | pland. | _ | | 1 |
| Prostatic obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz stream, and incomplete emptying | | secondary to enlargement of the p | prostate gland. This results in voidi | ng difficulties (straining to void, slo | ow urine |
| Prostatic pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | _ |
| · | | instrumental ADL | ADL | | |
| | ed by a sensation of marked disco | 1 | | | |
| Scrotal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n in the scrotal area. | | | |
| Spermatic cord hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the spermation | cord. | | | |
| Spermatic cord obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by blockage of the normal flow | of the contents of the spermatic c | ord. | | |
| Testicular disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic but not interfering with urination or sexual activities; intervention not indicated; limiting instrumental ADL | Severe symptoms; interfering with urination or sexual function; limiting self care ADL; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by involvement of the testis. | | | | |
| Testicular hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the testis. | T | T | Т | 1 |
| Testicular pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the testis. | | | |
| Uterine fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | n between the uterus and another | organ or anatomic site. | | |
| Uterine hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the uterus. | | | | |
| Uterine obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by blockage of the uterine outle | et. | | | |
| Uterine pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the uterus. | | • | |
| Vaginal discharge | Mild vaginal discharge (greater than baseline for patient) | Moderate to heavy vaginal discharge; use of perineal pad or tampon indicated | - | - | - |
| Definition: A disorder characteriz | ed by vaginal secretions. Mucus n | 1 | ।<br>discharged from the vagina natura | lly, especially during the childbear | ing years. |
| Vaginal dryness | Mild vaginal dryness not interfering with sexual function | Moderate vaginal dryness interfering with sexual function or causing frequent discomfort | Severe vaginal dryness resulting in dyspareunia or severe discomfort | - | - |
| Definition: A disorder characteriz | ed by an uncomfortable feeling of | | | 1 | 1 |

| Reproductive system and breast disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Vaginal fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the vagina and another | organ or anatomic site. | | |
| Vaginal hemorrhage | Minimal bleeding identified on clinical exam or imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the vagina. | | | | |
| Vaginal inflammation | Mild discomfort or pain, edema, or redness | Moderate discomfort or pain,<br>edema, or redness; limiting<br>instrumental ADL | Severe discomfort or pain,<br>edema, or redness; limiting self<br>care ADL; small areas of<br>mucosal ulceration | Widespread areas of mucosal<br>ulceration; life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation involving the v | agina. Symptoms may include red | lness, edema, marked discomfort | and an increase in vaginal dischar | ge. |
| Vaginal obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by blockage of vaginal canal. | | | _ | |
| Vaginal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | mfort in the vagina. | | | |
| Vaginal perforation | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the vaginal wall. | ' | ' | ' | |
| Vaginal stricture | Asymptomatic; mild vaginal shortening or narrowing | Vaginal narrowing and/or<br>shortening not interfering with<br>physical examination | Vaginal narrowing and/or<br>shortening interfering with the<br>use of tampons, sexual activity<br>or physical examination | - | Death |
| Definition: A disorder characteriz | ed by a narrowing of the vaginal ca | anal. | • | • | |
| Vaginismus | Mild discomfort or pain<br>associated with vaginal<br>spasm/tightening; no impact<br>upon sexual function or physical<br>examination | Moderate discomfort or pain<br>associated with vaginal<br>spasm/tightening; disruption in<br>sexual function and physical<br>examination | Severe discomfort or pain<br>associated with vaginal<br>spasm/tightening; unable to<br>tolerate vaginal penetration or<br>physical examination | - | - |
| Definition: A disorder characteriz intercourse. | ed by involuntary spasms of the pe | elvic floor muscles, resulting in pa | thologic tightness of the vaginal w | all during penetration such as duri | ng sexua |
| Reproductive system and breast<br>disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Respi | ratory, thoracic and med | iastinal disorders | | |
|---|---|---|---|---|---|
| | · | • | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Adult respiratory distress syndrome | - | - | Present with radiologic findings; intubation not indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characterize surgery. | ed by progressive and life-threater | ning pulmonary distress in the abs | ence of an underlying pulmonary | condition, usually following major t | rauma or |
| Allergic rhinitis | Mild symptoms; intervention not indicated | intervention indicated | - | - | - |
| | ed by an inflammation of the nasal<br>of the sinuses, eyes, middle ear, a | - | - : | - | ay aiso |
| Apnea | - | - | Present; medical intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characterize | | A4 | D | 1 :6- 41 | D41- |
| Aspiration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Altered eating habits; coughing or choking episodes after eating or swallowing; medical intervention indicated (e.g., suction or oxygen) | Dyspnea and pneumonia<br>symptoms (e.g., aspiration<br>pneumonia); hospitalization<br>indicated; unable to aliment<br>orally | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characterize | ed by inhalation of solids or liquids | into the lungs. | 1 | ı | ı |
| Atelectasis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., dyspnea, cough); medical intervention indicated (e.g., chest physiotherapy, suctioning); bronchoscopic suctioning | Oxygen indicated;<br>hospitalization or elective<br>operative intervention indicated<br>(e.g., stent, laser) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characterize | ed by the collapse of part or the er | ntire lung. | T | T | |
| Bronchial fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder characterize | ed by an abnormal communication | between the bronchus and anoth | ner organ or anatomic site. | | |
| Bronchial obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., mild<br>wheezing); endoscopic<br>evaluation indicated;<br>radiographic evidence of<br>atelectasis/lobar collapse;<br>medical management indicated<br>(e.g., steroids, bronchodilators) | Shortness of breath with stridor; endoscopic intervention indicated (e.g., laser, stent placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characterize | ed by blockage of a bronchus pass | sage, most often by bronchial seci | retions and exudates. | | |
| Bronchial stricture | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., rhonchi or wheezing) but without respiratory distress; medical intervention indicated (e.g., steroids, bronchodilators) | Shortness of breath with stridor; endoscopic intervention indicated (e.g., laser, stent placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| | ed by a narrowing of the bronchial | | T_ | | |
| Bronchopleural fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL; endoscopic or operative intervention indicated (e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder characterize | ed by an abnormal communication | between a bronchus and the pleu | ural cavity. | Г | |
| Bronchopulmonary hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characterize | ed by bleeding from the bronchial | wall and/or lung parenchyma. | | | |

| | Respi | ratory, thoracic and med | iastinal disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Bronchospasm | Mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Limiting self care ADL; oxygen saturation decreased | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by a sudden contraction of the | smooth muscles of the bronchial | wall. | T | I |
| Chylothorax | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thoracentesis or tube drainage indicated | Severe symptoms; elective operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by milky pleural effusion (abnor | rmal collection of fluid) resulting fr | om accumulation of lymph fluid in | the pleural cavity. | |
| Cough | Mild symptoms; nonprescription intervention indicated | Moderate symptoms, medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteri by a distinctive sound. | zed by sudden, often repetitive, spa | asmodic contraction of the thoracion | c cavity, resulting in violent release | e of air from the lungs and usually | accompanied |
| Dyspnea | Shortness of breath with moderate exertion | Shortness of breath with minimal exertion; limiting instrumental ADL | Shortness of breath at rest;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an uncomfortable sensation | of difficulty breathing. | | 1 | T |
| Epistaxis | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated (e.g., nasal packing, cauterization; topical vasoconstrictors) | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by bleeding from the nose. | | | • | |
| Hiccups | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe symptoms; interfering with sleep; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by repeated gulp sounds that re | esult from an involuntary opening | and closing of the glottis. This is a | ttributed to a spasm of the diaphra | igm. |
| Hoarseness | Mild or intermittent voice change; fully understandable; self-resolves | Moderate or persistent voice changes; may require occasional repetition but understandable on telephone; medical evaluation indicated | Severe voice changes including predominantly whispered speech | - | - |
| Definition: A disorder characteri | zed by harsh and raspy voice arisir | g from or spreading to the larynx. | | | |
| Hypoxia | - | Decreased oxygen saturation<br>with exercise (e.g., pulse<br>oximeter <88%); intermittent<br>supplemental oxygen | Decreased oxygen saturation at<br>rest (e.g., pulse oximeter <88%<br>or PaO2 <=55 mm Hg) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | zed by a decrease in the level of ox | İ | <u> </u> | | |
| Laryngeal edema | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated (e.g., dexamethasone, epinephrine, antihistamines) | Stridor; respiratory distress;<br>hospitalization indicated | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| | zed by swelling due to an excessive | | | | <b>.</b> |
| Laryngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube thoracostomy or medical management indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; endoscopic or operative intervention indicated (e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder characteri | zed by an abnormal communication | between the larynx and another | organ or anatomic site. | | |
| Laryngeal hemorrhage | Mild cough or trace hemoptysis; laryngoscopic findings | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder characteri | zed by bleeding from the larynx. | I | | T | T |
| Laryngeal inflammation | Mild sore throat; raspy voice | Moderate sore throat; analgesics indicated | Severe throat pain; endoscopic intervention indicated | - | - |
| Definition: A disorder characteri | zed by an inflammation involving th | e larynx. | | | |

| | Respi | ratory, thoracic and med | iastinal disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Laryngeal mucositis | Endoscopic findings only; mild discomfort with normal intake | Moderate discomfort; altered oral intake | Severe pain; severely altered eating/swallowing; medical intervention indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | , | e mucous membrane of the larynx | | | |
| Laryngeal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by blockage of the laryngeal ai | rway. | | | |
| Laryngeal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids) | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a narrowing of the laryngeal | airway. | | | |
| Laryngopharyngeal dysesthesia | Mild symptoms; no anxiety; intervention not indicated | Moderate symptoms; mild<br>anxiety, but no dyspnea; short<br>duration of observation and or<br>anxiolytic indicated; limiting<br>instrumental ADL | Severe symptoms; dyspnea and swallowing difficulty; limiting self care ADL | Life-threatening consequences | Death |
| Definition: A disorder characterize | ed by an uncomfortable persistent | sensation in the area of the laryn | gopharynx. | | |
| Laryngospasm | - | Transient episode; intervention not indicated | Recurrent episodes;<br>noninvasive intervention<br>indicated (e.g., breathing<br>technique, pressure point<br>massage) | Persistent or severe episodes<br>associated with syncope; urgent<br>intervention indicated (e.g.,<br>fiberoptic laryngoscopy,<br>intubation, botox injection) | Death |
| Definition: A disorder characterize | ed by paroxysmal spasmodic mus | cular contraction of the vocal cord | s. | • | • |
| Mediastinal hemorrhage | Radiologic evidence only;<br>minimal symptoms; intervention<br>not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated<br>(e.g., hemostasis of bleeding<br>site) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by bleeding from the mediastin | um. | T | Γ | T |
| Nasal congestion | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Associated with bloody nasal discharge or epistaxis | - | - |
| Definition: A disorder characterize | ed by obstruction of the nasal pas | sage due to mucosal edema. | 1 | I | ı |
| Pharyngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an abnormal communication | n between the pharynx and anothe | er organ or anatomic site. | Т | l |
| Pharyngeal hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characterize | | | | | |
| Pharyngeal mucositis | Endoscopic findings only;<br>minimal symptoms with normal<br>oral intake; mild pain but<br>analgesics not indicated | Moderate pain and analgesics indicated; altered oral intake; limiting instrumental ADL | Severe pain; unable to<br>adequately aliment or hydrate<br>orally; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an inflammation involving th | e mucous membrane of the phary | nx. | r | T |
| Pharyngeal necrosis | - | - | Inability to aliment adequately<br>by GI tract; tube feeding or TPN<br>indicated; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the pharynx. | | | |
| Pharyngeal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor; endoscopic intervention indicated (e.g., stent, laser) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder characteriz | ed by a narrowing of the pharynge | al airway. | | | |
| Pharyngolaryngeal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the pharyngolaryngeal region. | | T | Т |
| Pleural effusion | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; intervention indicated (e.g., diuretics or limited therapeutic thoracentesis) | Symptomatic with respiratory distress and hypoxia; surgical intervention including chest tube or pleurodesis indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by an increase in amounts of flu | uid within the pleural cavity. Symp | toms include shortness of breath, | cough and marked chest discomfo | ort. |
| Pleural hemorrhage | Asymptomatic; mild hemorrhage confirmed by thoracentesis | Symptomatic or associated with pneumothorax; chest tube drainage indicated | >1000 ml of blood evacuated;<br>persistent bleeding (150-200<br>ml/hr for 2 - 4 hr); persistent<br>transfusion indicated; elective<br>operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the pleural ca | vity. | | | |
| Pleuritic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the pleura. | <b>.</b> | <b>.</b> | ı |
| Pneumonitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; oxygen indicated | Life-threatening respiratory compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder characteriz | ed by inflammation focally or diffus | sely affecting the lung parenchyma | a.<br>T | Ι | |
| Pneumothorax | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; intervention indicated (e.g., tube placement without sclerosis) | Sclerosis and/or operative intervention indicated; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by abnormal presence of air in | the pleural cavity resulting in the c | collapse of the lung. | | |
| Postnasal drip | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder characteriz | ed by excessive mucous secretion | in the back of the nasal cavity or | throat, causing sore throat and/or | coughing. | ı |
| Productive cough | Occasional/minimal production of sputum with cough | Moderate sputum production;<br>limiting instrumental ADL | Persistent or copious production of sputum; limiting self care ADL | | - |
| | ed by expectorated secretions upo | | | I | |
| Pulmonary edema | Radiologic findings only;<br>minimal dyspnea on exertion | Moderate dyspnea on exertion;<br>medical intervention indicated;<br>limiting instrumental ADL | Severe dyspnea or dyspnea at rest; oxygen indicated; limiting self care ADL | Life-threatening respiratory<br>compromise; urgent intervention<br>or intubation with ventilatory<br>support indicated | Death |
| Definition: A disorder characteriz | ed by accumulation of fluid in the I | ung tissues that causes a disturba | ance of the gas exchange that may | lead to respiratory failure. | |
| Pulmonary fibrosis | Mild hypoxemia; radiologic pulmonary fibrosis <25% of lung volume | radiographic pulmonary fibrosis<br>25 - 50% | Severe hypoxemia; evidence of right-sided heart failure; radiographic pulmonary fibrosis >50 - 75% | Life-threatening consequences (e.g., hemodynamic/pulmonary complications); intubation with ventilatory support indicated; radiographic pulmonary fibrosis >75% with severe honeycombing | Death |
| | ed by the replacement of the lung | tissue by connective tissue, leadir | ī i i i i i i i i i i i i i i i i i i i | tory failure or right heart failure. | |
| Pulmonary fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Limiting self care ADL;<br>endoscopic stenting or<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characte | erized by an abnormal communication | between the lung and another or | gan or anatomic site. | T | 1 |
| Pulmonary hypertension | Minimal dyspnea; findings on physical exam or other evaluation | Moderate dyspnea, cough;<br>requiring evaluation by cardiac<br>catheterization and medical<br>intervention | Severe symptoms, associated<br>with hypoxemia, right heart<br>failure; oxygen indicated | Life-threatening airway<br>consequences; urgent<br>intervention indicated (e.g.,<br>tracheotomy or intubation) | Death |
| Definition: A disorder characte | erized by an increase in pressure with | nin the pulmonary circulation due to | o lung or heart disorder. | T | 1 |
| Respiratory failure | - | - | - | Life-threatening consequences; urgent intervention, intubation, or ventilatory support indicated | Death |
| | erized by impaired gas exchange by t | he respiratory system resulting in | nypoxemia and a decrease in oxy | genation of the tissues that may be | e associate |
| with an increase in arterial lev | rels of carbon dioxide. | | | | |
| Retinoic acid syndrome | Fluid retention; <3 kg of weight<br>gain; intervention with fluid<br>restriction and/or diuretics<br>indicated | Moderate signs or symptoms; steroids indicated | Severe symptoms;<br>hospitalization indicated | Life-threatening consequences; ventilatory support indicated | Death |
| | erized by weight gain, dyspnea, pleur | al and pericardial effusions, leukoo | cytosis and/or renal failure original | ly described in patients treated wit | h all-trans |
| retinoic acid.<br>Sinus disorder | Asymptomatic mucosal crusting; blood-tinged secretions | Symptomatic stenosis or edema/narrowing interfering with airflow; limiting instrumental ADL | Stenosis with significant nasal obstruction; limiting self care ADL | Necrosis of soft tissue or bone; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by involvement of the paranasa | al sinuses. | | | |
| Sleep apnea | Snoring and nocturnal sleep arousal without apneic periods | Moderate apnea and oxygen desaturation; excessive daytime sleepiness; medical evaluation indicated; limiting instrumental ADL | Oxygen desaturation;<br>associated with hypertension;<br>medical intervention indicated;<br>limiting self care ADL | Cardiovascular or<br>neuropsychiatric symptoms;<br>urgent operative intervention<br>indicated | Death |
| | | 1 | | | |
| Sneezing | Mild symptoms; intervention not indicated | intervention indicated | - | - | - |
| Definition: A disorder characte | erized by the involuntary expulsion of | air from the nose. | | | |
| Sore throat | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL; limiting ability to swallow | - | - |
| Definition: A disorder characte | erized by of marked discomfort in the | throat | | <b>.</b> | 1 |
| Stridor | - | - | Respiratory distress limiting self care ADL; medical intervention indicated | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder characte | erized by a high pitched breathing sou | und due to laryngeal or upper airw | ay obstruction. | | |
| Tracheal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder characte | erized by an abnormal communication | between the trachea and another | r organ or anatomic site. | Τ | |
| Tracheal mucositis | Endoscopic findings only;<br>minimal hemoptysis, pain, or<br>respiratory symptoms | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe pain; hemorrhage or respiratory symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an inflammation involving th | e mucous membrane of the trache | ea.<br>I | <u> </u> | 1 |
| Tracheal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids) | Stridor or respiratory distress<br>limiting self care ADL;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| | | I to the state of | 1 | T . | 1 |

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Voice alteration | Mild or intermittent change from normal voice | Moderate or persistent change<br>from normal voice; still<br>understandable | Severe voice changes including predominantly whispered speech; may require frequent repetition or face-to-face contact for understandability; may require assistive technology | - | - |
| Definition: A disorder characterize | zed by a change in the sound and/o | or speed of the voice. | | | |
| Wheezing | Detectable airway noise with minimal symptoms | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | . , , , . | | Death |
| Definition: A disorder characterize | zed by a high-pitched, whistling sou | and during breathing. It results from | m the narrowing or obstruction of t | he respiratory airways. | |
| Respiratory, thoracic and mediastinal disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Sk | in and subcutaneous tis | sue disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Alopecia | Hair loss of <50% of normal for that individual that is not obvious from a distance but only on close inspection; a different hair style may be required to cover the hair loss but it does not require a wig or hair piece to camouflage | Hair loss of >=50% normal for that individual that is readily apparent to others; a wig or hair piece is necessary if the patient desires to completely camouflage the hair loss; associated with psychosocial impact | - | - | - |
| Definition: A disorder characteri | zed by a decrease in density of hair | ı | l<br>ndividual at a given age and body | location | |
| Body odor | Mild odor; physician intervention<br>not indicated; self care<br>interventions | | - | - | - |
| Definition: A disorder characterization | zed by an abnormal body smell res | ulting from the growth of bacteria | on the body. | | |
| Bullous dermatitis | Asymptomatic; blisters covering <10% BSA | Blisters covering 10 - 30% BSA;<br>painful blisters; limiting<br>instrumental ADL | Blisters covering >30% BSA;<br>limiting self care ADL | Blisters covering >30% BSA;<br>associated with fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| Definition: A disorder characterization | zed by inflammation of the skin cha | racterized by the presence of bull | ae which are filled with fluid. | | |
| Dry skin | Covering <10% BSA and no associated erythema or pruritus | Covering 10 - 30% BSA and associated with erythema or pruritus; limiting instrumental ADL | Covering >30% BSA and associated with pruritus; limiting self care ADL | - | - |
| Definition: A disorder characterization | zed by flaky and dull skin; the pores | are generally fine, the texture is | a papery thin texture. | | |
| Erythema multiforme | Target lesions covering <10%<br>BSA and not associated with<br>skin tenderness | Target lesions covering 10 -<br>30% BSA and associated with<br>skin tenderness | Target lesions covering >30%<br>BSA and associated with oral or<br>genital erosions | Target lesions covering >30%<br>BSA; associated with fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| Definition: A disorder characterization | zed by target lesions (a pink-red rin | g around a pale center). | | | |
| Erythroderma | - | Erythema covering >90% BSA without associated symptoms; limiting instrumental ADL | Erythema covering >90% BSA with associated symptoms (e.g., pruritus or tenderness); limiting self care ADL | Erythema covering >90% BSA with associated fluid or electrolyte abnormalities; ICU care or burn unit indicated | Death |
| Definition: A disorder characterize | zed by generalized inflammatory er | ythema and exfoliation. The inflan | nmatory process involves > 90% o | f the body surface area. | |
| Fat atrophy | Covering <10% BSA and asymptomatic | Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL | Covering >30% BSA;<br>associated with erythema or<br>tenderness; limiting self-care<br>ADL | - | - |
| Definition: A disorder characterization | zed by shrinking of adipose tissue. | <u> </u> | T | T | |
| Hirsutism | In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or removal of hair | In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair removal to camouflage; associated with psychosocial impact | - | - | - |
| Definition: A disorder characterizandrogen control (beard, moust | zed by the presence of excess hair<br>ache, chest, abdomen) | growth in women in anatomic site | s where growth is considered to b | e a secondary male characteristic | and under |
| Hyperhidrosis | Limited to one site (palms, soles, or axillae); self care interventions | Involving >1 site; patient seeks medical intervention; associated with psychosocial impact | Generalized involving sites<br>other than palms, soles, or<br>axillae; associated with<br>electrolyte/hemodynamic<br>imbalance | - | - |
| Definition: A disorder abarestori | zed by excessive perspiration. | , | • | • | , |

| | Sk | in and subcutaneous tis | sue disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypertrichosis | Increase in length, thickness or<br>density of hair that the patient is<br>either able to camouflage by<br>periodic shaving or removal of<br>hairs or is not concerned | Increase in length, thickness or<br>density of hair at least on the<br>usual exposed areas of the<br>body [face (not limited to<br>beard/moustache area) | - | - | - |
| | enough about the overgrowth to use any form of hair removal | plus/minus arms] that requires<br>frequent shaving or use of<br>destructive means of hair<br>removal to camouflage;<br>associated with psychosocial<br>impact | | | |
| Definition: A disorder characteriz | zed by hair density or length beyon | d the accepted limits of normal in | a particular body region, for a part | icular age or race. | |
| Hypohidrosis | - | Symptomatic; limiting instrumental ADL | Increase in body temperature;<br>limiting self care ADL | Heat stroke | Death |
| Definition: A disorder characteriz | 1 | Cavaring 10, 200/ DCA and | Covering > 200/ DCA and | | |
| Lipohypertrophy | Asymptomatic and covering <10% BSA | Covering 10 - 30% BSA and associated tenderness; limiting instrumental ADL | Covering >30% BSA and<br>associated tenderness and<br>narcotics or NSAIDs indicated;<br>lipohypertrophy; limiting self<br>care ADL | | - |
| Definition: A disorder characterize | zed by hypertrophy of the subcutan | eous adipose tissue at the site of | multiple subcutaneous injections of | of insulin. | |
| Nail discoloration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characterize | zed by a change in the color of the | nail plate. | _ | | |
| Nail loss | Asymptomatic separation of the nail bed from the nail plate or nail loss | Symptomatic separation of the nail bed from the nail plate or nail loss; limiting instrumental ADL | - | - | - |
| Definition: A disorder characteriz | ed by loss of all or a portion of the | nail. | | | |
| Nail ridging | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characteriz | red by vertical or horizontal ridges | on the nails. | ' | ' | |
| Pain of skin | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characterize | zed by marked discomfort sensation | n in the skin. | Т | Т | 1 |
| Palmar-plantar erythrodysesthesia syndrome | Minimal skin changes or<br>dermatitis (e.g., erythema,<br>edema, or hyperkeratosis)<br>without pain | Skin changes (e.g., peeling,<br>blisters, bleeding, edema, or<br>hyperkeratosis) with pain;<br>limiting instrumental ADL | Severe skin changes (e.g.,<br>peeling, blisters, bleeding,<br>edema, or hyperkeratosis) with<br>pain; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by redness, marked discomfort | , swelling, and tingling in the palm | s of the hands or the soles of the | feet. | 1 |
| Periorbital edema | Soft or non-pitting | Indurated or pitting edema; topical intervention indicated | Edema associated with visual disturbance; increased intraocular pressure, glaucoma or retinal hemorrhage; optic neuritis; diuretics indicated; operative intervention indicated | - | - |
| Definition: A disorder characteriz | zed by swelling due to an excessive | e accumulation of fluid around the | orbits of the face. | | |
| Photosensitivity | Painless erythema and<br>erythema covering <10% BSA | Tender erythema covering 10 - 30% BSA | Erythema covering >30% BSA and erythema with blistering; photosensitivity; oral corticosteroid therapy indicated; pain control indicated (e.g., narcotics or NSAIDs) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | l<br>zed by an increase in sensitivity of | l<br>the skin to light. | maroonoo or Noriba) | I<br> | [ |

| | Sk | in and subcutaneous tis | sue disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pruritus | Mild or localized; topical intervention indicated | Intense or widespread;<br>intermittent; skin changes from<br>scratching (e.g., edema,<br>papulation, excoriations,<br>lichenification, oozing/crusts);<br>oral intervention indicated;<br>limiting instrumental ADL | Intense or widespread;<br>constant; limiting self care ADL<br>or sleep; oral corticosteroid or<br>immunosuppressive therapy<br>indicated | - | - |
| Definition: A disorder characteriz | ed by an intense itching sensation | • | | | |
| Purpura Definition: A disorder characteriz | Combined area of lesions covering <10% BSA ed by hemorrhagic areas of the sk | Combined area of lesions<br>covering 10 - 30% BSA;<br>bleeding with trauma<br>in and mucous membrane. Newel | Combined area of lesions covering >30% BSA; spontaneous bleeding resions appear reddish in color. C | -<br>Dider lesions are usually a darker i | -<br>ourple color |
| and eventually become a browni | sh-yellow color. | | T | T | |
| Rash acneiform | Papules and/or pustules<br>covering <10% BSA, which may<br>or may not be associated with<br>symptoms of pruritus or<br>tenderness | Papules and/or pustules covering 10 - 30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| Definition: A disorder characteriz | ed by an eruption of papules and p | pustules, typically appearing in fac | e, scalp, upper chest and back. | | |
| Rash maculo-papular | Macules/papules covering<br><10% BSA with or without<br>symptoms (e.g., pruritus,<br>burning, tightness) | Macules/papules covering 10 -<br>30% BSA with or without<br>symptoms (e.g., pruritus,<br>burning, tightness); limiting<br>instrumental ADL | Macules/papules covering<br>>30% BSA with or without<br>associated symptoms; limiting<br>self care ADL | - | - |
| Definition: A disorder characteriz | ed by the presence of macules (fla | t) and papules (elevated). Also kr | nown as morbillform rash, it is one | of the most common cutaneous a | dverse |
| events, frequently affecting the u | pper trunk, spreading centripetally | and associated with pruritus. | I | T | 1 |
| Scalp pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the skin covering the top and | the back of the head. | | 1 |
| Skin atrophy | Covering <10% BSA;<br>associated with telangiectasias<br>or changes in skin color | Covering 10 - 30% BSA;<br>associated with striae or<br>adnexal structure loss | Covering >30% BSA; associated with ulceration | - | - |
| Definition: A disorder characteriz | ed by the degeneration and thinnir | ng of the epidermis and dermis. | T | T | 1 |
| Skin hyperpigmentation | Hyperpigmentation covering <10% BSA; no psychosocial impact | Hyperpigmentation covering >10% BSA; associated psychosocial impact | - | - | - |
| Definition: A disorder characteriz | ed by darkening of the skin due to | excessive melanin deposition. | | | |
| Skin hypopigmentation | Hypopigmentation or<br>depigmentation covering <10%<br>BSA; no psychosocial impact | Hypopigmentation or<br>depigmentation covering >10%<br>BSA; associated psychosocial<br>impact | - | - | - |
| Definition: A disorder characteriz | ed by loss of skin pigment. | | | | _ |
| Skin induration | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration, unable to<br>slide or pinch skin; limiting joint<br>movement or orifice (e.g.,<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| Definition: A disorder characteriz | ed by an area of hardness in the s | kin. | I | T | |
| Skin ulceration | Combined area of ulcers <1 cm;<br>nonblanchable erythema of<br>intact skin with associated<br>warmth or edema | Combined area of ulcers 1 - 2<br>cm; partial thickness skin loss<br>involving skin or subcutaneous<br>fat | Combined area of ulcers >2 cm;<br>full-thickness skin loss involving<br>damage to or necrosis of<br>subcutaneous tissue that may<br>extend down to fascia | Any size ulcer with extensive destruction, tissue necrosis, or damage to muscle, bone, or supporting structures with or without full thickness skin loss | Death |
| Definition: A disorder characteriz | ed by circumscribed, inflammatory | and necrotic erosive lesion on the | e skin. | | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Stevens-Johnson syndrome | - | - | Skin sloughing covering <10%<br>BSA with associated signs (e.g.,<br>erythema, purpura, epidermal<br>detachment and mucous<br>membrane detachment) | Skin sloughing covering 10 - 30% BSA with associated signs (e.g., erythema, purpura, epidermal detachment and mucous membrane detachment) | Death |
| Definition: A disorder characteriz nucous membranes. | ed by less than 10% total body ski | n area separation of dermis. The | syndrome is thought to be a hyper | sensitivity complex affecting the sl | kin and the |
| Telangiectasia | Telangiectasias covering <10%<br>BSA | Telangiectasias covering >10%<br>BSA; associated with<br>psychosocial impact | - | - | - |
| Definition: A disorder characteriz | ed by local dilatation of small vess | els resulting in red discoloration o | f the skin or mucous membranes. | _ | |
| Toxic epidermal necrolysis | - | - | - | Skin sloughing covering >=30%<br>BSA with associated symptoms<br>(e.g., erythema, purpura, or<br>epidermal detachment) | Death |
| Definition: A disorder characteriz mucous membranes. | ed by greater than 30% total body | skin area separation of dermis. The | he syndrome is thought to be a hy | persensitivity complex affecting the | e skin and |
| Urticaria | Urticarial lesions covering <10%<br>BSA; topical intervention<br>indicated | Urticarial lesions covering 10 - 30% BSA; oral intervention indicated | Urticarial lesions covering >30%<br>BSA; IV intervention indicated | - | - |
| Definition: A disorder characteriz | ed by an itchy skin eruption charac | cterized by wheals with pale interi | ors and well-defined red margins. | | |
| Skin and subcutaneous tissue disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |

| Social circumstances | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Menopause | Menopause occurring at age 46 - 53 years of age | Menopause occurring at age 40 - 45 years of age | Menopause occurring before age 40 years of age | - | - |
| Definition: A disorder characteriz | ed by the permanent cessation of | menses, usually defined by 12 cor | nsecutive months of amenorrhea i | n a woman over 45 years of age. | |
| Social circumstances - Other, specify | , | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Surgical and medical procedures | | | | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Surgical and medical procedures - Other, specify | 1 | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Vascular disord | ers | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Capillary leak syndrome | - | Symptomatic; medical intervention indicated | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by leakage of intravascular fluid<br>syndromes, low-flow states, ischer | · · | - | <del>-</del> | |
| Flushing | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Symptomatic, associated with hypotension and/or tachycardia; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by episodic reddening of the fa | ce. | T | I | |
| Hematoma | Mild symptoms; intervention not indicated | Minimally invasive evacuation or aspiration indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a localized collection of bloc | od, usually clotted, in an organ, sp | ace, or tissue, due to a break in th | e wall of a blood vessel. | |
| Hot flashes | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by an uncomfortable and temp | orary sensation of intense body w | armth, flushing, sometimes accom | panied by sweating upon cooling. | |
| Hypertension | Prehypertension (systolic BP<br>120 - 139 mm Hg or diastolic<br>BP 80 - 89 mm Hg) | Stage 1 hypertension (systolic<br>BP 140 - 159 mm Hg or<br>diastolic BP 90 - 99 mm Hg);<br>medical intervention indicated;<br>recurrent or persistent (>=24<br>hrs); symptomatic increase by<br>>20 mm Hg (diastolic) or to | Stage 2 hypertension (systolic BP >=160 mm Hg or diastolic BP >=100 mm Hg); medical intervention indicated; more than one drug or more intensive therapy than previously used indicated | Life-threatening consequences<br>(e.g., malignant hypertension,<br>transient or permanent<br>neurologic deficit, hypertensive<br>crisis); urgent intervention<br>indicated<br>Pediatric: Same as adult | Death |
| | | >140/90 mm Hg if previously<br>WNL; monotherapy indicated<br>Pediatric: recurrent or persistent<br>(>=24 hrs) BP >ULN;<br>monotherapy indicated | Pediatric: Same as adult | | |
| | ed by a pathological increase in bl | T . | i i | Ī | D#- |
| Hypotension | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | hospitalization indicated | Life-threatening and urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a blood pressure that is belo | ow the normal expected for an indi | ividual in a given environment. | | |
| Lymph leakage | - | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the loss of lymph fluid into the | ne surrounding tissue or body cavi | ity. | T | |
| Lymphedema | Trace thickening or faint discoloration | Marked discoloration; leathery skin texture; papillary formation; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by excessive fluid collection in | tissues that causes swelling. | | | |
| Lymphocele | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | - | - |
| Definition: A disorder characteriz | ed by a cystic lesion containing lyr | mph. | 1 | | |
| Peripheral ischemia | - | Brief (<24 hrs) episode of ischemia managed non-surgically and without permanent deficit | Recurring or prolonged (>=24 hrs) and/or invasive intervention indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by impaired circulation to an ex | ctremity. | 1 | 1 | 1 |
| Phlebitis | - | Present | - | - | - |
| Definition: A disorder characteriz | ed by inflammation of the wall of a | vein. | , | | |
| Superficial thrombophlebitis | - | Present | - | - | - |
| Definition: A disorder characteriz | ed by a blood clot and inflammatic | on involving a superficial vein of the | e extremities. | | |

| Vascular disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Superior vena cava syndrome | Asymptomatic; incidental finding of SVC thrombosis | Symptomatic; medical intervention indicated (e.g., anticoagulation, radiation or chemotherapy) | Severe symptoms; multi-<br>modality intervention indicated<br>(e.g., anticoagulation,<br>chemotherapy, radiation,<br>stenting) | Life-threatening consequences;<br>urgent multi-modality<br>intervention indicated (e.g.,<br>lysis, thrombectomy, surgery) | Death |
| Definition: A disorder characteriz cough, orthopnea and headache | ed by obstruction of the blood flow . | in the superior vena cava. Signs | and symptoms include swelling an | d cyanosis of the face, neck, and | upper arms, |
| Thromboembolic event | Venous thrombosis (e.g., superficial thrombosis) | Venous thrombosis (e.g.,<br>uncomplicated deep vein<br>thrombosis), medical<br>intervention indicated | thrombus), medical intervention | Life-threatening (e.g.,<br>pulmonary embolism,<br>cerebrovascular event, arterial<br>insufficiency); hemodynamic or<br>neurologic instability; urgent<br>intervention indicated | Death |
| Definition: A disorder characteriz | ed by occlusion of a vessel by a th | rombus that has migrated from a | distal site via the blood stream. | | |
| Vasculitis | Asymptomatic, intervention not indicated | ntervention not Moderate symptoms, medical intervention indicated intervention indicated steroids) Moderate symptoms, medical intervention indicated (steroids) | | Life-threatening; evidence of peripheral or visceral ischemia; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation involving the w | rall of a vessel. | ' | | , |
| Visceral arterial ischemia | - | Brief (<24 hrs) episode of ischemia managed medically and without permanent deficit | Prolonged (>=24 hrs) or recurring symptoms and/or invasive intervention indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by a decrease in blood supply | due to narrowing or blockage of a | visceral (mesenteric) artery. | | |
| Vascular disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |







NIH Publication No. 09-5410 Revised June 2010 Reprinted June 2010



## 13.5 Appendix 5: Acute Radiation Morbidity Scoring Criteria (RTOG)

| | [0] | [1] | [2] | [3] | [4] |
|---|---|---|---|---|---|
| | No change<br>over baseline | Follicular, faint or dull erythema/ epilation/dry desquamation/ decreased sweating | Tender or bright erythema, patchy moist desquamation/moderate edema | Confluent, moist<br>desquamation other than<br>skin folds, pitting edema | Ulceration, hemorrhage, necrosis |
| UPPER G.I. | No change | weight loss from pretreatment baseline/ nausea not requiring antiemetics/ abdominal discomfort not requiring parasympatholytic drugs or | Anorexia with <=15% weight loss from pretreatment baseline/nausea &/ or vomiting requiring antiemetics/ abdominal pain requiring analgesics | Anorexia with >15% weight loss from pretreatment baseline or requiring N-G tube or parenteral support. Nausea &/or vomiting requiring tube or parenteral support/abdominal pain, severe despite medication/hematemesis or melena/ abdominal distention (flat plate radiograph demonstrates distended bowel loops | Ileus, subacute or acute obstruction, perforation, GI bleeding requiring transfusion/abdominal pain requiring tube decompression or bowel diversion |
| LOWER G.I.<br>INCLUDING<br>PELVIS | No change | change in quality of bowel habits not requiring medication/ rectal discomfort not requiring analgesics | mucous discharge not | Diarrhea requiring parenteral support/ severe mucous or blood discharge necessitating sanitary pads/abdominal distention (flat plate radiograph demonstrates distended bowel loops) | Acute or subacute obstruction, fistula or perforation; GI bleeding requiring transfusion; abdominal pain or tenesmus requiring tube decompression or bowel diversion |

Date: 27 April 2016 v 2.1

| | [0] | [1] | [2] | [3] | [4] |
|---|---|---|---|---|---|
| GENITOURINARY | No change | Frequency of urination or nocturia twice pretreatment habit/ dysuria, urgency not requiring medication | which is less frequent<br>than every hour.<br>Dysuria, urgency,<br>bladder spasm<br>requiring local | more frequently/ dysuria,<br>pelvis pain or bladder<br>spasm requiring regular,<br>frequent narcotic/gross | Hematuria requiring transfusion/ acute bladder obstruction not secondary to clot passage, ulceration or necrosis |
| HEMATOLOGIC<br>WBC (X 1000) | >=4.0 | 3.0 - <4.0 | 2.0 - <3.0 | 1.0 - <2.0 | <1.0 |
| PLATELETS<br>(X 1000) | >=100 | 75 - <100 | 50 - <75 | 25 - <50 | <25 or spontaneous bleeding |
| NEUTROPHILS | >=1.9 | 1.5 - <1.9 | 1.0 - <1.5 | 0.5 - <1.0 | <0.5 or sepsis |
| HEMOGLOBIN<br>(GM %) | >11 | 11-9.5 | <9.5 - 7.5 | <7.5 - 5.0 | |
| HEMATOCRIT (%) | >=32 | 28 - <32 | K / X | Packed RBC transfusion required | |

GUIDELINES: The acute morbidity criteria are used to score/grade toxicity from radiation therapy. The criteria are relevant from day 1, the commencement of therapy, through day 90.

The evaluator must attempt to discriminate between disease- and treatment-related signs and symptoms.

An accurate baseline evaluation prior to commencement of therapy is necessary.

All toxicities Grade 3, 4 or 5\* must be verified by the Principal Investigator.

\*ANY TOXICITY WHICH CAUSED DEATH IS GRADED 5.

#### 13.6 Appendix 6: Preparation of Investigational Products

VGX-3100 and INO-9012 will be combined by the site pharmacist into a single syringe for subjects using the following procedure:

- 0. Using aseptic technique, withdraw 1.2 mL from the vial SynCon<sup>TM</sup> VGX-3100 with a 3 mL syringe and inject into an empty sterile vial. Set this "mixing" vial which now contains 1.2 mL of VGX-3100 aside.
- 1. Using a new 1 mL syringe, withdraw 0.12 mL from the vial SynCon<sup>TM</sup> INO-9012 and add the 0.12 mL to the "mixing" vial containing 1.2 mL of VGX-3100. The final volume of this vial should now be 1.32 mL of INO-3112(VGX-3100 / INO-9012).
- 2. Using a 3 mL syringe, withdraw 1.1 mL of INO-3112 from the "mixing" vial. This syringe will be used for dosing of subjects.

# 13.7 Appendix 7: CELLECTRA®-5P Error Reporting Form

| Please complete the form and fax to | or scan th | e form to | | |
|---|---|---|---|---|
| Protocol# Site# | Subject ID | Wee | k# | Visit Date |
| | ~u0]000 ID | | | , 2010 15 1010 |
| DEVICE INFORMATION CELLECTRA®-5P Serial No: | | | | |
| Located on label on the front cover | | | | |
| CELLECTRA®-5P Applicator Serial No: | | | | |
| Located on label on the handle | | | | |
| CELLECTRA®-5P Array Lot No: | | | | |
| Located on label on the package | | | | |
| Time of Electroporation: | <b>Location of Treat</b> | ment/EP: | Deltoid Right/Lo | eft |
| ☐ Other Location, specify: | IN | I-5P, was the | | I? □ YES □ NO |
| If EP Guide was used, please provide reason | on and include subject' | s BMI. | | |
| Was injection successful? | □YES | □N | O | |
| If NO, please provide reason and include n | | | | |
| Did the display on the device read EP su | ooossful? □ VES | | □NO | |
| If NO, please check all complications that | | ihe complicat | | |
| ☐ Impedance Test Error message displayed | | _ | | |
| ☐ Electroporation Error message displayed | = | | | |
| | • | on Error secu | on below | |
| ☐ EP aborted by trigger or keypad error m | | | | |
| ☐ Battery level too low for electroporation | | | | |
| ☐ Difficulty inserting array into muscle or | skın | | | |
| ☐ Other, please specify below | | | | |
| Describe device complication below (con | tinue on back if neces | ssary): | | |
| Total # of arrays used: | | | | |
| Impedance Test Error | | | | |
| Was the array inserted in subject's arm? | $\square$ YES | $\square$ NO | Total # of atter | mpts: |
| Were all attempts performed on the same d | ay? □ YES | $\square$ NO | | |
| | (provid | e other date(s) | ): | |
| Was a different location used for each atter | npt? □ YES | | NO | |
| Was a new array used for each attempt? | $\square$ YES | | NO | |
| Please provide any additional information | on below (continue on | back if neces | ssary): | |
| Electroporation Error | | | | |
| Were there 3 (IM) or 4 (ID) involuntary mu | iscle contractions? | □ YES | □ NO (how m | nanv |
| Was the array fully inserted in the subject's | | □ YES | | папу |
| Was the array inserted in the subject s | | □ YES | □ NO | |
| | • | □ YES | □ NO | |
| Did the needles of the array appear damage | | | | |
| If you were provided a sharps shuttle, please Please provide any additional information | | | | |
| any additional miormatic | in perow (continue on | DACK II HECE | 55a1 y j. | |

Date: 27 April 2016 v 2.1

### 13.8 Appendix 8: New York Heart Association (NYHA) Functional Classification

The NYHA classifies heart failure into classes based on functional limitations and severity.

| Class | Patient Symptoms |
|---|---|
| Class I (Mild) | No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea (shortness of breath). |
| Class II (Mild) | Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea. |
| Class III<br>(Moderate) | Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea. |
| Class IV (Severe) | Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased. |

<sup>\*</sup>The Criteria Committee of the New York Heart Association. *Nomenclature and Criteria for Diagnosis of Diseases of the Heart and Great Vessels.* 9th ed. Boston, Mass: Little, Brown & Co; 1994:253-256.

## 13.9 Appendix 9: Participant Reminder Card

## **Appendix 10. Participant Reminder Card**

| Participant ID: | Date of Study Treatment |
|---|---|
| Site of Injection: | Right Arm Left Arm Right Leg Left Leg |
| study treatment. The you received the stu | e complete this reminder card in the evening after and for three days following your ne "Evening of study treatment" column should include any side effects from the time dy treatment until 11:59pm of that day. Days 1, 2 and 3 should include any side effects 00 am) to 11:59 pm of that day (1 day, 2 days or 3 days after receiving the study |
| Take this card with y | you to your next study visit for review with the study team. If you have any questions, |

To describe the size of any area that is red or swollen, please use the measuring tool provided with this reminder card to indicate the approximate size of a circle that could fully cover the area of redness or swelling.

or if you have any concerns or side effects that you'd like to discuss, please contact your study team.

| Possible side effects | Evening of study treatment | 1 day after study<br>treatment | 2 days after study treatment | 3 days after study treatment | Date Resolved |
|---|---|---|---|---|---|
| Redness or | □None | □None | □None | □None | |
| bruising at | □ Diameter (in cm) | □ Diameter (in cm) | □ Diameter (in cm) | □ Diameter (in cm) | If date |
| treatment | from measuring | from measuring | from measuring | from measuring | unknown: |
| site | tool: | tool: | tool: | tool: | □ 1 week** |
| | | | | | □ 2 weeks** |
| | ☐ Greater than 7cm | ☐ Greater than 7cm | ☐ Greater than 7cm | ☐ Greater than 7cm | □ 3 weeks** |
| | □None | □None | □None | □None | |
| | ☐ A little, controlled | □ A little, | □ A little, | □ A little, | |
| Pain at | with OTC* meds | controlled with | controlled with | controlled with | If date |
| treatment | ☐ A lot, OTC meds | OTC* meds | OTC* meds | OTC* meds | unknown: |
| site | didn't work, | ☐ A lot, OTC meds | ☐ A lot, OTC meds | ☐ A lot, OTC meds | □ 1 week** |
| Site | prevented normal | didn't work, | didn't work, | didn't work, | □ 2 weeks** |
| | activity | prevented | prevented | prevented | □ 3 weeks** |
| | | normal activity | normal activity | normal activity | |
| | □None | □ None | □None | □None | |
| Swelling/ | ☐ Diameter (in cm) | ☐ Diameter (in cm) | ☐ Diameter (in cm) | ☐ Diameter (in cm) | If date |
| Edema at | from measuring | from measuring | from measuring | from measuring | unknown: |
| treatment | tool: | tool: | tool: | tool: | □ 1 week** |
| site | | | | | □ 2 weeks** |
| | ☐ Greater than 7cm | ☐ Greater than 7cm | ☐ Greater than 7cm | ☐ Greater than 7cm | □ 3 weeks** |
| | Please record | Please record | Please record | Please record | |
| Oral | below: | below: | below: | below: | |
| Temperature | □°F | □°F | □°F | □°F | |
| remperature | □ °C | □ °C | □ °C | □ °C | |

<sup>\*</sup> OTC – Over the counter analgesics or painkillers such as paracetamol, acetaminophen (e.g. Tylenol®) or ibuprofen (e.g. Advil® or Motrin®).

<sup>\*\*</sup> After study treatment

| Did you have | Did you have any other side effects? | | | | |
|---|---|---|---|---|---|
| Other side<br>effects<br>(insert below) | Evening of study treatment | 1 day after study<br>treatment | 2 days after study treatment | 3 days after study treatment | Date Resolved |
| | ☐ Mild, barely | ☐ Mild, barely | ☐ Mild, barely | ☐ Mild, barely | |
| | noticeable | noticeable | noticeable | noticeable | If date |
| | □ Moderate, | □ Moderate, | □ Moderate, | □ Moderate, | unknown: |
| | slowed me | slowed me | slowed me | slowed me | □ 1 week** |
| | down | down | down | down | □ 2 weeks** |
| | □ Severe | □ Severe | □ Severe | □ Severe | □ 3 weeks** |
| | ☐ Mild, barely | ☐ Mild, barely | ☐ Mild, barely | □ Mild, barely | |
| | noticeable | noticeable | noticeable | noticeable | If date |
| | □ Moderate, | □ Moderate, | □ Moderate, | □ Moderate, | unknown: |
| | slowed me | slowed me | slowed me | slowed me | □ 1 week** |
| | down | down | down | down | □ 2 weeks** |
| | □ Severe | □ Severe | □ Severe | □ Severe | □ 3 weeks** |
| Did you contact the study team for any symptoms that were not listed here or the severity was worse than the available choices? Yes No About Injection Site Reaction The most common reactions to the study treatment are reactions at the injection site such as an area of redness, a little bruising, possible swelling, and temporary pain. For most people, it is not bothersome at all and disappears in a day or two. However, it may last a week or more. If you have any concerns about your symptoms, have any ongoing injection site reactions or side effects that are still present more than 3 days after the study treatment, please contact your study team. | | | | | |
| Coord | Coordinator Name: Coordinator Telephone Number: | | | | |
| | Did you take any medications for your injection site reactions or other symptoms? Yes (record below) No | | | | |
| | Is there anything else that you would like to discuss with the study team? Yes (record below) No | | | | |

#### 13.10 Appendix 10: RECIST

A. Response will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria:

#### i. Definitions

Evaluable for Target Disease response: Only those participants who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for target disease response. These participants will have their response classified according to the definitions stated below. (Note: Participants who exhibit objective disease progression prior to the end of cycle 1 will also be considered evaluable.)

Evaluable Non-Target Disease Response: Participants who have lesions present at baseline that are evaluable but do not meet the definitions of measurable disease, have received at least one cycle of therapy, and have had their disease reevaluated will be considered evaluable for non-target disease. The response assessment is based on the presence, absence, or unequivocal progression of the lesions.

#### ii. <u>Disease Parameters</u>

<u>Measurable disease</u>. Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as  $\geq 20$  mm by chest x-ray or  $\geq 10$  mm with CT scan, MRI, or calipers by clinical exam. All tumor measurements must be recorded in <u>millimeters</u> (or decimal fractions of centimeters).

<u>Malignant lymph nodes.</u> To be considered pathologically enlarged and measurable, a lymph node must be  $\geq 15$  mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.

Non-measurable disease. All other lesions (or sites of disease), including small lesions (longest diameter <10 mm or pathological lymph nodes with ≥10 to <15 mm short axis), are considered non-measurable disease. Bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusions, lymphangitis cutis/pulmonitis, inflammatory breast disease, abdominal masses (not followed by CT or MRI), and cystic lesions are all considered non-measurable.

Note: Cystic lesions that meet the criteria for radiographically defined simple cysts should not be considered as malignant lesions (neither measurable nor non-measurable) since they are, by definition, simple cysts.

'Cystic lesions' thought to represent cystic metastases can be considered as measurable lesions, if they meet the definition of measurability described above. However, if non-cystic lesions are present in the same participant, these are preferred for selection as target lesions.

Target lesions. All measurable lesions up to a maximum of 2 lesions per organ and 5 lesions in total, representative of all involved organs, should be identified as target lesions and recorded and measured at baseline. Target lesions should be selected on the basis of their size (lesions with the longest diameter), be representative of all involved organs, but in addition should be those that lend themselves to reproducible repeated measurements. It may be the case that, on occasion, the largest lesion does not lend itself to reproducible measurement in which circumstance the next largest lesion which can be measured reproducibly should be selected. A sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) for all target lesions will be calculated and reported as the baseline sum diameters. If lymph nodes are to be included in the sum, then only the short axis is added into the sum. The baseline sum diameters will be used as reference to further characterize any objective tumor regression in the measurable dimension of the disease.

<u>Non-target lesions</u>. All other lesions (or sites of disease) including any measurable lesions over and above the 5 target lesions should be identified as **non-target lesions** and should also be recorded at baseline. Measurements of these lesions are not required, but the presence, absence, or in rare cases unequivocal progression of each should be noted throughout follow up.

#### iii. Response Criteria

Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.

<u>Partial Response (PR)</u>: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

<u>Progressive Disease (PD)</u>: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).

<u>Stable Disease (SD)</u>: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

### iv. Evaluation of Non-Target Lesions

<u>Complete Response (CR)</u>: Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).

Note: If tumor markers are initially above the upper normal limit, they must normalize for a patient to be considered in complete clinical response.

<u>Non-CR/Non-PD:</u> Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits.

<u>Progressive Disease (PD)</u>: Appearance of one or more new lesions and/or *unequivocal progression* of existing non-target lesions. *Unequivocal progression* should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.

Although a clear progression of "non-target" lesions only is exceptional, the opinion of the treating physician should prevail in such circumstances, and the progression status should be confirmed at a later time by the review panel (or Principal Investigator).

#### v. Evaluation of New Lesions

The finding of a new lesion should be unequivocal (i.e. not due to difference in scanning technique, imaging modality, or findings thought to represent something other than tumor (for example, some 'new' bone lesions may be simply healing or flare of pre-existing lesions). However, a lesion identified on a follow-up scan in an anatomical location that was not scanned at baseline is considered new and will indicate PD. If a new lesion is equivocal (because of small size etc.), follow-up evaluation will clarify if it truly represents new disease and if PD is confirmed, progression should be declared using the date of the initial scan on which the lesion was discovered.

#### vi. Evaluation of Best Overall Response

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The

patient's best response assignment will depend on the achievement of both target and non-target disease.

#### Time point response: patients with target (+/- non-target disease)

| <b>Target Lesions</b> | Non-Target | New Lesions | Overall |
|-----------------------|------------------|-------------|----------|
| | Lesions | | Response |
| CR | CR | No | CR |
| CR | Non-CR/Non- | No | PR |
| | PD | | |
| CR | Not evaluated | No | PR |
| PR | Non-CR/Non- | No | PR |
| | PD/not evaluated | | |
| SD | Non-CR/Non- | No | SD |
| | PD/not evaluated | | |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |

#### Time point response: patients with non-target disease only

| Non-Target Lesions | New Lesions | <b>Overall Response</b> |
|---|---|---|
| CR | No | CR |
| Non-CR/non-PD | No | Non-CR/non-PD* |
| Not all evaluated | No | not evaluated |
| Unequivocal PD | Yes or No | PD |
| Any | Yes | PD |
| * 'Non-CR/non-PD' is preferred over 'stable disease' for non-target | | |
| disease since SD is increasingly used as an endpoint for assessment | | |
| of efficacy in some trials so to assign this category when no lesions | | |

#### vii. Confirmation/Duration of Response

can be measured is not advised

Confirmation: Confirmation of PR and CR is required to ensure responses identified are not the results of measurement error. This will also permit appropriate interpretation of results in the context of historical data where response has traditionally required confirmation.

<u>Duration of overall response</u>: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded on study)

Date: 27 April 2016 v 2.1

<u>Duration of overall complete response</u>: The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented.

<u>Duration of stable disease</u>: Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest sum on study (if baseline sum is the smallest, this is the reference for calculation of PD).

B. **Progression Free Survival**- any progression of disease as defined below will be recorded and summarized for subjects in the individual cohorts and overall

Overall Survival: Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive.

<u>Progression-Free Survival</u>: Progression-Free Survival (PFS) is defined as the time from randomization (or registration) to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.

<u>Time to Progression</u>: Time to Progression (TTP) is defined as the time from randomization (or registration) to progression, or censored at date of last disease evaluation for those without progression reported